

# CLINICAL TRIAL PROTOCOL INCLUDING AMENDMENTS NOS. 01 TO 09 BNT162-01

**Version:** 13.0 **Date:** 12 JAN 2022

Sponsor: BioNTech SE

Trial title: A multi-site, Phase I/II, 2-part, dose escalation trial investigating the safety and

immunogenicity of four prophylactic SARS-CoV-2 RNA vaccines against

COVID-19 using different dosing regimens in healthy and

immunocompromised adults

Brief title: A multi-site Phase I/II trial investigating the safety and effects of four BNT162

vaccines against COVID-19 in healthy and immunocompromised adults

Trial phase: Phase I/II

**Indication:** Protection against COVID-19

**Product:** BNT162: SARS-CoV-2 - RNA lipid nanoparticle (RNA-LNP) vaccines utilizing

different RNA formats, i.e., BNT162a1, BNT162b1, BNT162b2 and BNT162c2.

Coordinating and Dr. Dr. med. Armin Schultz, CRS Clinical Research Services

Principal investigator: Mannheim GmbH, Germany (tel.: +49 621 15045

**Trial sites:** Multiple sites in Germany. For further details of the study sites and site

personnel, see the Trial Master File (TMF).

Contract research organization (CRO):

CRS Clinical Research Services Mannheim GmbH, Germany

Sponsor's medical

representative:

Dr. Svetlana Shpyro, Director Clinical Development, BioNTech SE

**Sponsor:** BioNTech SE, An der Goldgrube 12, 55131 Mainz, Germany

Regulatory identifiers: EudraCT no.: 2020-001038-36; ClinicalTrials.gov: NCT04380701; WHO UTN:

U1111-1249-4220

**Medical Monitor:** Contact information will be provided separately

See the next page for a history of all sponsor-approved document versions and Section 10.10 for the rationale for all approved versions.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| Document history | Date | Version number | Valid for |
|------------------------|-------------|----------------|-----------|
| First approved version | 09 Apr 2020 | 2.0 | Germany |
| Amendment No. 1 | 17 Apr 2020 | 3.0 | Germany |
| Amendment No. 2 | 13 May 2020 | 4.0 | Germany |
| Amendment No. 3 | 26 May 2020 | 5.0 | Germany |
| Amendment No. 4 | 09 Jun 2020 | 6.0 | Germany |
| Amendment No. 4 | 26 Jun 2020 | 7.0 | Germany |
| Amendment No. 5 | 21 Jul 2020 | 8.0 | Germany |
| Amendment No. 6 | 05 OCT 2020 | 9.0 | Germany |
| Amendment No. 6 | 28 OCT 2020 | 10.0 | Germany |
| Amendment No. 7 | 04 DEC 2020 | 11.0 | Germany |
| Amendment No. 8 | 01 MAR 2021 | 12.0 | Germany |
| Amendment No. 9 | 12 JAN 2022 | 13.0 | Germany |


### 1 PROTOCOL SUMMARY

### 1.1 Trial synopsis

Trial number: BNT162-01

#### Trial title

A multi-site, Phase I/II, 2-part, dose escalation trial investigating the safety and immunogenicity of four prophylactic SARS-CoV-2 RNA vaccines against COVID-19 using different dosing regimens in healthy and immunocompromised adults

### **Objectives and endpoints**

| Objectives | Endpoints <sup>a</sup> |
|---|---|
| Primary objective | |
| (All cohorts) To describe the safety and tolerability profiles of | <ul> <li>Solicited local reactions at the injection site (pain, tenderness,<br/>erythema/redness, induration/swelling) recorded up to 7 d after each<br/>immunization (trial days 8 and 29).</li> </ul> |
| prophylactic BNT162<br>vaccines in healthy adults<br>after single dose (SD;<br>prime only) or prime/boost | <ul> <li>Solicited systemic reactions (nausea, vomiting, diarrhea, headache,<br/>fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and<br/>fever) recorded up to 7 d after each immunization (trial days 8<br/>and 29).</li> </ul> |
| (P/B) immunization. | <ul> <li>The proportion of subjects with at least 1 unsolicited treatment-<br/>emergent adverse event (TEAE):</li> </ul> |
| | <ul> <li>For BNT162a1, BNT162b1, BNT162b2, and BNT162c2 (P/B):<br/>occurring up to 21 d after the prime immunization (trial day 22)<br/>and 28 d after the boost immunization (trial day 50).</li> </ul> |
| | <ul> <li>For BNT162c2 (SD): The proportion of subjects with at least<br/>1 unsolicited TEAE occurring up to 28 d after the immunization<br/>(trial day 29).</li> </ul> |

### Secondary objectives

#### (All cohorts)

To describe the immune response in healthy adults after SD or P/B immunization measured by a functional antibody titer, e.g., virus neutralization test (VNT) or an equivalent assay available by the time of trial conduct.

#### For BNT162a1, BNT162b1, BNT162b2, and BNT162c2 (P/B)

As compared to baseline at 7 and 21 d after primary immunization (trial days 8 and 22) and at 7, 14 b, 21, 28, 63, and 162 d after the boost immunization (trial days 29 to 184):

- Functional antibody responses (titers).
- Fold increase in functional antibody titers.
- Number of subjects with seroconversion defined as a minimum of 4-fold increase of functional antibody titers as compared to baseline.

#### For BNT162c2 (SD)

As compared to baseline at 7, 21, 28, 42, 84, and 183 d after the primary immunization (trial days 8 to 184):

- Functional antibody responses (titers).
- Fold increase in functional antibody titers.
- Number of subjects with seroconversion defined as a minimum of
   4-fold increase of functional antibody titers as compared to baseline.

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


#### **Objectives** Endpoints a

### For Cohort 14 with BNT162b2

As compared to baseline at 7, 14, and 21 d after primary immunization (trial days 8, 15, and 22) and at 7, 28, and 162 d after the boost immunization (trial days 29, 50, and 184):

- Functional antibody responses (titers).
- Fold increase in functional antibody titers.
- Number of subjects with seroconversion defined as a minimum of 4-fold increase of functional antibody titers as compared to baseline.

#### **Exploratory objectives**



# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01




### Trial design

This trial has two parts. Part A and Part B. Due to changes in the overall clinical development plan, Part B will no longer be conducted. The objectives originally described for Part B have been implemented in the ongoing development via a pivotal Phase I/II/III trial BNT162-02/C4591001 (NCT04368728).

Part A is for dose ranging of four different vaccines (BNT162a1, BNT162b1, BNT162b2, and BNT162c2) will be undertaken with dose escalation and de-escalation plus the evaluation of interim dose levels. It also includes dose ranging in older subjects.

The vaccines BNT162a1, BNT162b1, BNT162b2, and BNT162c2 will be administered using a P/B regimen. The vaccine BNT162c2 will also be administered using a SD regimen.

BNT162b2, for which the dose regimen has been determined in the dose ranging in Part A of this trial, has now entered efficacy evaluation in the ongoing development via a pivotal Phase I/II/III trial BNT162-02/C4591001 (NCT04368728). Therefore, for BNT162b2, amendment 06 introduced expansion cohorts designed to expand the existing safety profiling to a broader population and to enable detailed characterization of the adaptive immune responses, including determine factors that impact them. These cohorts will involve healthy and immunocompromised populations treated according to the selected dosing posology and exploring an alternative posology.

The chosen trial design reflects discussion and advice from the Paul-Ehrlich-Institut (PEI) obtained in scientific advice meetings held in February, March, and June 2020 in response to a fast-changing situation.

For a summary of the trial as a flow diagram, see the Schema in Section 1.2. For the planned assessments and visits, see the Schedule of Activities (SoA) in Section 1.3.

#### Part A

The first part of the trial (Part A) will follow a dose escalation design. Discretionary dose de-escalation and refinement is also planned. Part A will consist of a screening/treatment phase and a follow-up phase.

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### **Dose ranging cohorts:**

Trial subjects with the first-in-human (FIH) immunization will be immunized using a sentinel dosing/subject staggering (EMA 2017 guidance "Strategies to Identify and Mitigate Risks for First-in-Human and Early Clinical Trials with Investigational Medicinal Products"). The FIH starting dose and the planned escalation/de-escalation doses are given in Table 1. Dose escalation rules have been defined in this protocol to guide dose escalation.

For all cohorts, if the investigator considers necessary, the planned observation periods before proceeding to dose further subjects in the same group may be prolonged by 24 hours (h).

Dose de-escalation in the case of possible vaccine-related toxicities will be guided by the Safety Review Committee (SRC), as required.

In Cohort 1, the sentinel dosing/subject staggering process will be as follows:

- One sentinel subject will be dosed on one day.
- If the dosing in this subject was considered to be safe and well tolerated by the investigator after 24±2 h observation on site, a 5 further subjects will be dosed (with intervals of at least 1 h between subjects).
- If the dosing in these 5 subjects was considered to be safe and well tolerated by the investigator based on 48 h data (24±2 h observation on site and phone interview for assessment 48±2 h after immunization; in addition to the available 48±2 h data from the sentinel subject):
  - The remaining 6 subjects in the group will be dosed (with intervals of at least 30 minutes [min] between subjects).
  - o If approved by the SRC, the next planned escalation dose (see Table 1) will be initiated. The data assessed by the SRC comprises 48 h data for 6 subjects including observation on site, short summary of phone interview (including statement about diary reports), vital signs, investigator reported local and systemic reactions, treatment-emergent adverse events (TEAEs), solicited local & systemic reactions, blood/clinical laboratory data, and brief physical examination outcome.
  - If approved by the SRC, the planned de-escalation dose in Cohort 3 will be initiated.

For any subsequent dose escalation cohorts (to doses higher than the maximum already tested for a vaccine candidate), the sentinel/subject staggering process will be as follows:

- Two sentinel subjects will be dosed on one day (with intervals of at least 30 min between subjects).
- If the dosing in these subjects was considered to be safe and well tolerated by the investigator after 24±2 h observation on site, a 4 further subjects will be dosed (with intervals of at least 30 min between subjects).
- If the dosing in these 4 subjects was considered to be safe and well tolerated by the investigator based on 48 h data (24±2 h observation on site and phone interview for

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


assessment 48±2 h after immunization; in addition to the available 48 h data from the sentinel subjects):

- The remaining 6 subjects in the group will be dosed (with intervals of at least 30 min between subjects).
- o If approved by the SRC, the next planned escalation dose (see Table 1) will be initiated. The data assessed by the SRC comprises 48 h data for 6 subjects including observation on site, short summary of phone interview (including statement about diary reports), vital signs, investigator reported local and systemic reactions, TEAEs, solicited local & systemic reactions, blood/clinical laboratory data, and brief physical examination outcome.

The maximum allowed dose for each vaccine candidate is defined in Table 1.

For the planned dose de-escalation cohorts, 12 subjects may be dosed on one day (with intervals of at least 30 min between subjects). The doses in these cohorts in younger adults must be lower than doses that have shown acceptable tolerability in younger adults (based on the data from 12 subjects up until 48 h after the first dose). The same dose will not be administered twice, i.e., in two cohorts.

For BNT162b1 and BNT162b2, administration of the planned 10 μg dose in older subjects (Cohort 8) may start once at least a 30 μg dose has shown acceptable tolerability in younger adults (based on the data from 12 subjects up until 48 h after the boost dose).

The dose in Cohort 8 must also be confirmed by the SRC. In Cohort 8, 12 subjects will be dosed using a sentinel dosing/subject staggering (2-4-6) process with intervals of at least 1 h between the first 6 subjects and then at least 30 min intervals for the remaining 6 subjects.

For BNT162b1 and BNT162b2, administration of the planned dose escalation cohorts in older adults (Cohorts 9 and 10), 12 subjects will be dosed using a sentinel dosing/subject staggering (2-4-6) process with intervals of at least 30 min between subjects. The doses planned in these cohorts will only be administered if the dose is confirmed by the SRC.

The doses planned for Cohorts 8 to 10 are defined in Table 2.

For the unplanned dose de-escalation cohorts, i.e., where the SRC requests the use of a reduced dose for safety reasons, 12 subjects may be dosed on one day with intervals of at least 30 min between subjects (as for planned de-escalation cohorts).

Note: BNT162b1 and BNT162b2 are nucleoside modified RNAs, while BNT162a1 and BNT162c2 are both non-modified uridine containing RNAs. RNA modification is known to impact the extent of innate immune activation at a given dose level, and thus potentially the extent of reactogenicity. Therefore, tolerability data obtained with one of the vaccine variants of each of these pairs may be potentially informative for the respective other one and should be taken in consideration by the SRC for recommendations of lower or interim doses.

In the case that an individual experiences dose limiting toxicities or that the frequency or pattern of adverse events (AEs) within a sub-cohort gives cause for concern, the

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


investigator may request by phone an ad hoc review by the SRC, at any time, before further doses of a given vaccine construct are administered.

### Expansion cohorts:

Protocol amendment 6.0 implemented three additional cohorts (Cohorts 11, 12, and 13) comprising additional 150 trial subjects aged from 18 to 85 years receiving BNT162b2 only.

BNT162b2 has entered a Phase II/III evaluation of efficacy, with the intent to support an application for marketing authorization. The dosing regimen under investigation is two 30 µg BNT162b2 doses given ~21 days (d) apart.

The expansion cohorts are intended to provide a more in-depth characterization of the adaptive immune responses induced by BNT162b2, associated vaccine safety, and the impact of factors such as subject disposition and dosing posology on humoral and cell-mediated immunity. These cohorts will extend the safety data of BNT162b2 to a broader trial population and thus closer to the vaccine target population.



The planned dose of BNT162b2, two 30  $\mu$ g BNT162b2 doses given 21 d apart, is the same regimen that has already been tested in the dose escalation phase of this trial and in more than 25,000 trial subjects (status 20 JAN 2021), including those with acute and chronic illnesses, in the ongoing global Phase I/II/III trial BNT162-02/C4591001 (NCT04368728). As such, all trial subjects in the three expansion cohorts can be treated in parallel.

For Cohort 13, the interval between the trial subjects for the prime and boost immunizations will be at least 30 min. For Cohorts 11 and 12, the interval between the trial subjects will be at least 15 min for the prime immunizations and at least 5 min for boost immunizations.

The three expansion cohorts (with comparable numbers of male and female subjects for each of the defined age groups, see the section Population below) are as follows:

- Cohort 11: Alternative posology cohort with 30 healthy adults who will receive BNT162b2 using one 3 μg prime dose and one 30 μg boost dose of BNT162b2 given approximately 21 d apart (P/B regimen).
- Cohort 12: Adaptive immune response cohort (including safety and long term immune response) with 90 healthy adults who will receive two 30 μg BNT162b2 doses given approximately 21 d apart (P/B regimen).

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


 Cohort 13: Population expansion cohort (including safety and long term immune response) with 30 immunocompromised adults who will receive of two 30 μg BNT162b2 doses given approximately 21 d apart (P/B regimen).

For the scientific rationale for the expansion cohorts, see Section 4.2.

All trial site visits for subjects in the expansion cohorts will be conducted on an outpatient basis, with the clinical judgment of the investigator determining whether a period of observation beyond that required for completion of study procedures is required, on a case by case basis. Standard measures to avoid cross-contamination of immunocompromised individuals with high risk pathogens should be followed for 24 months after the primary immunization.

The European Medicines Agency (EMA) approval of a third dose of Comirnaty® has impacted the planned 2-year follow-up for Cohorts 11 to 13, with the subjects in this trial having the option to receive non-trial SARS-CoV-2 vaccinations (e.g., an authorized Comirnaty® vaccine within another BNT trial or within the government vaccination program).

### Biomarker (in-depth B cell immunity to SARS-CoV-2) Cohort 14:

Protocol amendment 8.0 implements an additional cohort (Cohort 14) comprising an additional 20 healthy subjects aged from 18 to 85 years receiving BNT162b2 only. Two 30 µg BNT162b2 doses will be given approximately 21 d apart (P/B regimen).

Cohort 14 is intended to provide for additional characterization of B cell immune responses induced by BNT162b2. The planned dose of BNT162b2, two 30 µg BNT162b2 doses given 21 d apart, is the same regimen that has already been tested in the dose escalation phase of this trial and in more than 25,000 trial subjects (status 20 JAN 2021) in the ongoing global Phase I/II/III trial BNT162-02/C4591001 (NCT04368728).

For the scientific rationale for Cohort 14, see Section 4.2.

### Part B

Due to changes in the overall clinical development plan, Part B will no longer be conducted.


Table 1: Dose ranging: vaccine dose regimens for younger adults aged 18 to 55 years in Part A (Cohorts 1 to 7)

| | | | Part A – Cohort numbers & dose (μg) (12 subjects per cohort) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Vaccine /<br>mRNA type | Vaccine-encoded antigen | Vaccine IM<br>dosing regimen | 1<br>Starting<br>dose | 2 | 3<br>De-escalation<br>dose | 4 | 5<br>Optional de-<br>escalation dose | 6 | 7 |
| BNT162a1 / | RBD of the SARS-CoV-2 | Prime: Day 1 | 1Α | 2Α | 3Α | 4Α <sup>a</sup> | 5Α | 6Α | |
| uRNA | S protein | Boost: Day 22 | 3 μg <sup>b</sup> | 0.6 μg <sup>a</sup> | 0.1 μg | 2 μg <sup>e</sup> | 0.3 μg | 1 μg | |
| BNT162b1 / | RBD of the SARS-CoV-2 | Prime: Day 1 | 1B | 2B | 3Β | 4Β | 5Β | 6B | 7Β |
| modRNA | S protein | Boost: Day 22 | 10 μg | 30 μg | 1 μg | 60 μg <sup>d</sup> | 50 μg | 3 µg | 20 μg |
| BNT162b2 / | Modified version of the full length SARS-CoV-2 S protein | Prime: Day 1 | 1C | 2C | 3C | 4C <sup>a</sup> | 5C <sup>a</sup> | 6C <sup>a</sup> | 7С <sup>а</sup> |
| modRNA | | Boost: Day 22 | 10 μg | 30 μg | 1 μg | 60 μg <sup>d</sup> | 20 μg | 3 µg | 50 µg |
| BNT162c2 /<br>saRNA | Modified version of the full length SARS-CoV-2 S protein | Prime only: Day 1 | 1D<br>0.1 μg | 2D<br>0.3 μg | 3D<br>0.1 µg to <3 µg <sup>c</sup> | 4D<br>1 μg | 5D <sup>a</sup><br>0.6 μg | 6D <sup>a</sup><br>3 μg <sup>d</sup> | |
| BNT162c2 / | Modified version of the full length SARS-CoV-2 S protein | Prime: Day 1 | 1Ε | 2E | 3Ε | 4E <sup>a</sup> | 5Ε | 6Ε | 7Ε |
| saRNA | | Boost: Day 22 | 0.1 μg | 0.3 μg | 1 μg | 5-10 μg <sup>c, d</sup> | 0.6 μg | 3 μg | 5-10 μg <sup>c, d</sup> |

a) All dose escalation doses used must be judged acceptable by the Safety Review Committee (SRC) before use.

Note: Currently, dosing with BNT162a1 has been deferred. Dosing may be resumed if disease prevention data for the other vaccine candidates suggest the need for additional vaccine candidates.

b) Status 08 JUN 2020: This cohort was set on hold by the SRC after 6 subjects had been received their Day 1 dose, furthermore the SRC decided not to perform Day 22 dosing for these 6 subjects. Due to this hold, the starting dose is also the maximum dose.

c) Specific doses to be defined, but in the range given. Already given doses will not be repeated.

d) The planned maximum doses per vaccine candidate.

e) Dosing with this vaccine variant has been put on hold. Dosing may be resumed if disease prevention data for the other vaccine candidates suggest the need for additional vaccine candidates.

IM = intramuscular; RBD = Receptor Binding Domain; S protein = SARS-CoV-2 spike protein; tbd = to be defined.


Table 2: Dose ranging: vaccine dose regimens for older adults aged 56 to 85 years in Part A (Cohorts 8 to 10)

| | | Vaccine IM dosing | Part A – Cohort numbe | ers & dose (µg) (12 sub | jects per cohort) <sup>a</sup> |
|---|---|---|---|---|---|
| Vaccine / mRNA type | Vaccine-encoded antigen | regimen | 8<br>Older adults | 9<br>Older adults | 10<br>Older adults |
| BNT162b1 / modRNA | RBD of the SARS-CoV-2 S protein | Prime: Day 1<br>Boost: Day 22 | 8B<br>10 µg | 9Β <sup>a</sup><br>20 μg | 10B <sup>a</sup><br>30 µg |
| BNT162b2 / modRNA | Modified version of the full length SARS-CoV-2 S protein | Prime: Day 1<br>Boost: Day 22 | 8С<br>10 µg | 9C <sup>a</sup><br>20 μg | 10C <sup>a</sup><br>30 μg |

a) All dose escalation doses used must be judged acceptable by the Safety Review Committee (SRC) before use.

Note: The doses planned in this trial for older adults (i.e., adults aged between 56 and 85 years) reflect clinical data from the ongoing BNT162-01 and BNT162-02 trials with the vaccine candidates BNT162b1 and BNT162b2 in younger adults (aged between 18 and 55 years) and elderly (adults aged between 65 and 85 years). For details, see the BNT162 IB.

#### BNT162b1:

- BNT162b1 P/B doses of 1, 10, 30, and 50 µg showed acceptable tolerability in younger adults.
- Based on the tolerability profile after the prime dose at 60 μg (BNT162-01 trial) and 100 μg (BNT162-02 trial), the respective boost doses were not administered.
- BNT162b1 P/B doses of 10, 20, and 30 μg showed acceptable tolerability in elderly adults. This tolerability appears to be better than seen in younger adults at the same doses. BNT162b2:
- BNT162b2 P/B doses of 1, 10, and 30 µg showed acceptable tolerability in younger adults.
- BNT162b2 P/B doses of 10, 20, and 30 µg showed acceptable tolerability in elderly adults. This tolerability appears to be better than seen in younger adults at the same doses.

Based on the tolerability data summarized above, and the implemented safety measures (sentinel/staggered subject dosing, post-dose observations period, wellbeing questioning, etc.) as described in the section Risk assessment, the planned doses in older subjects in this trial are expected to show acceptable tolerability.

Based on the available immunogenicity data after dosing with BNT162b1 and BNT162b2 in younger adults in the BNT162-02 trial (see the BNT162 IB), the doses planned in this trial in older subjects are expected to show lower but measurable immunogenicity than in younger adults.

Altogether, the doses planned in older subjects in this trial are considered adequate to support the trial objectives and to pose an acceptable risk to trial subjects.

IM = intramuscular; RBD = Receptor Binding Domain; S protein = SARS-CoV-2 spike protein.


Table 3: Expansion cohorts for BNT162b2 (ages 18 to 85 years) in Part A (Cohorts 11 to 13)

| Vaccine / mRNA type V | | | Part A – Coho | rt numbers & dose (μg) (number | subjects per cohort) |
|---|---|---|---|---|---|
| Vaccine / mRNA type | Vaccine-encoded antigen Vaccine IM dosing regimen Modified version of the full length SARS-CoV-2 S protein Vaccine IM dosing regimen | 11C<br>(N = 30)<br>Healthy adults<br>(Alternative posology) | 12C<br>(N = 90)<br>Healthy adults<br>(Adaptive immune response<br>cohort) | 13C (N = 30) Immunocompromised but otherwise healthy adults (Population expansion cohort) | |
| I BNI 16202 / MODRNA I | | • | 3 µg<br>30 µg | 30 µg<br>30 µg | 30 µg<br>30 µg |

IM = intramuscular; N = number of subjects; S protein = SARS-CoV-2 sp ke protein.

Table 4: Cohort 14 for BNT162b2 (ages 18 to 85 years) in Part A

| | | | Part A – Cohort number & dose (μg) (number of subjects) |
|---|---|---|---|
| Vaccine / mRNA type | Vaccine-encoded antigen | Vaccine IM dosing regimen | 14<br>(N = 20)<br>Healthy adults<br>(B cell and plasma cell immune responses) |
| BNT162b2 / modRNA | Modified version of the full length SARS-CoV-2 S protein | Prime: Day 1<br>Boost: Day 22 | 30 µg<br>30 µg |

IM = intramuscular; N = number of subjects; S protein = SARS-CoV-2 sp ke protein.


#### **Trial duration**

In total, the planned trial duration (i.e., the sum of the screening, treatment, and follow-up phases) for subjects is expected to be approximately 223 d for Cohorts 1 to 10 and 14, and 760 d for Cohorts 11 to 13.

For logistical reasons, investigation of the different vaccines may not be able to start at the same time.

### **Population**

### Dose ranging Cohorts (Cohorts 1 to 10)

 Healthy adults aged 18 to 55 years (Cohorts 1 to 7; younger adults) or aged 56 to 85 years (Cohorts 8 to 10; older adults). Subjects aged 56 to 85 years must be enrolled such that at least 6 subjects per cohort are aged 65 to 85 years (i.e., are elderly). For each vaccine, 12 subjects are required for each of the dose ranging cohorts.

### Expansion cohorts (Cohorts 11 to 13)

- Cohort 11 Alternative posology cohort: 30 healthy adults aged 18 to 85 years with comparable numbers of male and female subjects for each of the following age groups: 18 to 55 years, 56 to 85 years (15 per age group).
- Cohort 12 Adaptive immune response cohort: 90 healthy adults, with comparable numbers of male and female subjects for each of the following age groups: 18 to 55 years, 56 to 64 years, and 65 to 85 years (30 per age group).
- Cohort 13 Population expansion cohort: 30 immunocompromised adults aged 18 to 85 years with comparable numbers of male and female subjects for each of the following age groups: 18 to 55 years, 56 to 85 years (and approximately comparable numbers within each age group).

#### Biomarker (B cell and plasma cell immunity directed to SARS-CoV-2) cohort (Cohort 14)

 20 healthy adults aged 18 to 85 years, ideally with 10 male and 10 female subjects and approximately comparable numbers of subjects for each of the following age groups: 18 to 55 years, 56 to 85 years.

Table 5: Overview of the total number of subjects for each vaccine in Part A

| Vaccine / mRNA type | Vaccine dosing regimen | Maximum number of subjects (assuming all cohorts planned in Table 1, Table 2, Table 3, and Table 4 are performed) |
|---|---|---|
| BNT162a1 / uRNA | Prime/Boost | 72 (6 cohorts) |
| BNT162b1 / modRNA | Prime/Boost | 120 (10 cohorts) |
| BNT162b2 / modRNA | Prime/Boost | 290 (14 cohorts) |
| BNT162c2 / saRNA | Prime only | 72 (6 cohorts) |
| BNT162c2 / saRNA | Prime/Boost | 84 (7 cohorts) |

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### Key inclusion criteria

Volunteers are only eligible to be enrolled in the trial if they meet the following criteria:

For younger adult cohorts, volunteers must be aged 18 to 55 years, have a BMI over 19 kg/m<sup>2</sup> and under 30 kg/m<sup>2</sup>, and weigh at least 50 kg at Visit 0.
 OR

For older adult cohorts, volunteers must be aged 56 to 85 years, have a BMI over 19 kg/m<sup>2</sup> and under 30 kg/m<sup>2</sup>, and weigh at least 50 kg at Visit 0. OR

For the immunocompromised adult cohort (Cohort 13), volunteers must be aged 18 to 85 years, have a BMI over 19 kg/m<sup>2</sup> and under 30 kg/m<sup>2</sup>, and weigh at least 50 kg at Visit 0.

 They must be healthy, in the clinical judgment of the investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs (systolic/diastolic blood pressure, pulse rate, body temperature, respiratory rate), and clinical laboratory tests (blood chemistry, hematology, and urine chemistry) at Visit 0.

Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks (wks) before enrollment, can be included.

For the immunocompromised cohort (Cohort 13); volunteers who have previously received solid organ transplant, or peripheral blood stem cell transplantation ≥6 months after transplantation, or individuals with human immunodeficiency virus (HIV) infection with a CD4+ T-cell count of ≥200 x 10<sup>6</sup>/L at Visit 0. Individuals with lower T-cell counts will be excluded from the trial on the basis that this represents a significant medical complication. In the clinical judgment of the investigator, volunteers must be immunocompromised but otherwise healthy. After consultation with the Medical Monitor, this may include individuals receiving immunosuppressant therapy due to another confounding disease at least 2 wks prior to enrollment and/or at least 6 wks following immunization with BNT162b2, and/or individuals with immunosuppressive treatment of an autoimmune disease if the disease is stable.

 Women of childbearing potential (WOCBP) must have a negative beta-human chorionic gonadotropin urine test at Visit 0 and Visit 1. Women that are postmenopausal or permanently sterilized will be considered as not having reproductive potential.

### Key exclusion criteria

Volunteers are excluded from the trial if they present any of the following criteria:

 Have had any acute illness, as determined by the investigator, with or without fever, within 72 h prior to any immunization. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the investigator, the residual symptoms will not compromise their wellbeing if they

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.

- Have a known allergy, hypersensitivity, or intolerance to the planned investigational medicinal product (IMP) including any excipients of the IMP.
- Had any medical condition or any major surgery (e.g., requiring general anesthesia) within the past 5 years which, in the opinion of the investigator, could compromise their wellbeing if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments. See the inclusion criteria for non-excluded medical conditions for Cohort 13.
- Have any surgery planned during the trial, starting after Visit 0 and continuously until at least 90 d after receiving the last immunization.
- Had any chronic use (more than 21 continuous days) of any systemic medications, including immunosuppressants or other immune-modifying drugs (except for Cohort 13) within the 6 months prior to Visit 0, unless in the opinion of the investigator the medication would not prevent, limit, or confound the protocol-specified assessments or could compromise subject safety.

Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 wks before enrollment, can be included.

- Regular receipt of inhaled/nebulized corticosteroids (except for Cohort 13).
- Had any vaccination within the 28 d prior to Visit 0.
- Had administration of any immunoglobulins and/or any blood products within the 3 months prior to Visit 0.
- Had administration of another IMP including vaccines within 60 d or 5 half-lives (whichever is longer), prior to Visit 0.
- Have a known history of active or ongoing hepatitis B or hepatitis C infection; or except for Cohort 13: HIV-1 or HIV-2 infection within the 30 d prior to Visit 0.
- Have a positive PCR-based test for SARS-CoV-2 within the 30 d prior to Visit 1.
- Previously participated in an investigational trial involving lipid nanoparticles.
- Have a history (within the past 5 years) of substance abuse or known medical, psychological, or social conditions which, in the opinion of the investigator, could compromise their wellbeing if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
- Have a history of hypersensitivity or serious reactions to previous vaccinations.
- Have a history of Guillain-Barré syndrome within 6 wks following a previous vaccination.
- Have a history of narcolepsy.

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- (Except for Cohort 13) Have a history of or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination at Visit 0.
- Have symptoms of the Coronavirus Disease 2019 (COVID-19), e.g., respiratory symptoms, fever, cough, shortness of breath and breathing difficulties.
- Have had contact with persons diagnosed with COVID-19 or who tested positive for SARS-CoV-2 by any diagnostic test within the 30 d prior to Visit 1.
- Are soldiers, volunteers in detention, CRO or sponsor staff or their family members.
- For older volunteers and for Cohort 13 only: Have a condition known to put them at high risk for severe COVID-19, including those with any of the following risk factors:
  - Uncontrolled hypertension.
  - Diabetes mellitus (HbA1c >8.5% ≥3 months, according to the medical history reported by the subject).
  - Chronic obstructive pulmonary disease.
  - Asthma.
  - Chronic liver disease.
  - Known Stage 3 or worse chronic kidney disease (glomerular filtration rate [GFR] of <60 mL/min/1.73 m²); Except for post-renal transplant patients who should have (estimated) GFR ≥40 mL/min/1.73 m².
  - Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies.
  - Sickle cell disease.
  - Cancer (except for Cohort 13).
  - Are immune compromised due to stem cell or organ-transplantation with significant medical complications such as acute or chronic graft rejection or graft versus host disease requiring intensive immunosuppressive treatment, transplant failure, or infectious complications or other conditions that would be considered a contraindication for vaccination.
  - Are immune compromised due to HIV infection with a CD4<sup>+</sup> count of <200 x 10<sup>6</sup>/L at screening (Visit 0) or significant medical complications such as opportunistic infections, malignant complications (e.g., lymphoma, Kaposi sarcoma), other organ manifestations consistent with advanced acquired immunodeficiency syndrome (AIDS) or other conditions that would be considered a contraindication for vaccination.
  - Resident in a long term facility.
  - Current vaping or smoking (occasional smoking is acceptable).
  - History of chronic smoking within the prior year.

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### Trial treatments (BNT162 vaccines)

Name: BNT162 vaccines - Antiviral RNA vaccines for active immunization against COVID-19

Type: RNA-LNP vaccines utilizing different BioNTech RNA formats, i.e., uRNA (product code

BNT162a1), modRNA (two variants, product codes BNT162b1 and BNT162b2),

saRNA (product code BNT162c2)

Dosage levels: Part A cohorts:

See Table 1, Table 2, Table 3, and Table 4. The planned dose per vaccine candidate will not exceed the pre-defined maximum dose (see Table 1 and Table 2). The planned dose per vaccine candidate will not exceed the listed pre-defined maximum doses.

Dosage

One injection or two injections 21 d apart. Injection volumes will be up to 1.5 mL.

frequency:

Intramuscular (IM); upper arm, musculus deltoideus. For the P/B regimens the same

Administration route:

arm may be used for both immunizations. The non-dominant arm is preferred.

#### **Statistics**

The final analysis will be performed once all subjects have completed the end of treatment (EoT as defined in Section 1.3). An analysis update will be performed once all subjects will have completed the last planned visit. No formal interim statistical analysis will be performed. However, preliminary analyses based on all data collected until a pre-defined data cut-off date (snapshot analyses) may be performed for each cohort once subjects within a cohort will have been followed up for at least 7 d following each dose.

### **Data Monitoring Committee (DMC)/SRC**

A DMC is not planned. A SRC is planned.


### 1.2 Schema (graphical representation of the trial)

For a graphical depiction of the cohorts in Part A, see Figure 1. For logistical reasons, investigation of the different vaccines may not be able to start at the same time. Should this happen, the expected overall trial duration may be extended.

Dose ranging cohort schema for BNT162a1, BNT162b1, BNT162b2, and BNT162c2 (P/B) c

Cohorts 1 to 7 with younger adults



#### Cohorts 8 to 10 with older adults



- a) The data assessed by the SRC for progressing comprises 48 h data for 6 subjects.
- b) Subjects will be dosed using a sentinel dosing/subject (2-4-6) staggering process unless the planned dose is the same or lower than previously found to show acceptable tolerability (in which case, all subjects may be dosed on one day).
- c) For the dose regimens, see Table 1 and Table 2.


### Dose ranging cohort schema for BNT162c2 (SD) b



- a) The data assessed by the SRC for progressing comprises 48 h data for 6 subjects.
- b) For the dose regimens, see Table 1.

### Expansion cohorts for BNT162b2 - Cohorts 11 to 13 a



a) For the dose regimens, see Table 3.

### Biomarker (B cell and plasma cell immunity) cohort for BNT162b2 - Cohort 14 a

a) For the dose regimen, see Table 4.

Figure 1: Graphical depiction of the dose-finding and expansion process in Part A

FIH = first-in-human; h = hour(s); SRC = Safety Review Committee.


### 1.3 Schedule of activities

Table 6: Schedule of trial procedures and assessments – BNT162a1, BNT162b1, BNT162b2, and BNT162c2 when tested P/B (excluding Cohorts 11 to 14)

| Procedure /<br>Assessment | Visit 0 | Visit 1<br>Pre-<br>dose | Visit 1<br>(Post-)<br>dosing | Visit 2<br>at<br>24±2 h | Phone<br>call at<br>48±2 h | Visit 3 | Visit 4<br>Pre-<br>dose | Visit 4<br>Dosing<br>& Post-<br>dose | Phone<br>call at<br>48±2 h | Visit 5 | Visit 5a | Visit 6 | Visit 7<br>(EoT<br>Visit) | Visit 8<br>(FU<br>Visit) | Visit 9<br>(FU<br>Visit) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day <sup>h</sup> | -30 to 0 | 1 | 1 | 2 | | 8 | 22 | 22 | | 29 | 36 <sup>q</sup> | 43 | 50 <sup>r</sup> | 85 | 184 |
| Days to last dose h | | 0 | 0 | | | 7 | 21 | 0 | | 7 | 14 | 21 | 28 | 63 | 162 |
| Informed consent | Х | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | х | X<br>(review) | | | | | | | | | | | | | |
| Medical history | х | X<br>(update) | | | | | | | | | | | | | |
| Physical examination incl. height | х | X a | | X a | | X a | X a | | | X a | | X a | X a | | |
| Vital signs, body<br>weight <sup>c</sup> | х | х | X b | х | | х | х | Χb | | х | | Х | х | Х | х |
| 12-lead ECG | Х | Х | | | | | | | | | | | | | |
| Urine pregnancy test for WOCBP | х | х | | | | | х | | | | | | | | |
| Urine drugs of abuse screen <sup>d</sup> | х | х | | | | | | | | | | | | | |
| Alcohol breath test | Х | Х | | | | | | | | | | | | | |
| Urine collection for clinical laboratory <sup>e</sup> | х | х | | х | | х | | | | х | | | х | | |
| Blood draw for clinical laboratory (15 mL) <sup>f</sup> | х | х | | х | | х | | | | х | | | х | | |
| Blood draw for viral screening <sup>g</sup> | X (5 mL) | | | | | | | | | | | | | | |

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| Procedure /<br>Assessment | Visit 0 | Visit 1<br>Pre-<br>dose | Visit 1<br>(Post-)<br>dosing | Visit 2<br>at<br>24±2 h | Phone<br>call at<br>48±2 h | Visit 3 | Visit 4<br>Pre-<br>dose | Visit 4<br>Dosing<br>& Post-<br>dose | Phone<br>call at<br>48±2 h | Visit 5 | Visit 5a | Visit 6 | Visit 7<br>(EoT<br>Visit) | Visit 8<br>(FU<br>Visit) | Visit 9<br>(FU<br>Visit) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day <sup>h</sup> | -30 to 0 | 1 | 1 | 2 | | 8 | 22 | 22 | | 29 | 36 <sup>q</sup> | 43 | 50 <sup>r</sup> | 85 | 184 |
| Days to last dose h | | 0 | 0 | | | 7 | 21 | 0 | | 7 | 14 | 21 | 28 | 63 | 162 |
| Blood draw for<br>SARS-CoV-2 testing <sup>k</sup> | X<br>(2.6 mL) | | | | | | | | | | | | | | |
| Oral swipe for<br>SARS-CoV-2 testing | | X <sup>m</sup> | | | | | | | | | | | | | |
| Allocation to IMP | | X | | | | | | | | | | | | | |
| Immunization | | | ΧI | | | | | X | | | | | | | |
| Blood draw for immunogenicity (10 mL) <sup>n</sup> | | X | | | | x | X | | | x | Х | x | х | х | x |
| Blood draw for HLA p | | | | | | | Х | (4 mL EDTA | A-blood) p | | | | | | |
| Blood draw for CMI<br>(100 mL) <sup>n, o</sup> | | Х | | | | | | | | х | | | | | |
| Blood draw for research n | | | | | | | | | | | | X<br>(≤100 mL) | | X<br>(≤50 mL) | X<br>(≤50 mL) |
| Subject hotline availability | Start | => | => | =^ | | => | => | => | | => | => | - | => | => | End |
| Issue subject diaries | | X | | X | | X | X | | | X | | X | X | | |
| Collect subject diaries | | | | Х | X | Х | Х | | | X | | Х | Х | X | |
| Record AEs since last visit | | X | | Х | | X | Х | | | х | X | Х | X | Χj | Χj |
| Local reaction<br>assessment/<br>systemic events | | | Χþ | Х | | х | Х | Хp | | х | | x | Х | | |
| Concomitant medication s | х | Х | | Х | | х | Х | | | X | | Х | Х | Х | Х |
| Subject wel being questioning | | | | | Χi | | | | Χ <sup>i</sup> | | | | | | |

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- a) Brief (symptom-directed) physical examination; no height measurement.
- b) At 1, 3, and 6 h (±15 min) after immunization.
- c) Vital signs: systolic/diastolic blood pressure, pulse rate, respiratory rate, and body temperature; body weight only at Visit 0.
- d) Urine screening for drugs of abuse (amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, tricyclic antidepressants).
- e) Dipstick urine analysis: glucose, bilirubin, ketone, specific gravity, blood, pH, protein, urobilinogen, nitrite, and leukocytes. Microscopic urinalysis: if warranted by dipstick results, urine sediment will be microscopically examined for the presence of red blood cells, white blood cells, casts, crystals, epithelial cells, and bacteria.
- f) Clinical laboratory tests: (Chemistry) alkaline phosphatase, creatinine, ferritin, C-reactive protein, albumin, alanine aminotransferase, amylase, aspartate aminotransferase, gamma glutamyl transpeptidase, total bilirubin, blood urea nitrogen, glucose, lipase, sodium, potassium, calcium; (Hematology) hemoglobin, hematocrit, red blood cell count, white blood cell count and differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count. Only in women who are not WOCBP (to confirm postmenopausal status): follicle stimulating hormone at Visit 0.
- g) Viral screening for human immunodeficiency virus (HIV) 1 or 2, hepatitis B, hepatitis C.
- h) Flexibility for visit days: Visit 3 Day 8±1 d; Visit 4 Day 22±2 d; Visit 5 Day 29±3 d; Visit 6 Day 43±4 d; Visit 7 Day 50±4 d; Visit 8 Day 85±7 d; Visit 9 Day 184±9 d.
- i) Only for the first 6 subjects per group. Questioning on and documentation of AEs as well as systemic and local reactions, the latter in case of upcoming dose decision meetings.
- j) Only IMP-related AEs and any SAEs except proven COVID-19 cases which have to be reported regardless on severity and relatedness to the trial drug until the last scheduled FU Visit as descr bed in Section 10.3.1.9.
- k) Blood draw for anti-SARS-CoV-2 antibodies.
- l) For Cohorts 1 and 8, immunization with at least 1 h intervals between subjects for the first 6 subjects and then with of at least 30 min intervals for the remaining 6 subjects. For all other cohorts and for all boost immunization, the intervals between subjects will be at least 30 min.
- m) Oral swipe for SARS-CoV-2 testing either on Day -1 or at the Visit 1 on Day 1.
- n) The timing of the listed "research" blood draw days may be adapted within the 200 mL maximum volume if justified by the collected data. Leftover blood after completion of the immunogenicity assessments may be used for additional analyses as described in Section 8.7 (Genetics) and/or Section 8.8 (Biomarkers).
- o) For subjects who have given consent, one aliquot of the blood sample drawn for analysis of CMI may be used for HLA typing to allow additional analysis of T-cell receptor repertoire and/or phenotypic characterization of T cells specific to vaccine-encoded antigens.
- p) If HLA typing using the blood sample collected with Lithium Heparin is not conclusive, EDTA-blood will be drawn for HLA testing.
- q) Only cohorts starting prime dosing after approval of protocol amendment 06.
- r) When entering the follow-up phase, i.e., after completing the EoT Visit, subjects are allowed to participate in other clinical trials not investigating COVID-19 vaccines or treatments.
- s) Record any medications that trial subjects receive during the trial in the CRF starting after Visit 0 and until the respective EoT Visit; record any vaccination, including SARS-CoV-2 vaccination, that subjects receive after the EoT Visit until the last FU Visit in the CRF.

#### Notes:

If the boost dose is not administered or if trial subjects permanently discontinue from IMP administration, subjects will complete all assessments listed in the SoA. The additional Visit 5a added by protocol amendment 06 will only apply for subjects who give consent.

AE = adverse event; CMI = cell-mediated immune testing; CRF = case report form; D or d = day; ECG = electrocardiogram; EDTA = ethylenediamine tetraacetic acid; EoT = end of treatment (Visit); FU = follow-up (visit); h = hour(s); HLA = human leukocyte antigen; Day 0 = one day before Day 1; IMP = investigational medicinal product; min = minute(s); SAE = serious adverse event; SARS-CoV-2 = the virus leading to COVID-19; SoA = Schedule of Activities; WOCBP = women of childbearing potential.


Table 7: Schedule of trial procedures and assessments – BNT162c2 (SD)

| Procedure/Assessment | Visit 0 | Visit 1<br>Pre-dose | Visit 1<br>Dosing &<br>Post-dose | Visit 2<br>at 24±2 h | Phone<br>call at<br>48±2 h | Visit 3 | Visit 4 | Visit 5 | Visit 6<br>(EoT Visit) | Visit 7<br>(FU Visit) | Visit 8<br>(FU Visit) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Day <sup>a</sup> | -30 to 0 | 1 | 1 | 2 | | 8 | 22 | 29 | 43 <sup>q</sup> | 85 | 184 |
| Informed consent | Х | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X (review) | | | | | | | | | |
| Medical history | X | X (update) | | | | | | | | | |
| Physical examination incl. height | X | X b | | ХÞ | | ХÞ | ХÞ | ΧÞ | ХÞ | | |
| Vital signs, body weight <sup>c</sup> | Х | Х | X q | X | | X | X | X | X | | |
| 12-lead ECG | X | Х | | | | | | | | | |
| Urine pregnancy test (for WOCBP) | X | Х | | | | | X | | | | |
| Urine drugs of abuse screen <sup>e</sup> | X | X | | | | | | | | | |
| Alcohol breath test | X | Х | | | | | | | | | |
| Urine for clinical laboratory <sup>f</sup> | Х | Х | | Х | | Х | | X | X | | |
| Blood draw for clinical laboratory <sup>g</sup> | X (15 mL) | X (15 mL) | | X (15 mL) | | X (15 mL) | | X (15 mL) | X (15 mL) | | |
| Blood draw for viral screening h | X (5 mL) | | | | | | | | | | |
| Blood draw for SARS-CoV-2 testing <sup>i</sup> | X<br>(2.6 mL) | | | | | | | | | | |
| Oral swipe for SARS-CoV-2 testing <sup>j</sup> | | Х | | | | | | | | | |
| Allocation to IMP | | Х | | | | | | | | | |
| Immunization k | | | X | | | | | | | | |
| Blood draw for immunogenicity | | X (10 mL) | | | | X (10 mL) | X (10 mL) | X (10 mL) | X (10 mL) | X (10 mL) | X (10 mL) |
| Blood draw for HLA testing <sup>p</sup> | | | | | X (4 mL | EDTA-blood) | | | | | |
| Blood draw for CMI testing I, m | | X (100 mL) | | | _ | | | X (100 mL) | | | |
| Blood draws for research | | | _ | | | | | | X (≤100 mL) | X (≤50 mL) | X (≤50 mL) |
| Subject hotline availability | Start | => | => | => | | => | => | => | => | => | End |
| Issue subject diaries | | Х | | X | | X | X | X | | | |

Procedure/Assessment

Collect subject diaries

systemic events

Record AEs since last visit

Local reaction assessment/

Concomitant medication r

Subject wel being questioning

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01

Phone

call at

48±2 h

Х

χo

Visit 3

8

Χ

Χ

Χ

Χ

Visit 4

22

Х

Χ

Х

Χ

Visit 5

29

Χ

X

Χ

Χ

Χ

Visit 2

at 24±2 h

2

Χ

Χ

Х

Χ

| Visit 6 (FU Visit) (FU Visit) 43 q 85 184 X | | |
|-----------------------------------------------|-----|-----|
| 43 <sup>q</sup> | 85 | 184 |
| Χ | | |
| Х | X n | X n |

Χ

Х


Version: 13.0

a) Flexibility for visit days: Visit 3 Day 8±1 d; Visit 4 Day 22±2 d; Visit 5 Day 29±3 d; Visit 6 Day 43±4 d; Visit 7 Day 85±7 d; Visit 8 Day 184±9 d.

Visit 1

Dosing &

Post-dose

1

X d

b) Brief (symptom-directed) physical examination; no height measurement.

Day <sup>a</sup>

c) Vital signs: systolic/diastolic blood pressure, pulse rate, respiratory rate, and body temperature; body weight only Visit 0.

Visit 1

Pre-dose

1

Χ

Х

- d) At 1, 3, and 6 h (±15 min) after immunization.
- e) Urine screening for drugs of abuse (amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, tricyclic antidepressants).
- f) Dipstick urine analysis: glucose, bilirubin, ketone, specific gravity, blood, pH, protein, urobilinogen, nitrite, and leukocytes. Microscopic urinalysis: if warranted by dipstick results, urine sediment will be microscopically examined for the presence of red blood cells, white blood cells, casts, crystals, epithelial cells, and bacteria.
- g) Clinical laboratory tests: (Chemistry) alkaline phosphatase, creatinine, ferritin, C-reactive protein, albumin, alanine aminotransferase, amylase, aspartate aminotransferase, gamma glutamyl transpeptidase, total bilirubin, blood urea nitrogen, glucose, lipase, sodium, potassium, calcium; (Hematology) hemoglobin, hematocrit, red blood cell count, white blood cell count and differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count. Only in women who are not WOCBP (to confirm postmenopausal status): follicle stimulating hormone at Visit 0.
- h) Viral screening for human immunodeficiency virus (HIV) 1 or 2, hepatitis B, hepatitis C.

Visit 0

-30 to 0

Χ

- i) Blood draw for anti-SARS-CoV-2 antibodies.
- Oral swipe for SARS-CoV-2 testing either on Day -1 or at the Visit 1 on Day 1.
- k) For Cohort 1, immunization with at least 1 h intervals between subjects for the first 6 subjects and then with at least 30 min intervals for the remaining 6 subjects. For all other cohorts, immunization with 30 min intervals between subjects.
- The listed blood draw days may be adapted if justified by the collected data. Leftover blood after completion of the immunogenicity assessments may be used for additional analyses as described in Section 8.7 (Genetics) and/or Section 8.8 (Biomarkers).
- m) For subjects who have given consent, one aliquot of the blood sample drawn for analysis of CMI may be used for human leukocyte antigen typing to allow additional analysis of T-cell receptor repertoire and/or phenotypic characterization of T cells specific to vaccine-encoded antigens.
- n) Only IMP-related AEs and any SAEs except proven COVID-19 cases which have to be reported regardless on severity and relatedness to the trial drug until the last scheduled FU Visit as descr bed in Section 10.3.1.9.
- o) Only for the first 6 subjects per group. Questioning on and documentation of AEs as well as systemic and local reactions, the latter in case of upcoming dose decision meetings.
- p) If HLA typing using the blood sample collected with Lithium Heparin is not conclusive. EDTA-blood will be drawn for HLA testing.
- d) When entering the follow-up phase, i.e., after completing the EoT Visit, subjects are allowed to participate in other clinical trials not investigating COVID-19 vaccines or treatments.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


r) Record any medications that trial subjects receive during the trial in the CRF starting after Visit 0 and until the respective EoT Visit; record any vaccination, including SARS-CoV-2 vaccination, that subjects receive after the EoT Visit until the last FU Visit in the CRF.

AE = adverse event; CMI = cell-mediated immune testing; CRF = case report form; d = day; ECG = electrocardiogram; EDTA = ethylenediamine tetraacetic acid; EoT = end of treatment (Visit); FU = follow-up (visit); h = hour(s); HLA = human leukocyte antigen; IMP = investigational medicinal product; min = minute(s); SAE = serious adverse event; SARS-CoV-2 = the virus leading to COVID-19; WOCBP = women of childbearing potential.


Table 8: Schedule of trial procedures and assessments – Cohorts 11 to 13 (Expansion cohorts only)

| Procedure /<br>Assessment | Visit 0 | Visit 1<br>Pre-dose | Visit 1<br>(Post-)<br>dosing | Visit 2 | Visit 3 | Visit 4<br>Pre-<br>dose | Visit 4<br>(Post-)<br>dosing | Visit 5 | Visit 5a | Visit 6 | Visit 7<br>(EoT<br>Visit) | Visit 8<br>(FU<br>Visit) | Visit 9<br>(FU<br>Visit) | Visit 10<br>(FU<br>Visit) <sup>s</sup> | Visit 11<br>(FU<br>Visit) <sup>s</sup> | Visit 12<br>(FU<br>Visit) <sup>s</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day <sup>h</sup> | -30 to 0 | 1 | 1 | 2 | 8 | 22 | 22 | 29 | 36 | 43 | 50 <sup>q</sup> | 85 | 184 | 365 | 547 | 730 |
| Days to last dose h | | 0 | 0 | 1 | 7 | 21 | 0 | 7 | 14 | 21 | 28 | 63 | 162 | 343 | 525 | 708 |
| Informed consent | X | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | х | X (review) | | | | | | | | | | | | | | |
| Medical history | X | X (update) | | | | | | | | | | | | | | |
| Physical exam. incl. height | х | X <sup>a</sup> | | Χª | X a | X a | | Χa | | X a | X a | | | | | |
| Vital signs, body<br>weight <sup>c</sup> | х | Х | X b | X | х | х | Χþ | X | | Х | х | Х | X | | | |
| 12-lead ECG | Х | Х | | | | | | | | | | | | | | |
| Urine pregnancy test for WOCBP | х | Х | | | | х | | | | | | | | | | |
| Urine drugs of abuse screen <sup>d</sup> | х | Х | | | | | | | | | | | | | | |
| Alcohol breath test | Х | Х | | | | | | | | | | | | | | |
| Urine collection for clinical laboratory <sup>e</sup> | х | Х | | X | х | | | X | | | х | | | | | |
| Blood draw for clin.<br>lab. (15 mL) <sup>f</sup> | х | Х | | x | х | | | X | | | х | | | | | |
| Blood draw for viral screening <sup>g</sup> | X<br>(5 mL) | | | | | | | | | | | | | | | |
| Blood draw for SARS-<br>CoV-2 testing (2.6 mL) k | х | | | | | | | | | | | | | | | |
| Oral swipe for<br>SARS-CoV-2 testing | | X <sup>m</sup> | | | | | | | | | | | | | | |
| Allocation to IMP | | X | | | | | | | | | | | | | | |

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| Procedure /<br>Assessment | Visit 0 | Visit 1<br>Pre-dose | Visit 1<br>(Post-)<br>dosing | Visit 2 | Visit 3 | Visit 4<br>Pre-<br>dose | Visit 4<br>(Post-)<br>dosing | Visit 5 | Visit 5a | Visit 6 | Visit 7<br>(EoT<br>Visit) | Visit 8<br>(FU<br>Visit) | Visit 9<br>(FU<br>Visit) | Visit 10<br>(FU<br>Visit) <sup>s</sup> | Visit 11<br>(FU<br>Visit) <sup>s</sup> | Visit 12<br>(FU<br>Visit) <sup>s</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day <sup>h</sup> | -30 to 0 | 1 | 1 | 2 | 8 | 22 | 22 | 29 | 36 | 43 | 50 <sup>q</sup> | 85 | 184 | 365 | 547 | 730 |
| Days to last dose h | | 0 | 0 | 1 | 7 | 21 | 0 | 7 | 14 | 21 | 28 | 63 | 162 | 343 | 525 | 708 |
| Immunization | | | ΧI | | | | Х | | | | | | | | | |
| Blood draw for immunogenicity <sup>n</sup> | | X<br>(10 mL) | | | X<br>(10 mL) | X<br>(10 mL) | | X<br>(10 mL) | X<br>(10 mL) | X<br>(10 mL) | X<br>(10 mL) | X<br>(10 mL) | X<br>(10 mL) | X<br>(10 mL) | X<br>(10 mL) | X<br>(10 mL) |
| Blood draw for HLA p | | | | | | X (4 mL E | DTA-blood) | | | | | | | | | |
| Blood draw for CMI<br>(100 mL) <sup>n, o</sup> | | Х | | | | | | х | | | | | х | х | Х | х |
| Blood draw for research <sup>n</sup> | | | | | X<br>(≤25 mL) | X<br>(≤25 mL) | | | | X<br>(≤100 mL) | | X<br>(≤50 mL) | | | | |
| Subject hotline availability | Start | => | => | => | => | => | => | => | => | => | => | => | => | => | => | End |
| Issue subject diaries | | X | | X | X | X | | X | | X | X | | | | | |
| Collect subject diaries | | | | X | X | X | | X | | X | X | X | | | | |
| Record AEs since last visit | | Х | | X | X | Х | | X | | X | х | Χj | Χj | Χj | Χj | <b>X</b> j |
| Local reaction<br>assessment/systemic<br>events | | | Хp | x | х | x | X p | x | | x | х | | | | | |
| Concomitant medication r | х | Х | | Х | Х | X | | х | | Х | х | Х | х | х | X | х |
| Subject wel being questioning by phone | | | | | | | X<br>At 24 h±2 h<br>post-second<br>dose | | | | | | | | | |
| Blood draw for CD <sup>4+</sup><br>T-cell count <sup>i</sup> | X<br>(3 mL) | | | | | | | | | | | | | | | |

a) Brief (symptom-directed) physical examination; no height measurement.

b) At 1, 3, and 6 h (±15 min) after immunization.

c) Vital signs: systolic/diastolic blood pressure, pulse rate, respiratory rate, and body temperature; body weight only at Visit 0.

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- d) Urine screening for drugs of abuse (amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, tricyclic antidepressants).
- e) Dipstick urine analysis: glucose, bilirubin, ketone, specific gravity, blood, pH, protein, urobilinogen, nitrite, and leukocytes. Microscopic urinalysis: if warranted by dipstick results, urine sediment will be microscopically examined for the presence of red blood cells, white blood cells, casts, crystals, epithelial cells, and bacteria.
- f) Clinical laboratory tests: (Chemistry) alkaline phosphatase, creatinine, ferritin, C-reactive protein, albumin, alanine aminotransferase, amylase, aspartate aminotransferase, gamma glutamyl transpeptidase, total bilirubin, blood urea nitrogen, glucose, lipase, sodium, potassium, calcium; (Hematology) hemoglobin, hematocrit, red blood cell count, white blood cell count and differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count. Only in women who are not WOCBP (to confirm postmenopausal status): follicle stimulating hormone at Visit 0.
- g) Viral screening for human immunodeficiency virus (HIV) 1 or 2, hepatitis B, hepatitis C.
- h) Flexibility for visit days: Visit 3 Day 8±1 d; Visit 4 Day 22±2 d; Visit 5 Day 29±3 d; Visit 5a Day 36±3 d; Visit 6 Day 43±4 d; Visit 7 Day 50±4 d; Visit 8 Day 85±7 d; Visit 9 Day 184±9 d; Visit 10 Day 365±14 d; Visit 11 Day 547±14 d; Visit 12 Day 730±14 d.
- i) Only for HIV-positive subjects (done locally).
- i) Visits 8 and 9, only IMP-related AEs and any SAEs. Visits 10, 11, and 12, only any SAEs except proven COVID-19 cases which have to be reported regardless on severity and relatedness to the trial drug until the last scheduled FU Visit as described in Section 10.3.1.9. For subjects who receive non-trial SARS-CoV-2 vaccinations, the AEs expected to be captured after these vaccinations are within the frame of post-marketing safety data reporting (see Section 8.3.1).
- k) Blood draw for anti-SARS-CoV-2 antibodies.
- 1) For first immunization in Cohort 13, immunization with at least 30 min intervals between the primary immunizations and 30 min between the boost immunizations. For Cohorts 11 and 12, the interval between the trial subjects will be at least 15 min for the prime immunizations and at least 5 min for the boost immunizations.
- m) Oral swipe for SARS-CoV-2 testing either on Day -1 or at the Visit 1 on Day 1.
- n) The timing of the listed "research" blood draw days may be adapted (within the 200 mL maximum volume) if justified by the collected data. Leftover blood after completion of the immunogenicity assessments may be used for additional analyses as described in Section 8.7 (Genetics) and/or Section 8.8 (Biomarkers). For subjects who receive non-trial SARS-CoV-2 vaccinations, there will be no blood sampling for immunogenicity or cell-mediated immune testing in the FU Visits.
- o) For subjects who have given consent, one aliquot of the blood sample drawn for analysis of CMI may be used for HLA typing to allow additional analysis of T-cell receptor repertoire and/or phenotypic characterization of T cells specific to vaccine-encoded antigens.
- p) If HLA typing using the blood sample collected with Lithium Heparin is not conclusive, EDTA-blood will be drawn for HLA testing.
- q) When entering the follow-up phase, i.e., after completing the EoT Visit, subjects are allowed to participate in other clinical trials not investigating COVID-19 vaccines or treatments (including immunosuppressants) except COVID-19 vaccine trials with booster BNT162b2 vaccines (i.e., where they are allowed).
- r) Record any medications that trial subjects receive during the trial in the CRF starting after Visit 0 and until the respective EoT Visit; record any vaccination, including SARS-CoV-2 vaccination, that subjects receive after the EoT Visit until the last FU Visit in the CRF.
- s) Subjects who receive non-trial SARS-CoV-2 vaccinations will be discontinued. Information about these vaccinations may be received outside of a planned visit and can be collected remotely, e.g., by phone.

If the boost dose is not administered or if trial subjects permanently discontinued from IMP administration, subjects will complete all assessments listed in the SoA. Updates introduced by amendment 07 only apply for new consenting subjects after approval of the amendment.

AE = adverse event; CMI = cell-mediated immune testing; CRF = case report form; D or d = day; ECG = electrocardiogram; EDTA = ethylenediamine tetraacetic acid; EoT = end of treatment (Visit); FU = follow-up (visit); h = hour(s); HLA = human leukocyte antigen; Day 0 = one day before Day 1; IMP = investigational medicinal product; min = minute(s); SAE = serious adverse event; SARS-CoV-2 = the virus leading to COVID-19; SoA = Schedule of Activities; WOCBP = women of childbearing potential.


### Table 9: Schedule of trial procedures and assessments – BNT162b2 and B cell immunity (Cohort 14)

Note that visit numbering conforms to the equivalent days from the other BNT162b2 cohorts.

| Procedure / Assessment | Visit 0 | Visit 1<br>Pre-dose | Visit 1<br>(Post-) dosing | Visit 3 | Visit 3a | Visit 4<br>Pre-dose | Visit 4<br>(Post-) dosing | Visit 5 | Visit 7<br>(EoT Visit) | Visit 9<br>(Final Visit) |
|---|---|---|---|---|---|---|---|---|---|---|
| Day <sup>h</sup> | -30 to 0 | 1 | 1 | 8 | 15 | 22 | 22 | 29 | 50 ° | 184 |
| Days to last dose <sup>h</sup> | | 0 | 0 | 7 | 14 | 21 | 0 | 7 | 28 | 162 |
| Informed consent | Х | | | | | | | | | |
| Inclusion/exclusion criteria | X | X (review) | | | | | | | | |
| Medical history | X | X (update) | | | | | | | | |
| Physical exam. incl. height | X | X <sup>a</sup> | | X <sup>a</sup> | | X a | | X <sup>a</sup> | X <sup>a</sup> | |
| Vital signs, body weight <sup>c</sup> | Х | X | X p | X | | X | Χþ | X | X | X |
| Urine pregnancy test for WOCBP | Х | X | | | | Х | | | | |
| Urine drugs of abuse screen <sup>d</sup> | X | X | | | | | | | | |
| Alcohol breath test | Х | X | | | | | | | | |
| Urine collection for clinical laboratory <sup>e</sup> | X | X | | X | | | | X | X | |
| Blood draw for clin. lab. (15 mL) <sup>f</sup> | Х | Х | | Х | | | | Х | Х | |
| Blood draw for viral screening (5 mL) <sup>g</sup> | Х | | | | | | | | | |
| Blood draw for SARS-CoV-2 testing (2.6 mL) j | Х | | | | | | | | | |
| Oral swipe for SARS-CoV-2 testing | | X <sup>k</sup> | | | | | | | | |
| Allocation to IMP | | Х | | | | | | | | |
| Immunization | | | X | | | | Х | | | |
| Blood draw for immunogenicity (10 mL) <sup>1</sup> | | X | | X | X | Х | | X | X | X |
| Blood draw for HLA <sup>m</sup> | | | | | | X (4 mL El | DTA-blood) | | | |
| Blood draw for CMI I, n | | X<br>(≤40 mL) | | | | | | X<br>(≤40 mL) | | X<br>(≤40 mL) |
| Blood draw for biomarkers (B cells) <sup>I, n</sup> | | X<br>(≤20 mL) | | X<br>(≤40 mL) | X<br>(≤40 mL) | X<br>(≤20 mL) | | X<br>(≤40 mL) | | X<br>(≤40 mL) |
| Saliva collection | | X | | X | X | X | | Х | | |

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| Procedure / Assessment | Visit 0 | Visit 1<br>Pre-dose | Visit 1<br>(Post-) dosing | Visit 3 | Visit 3a | Visit 4<br>Pre-dose | Visit 4<br>(Post-) dosing | Visit 5 | Visit 7<br>(EoT Visit) | Visit 9<br>(Final Visit) |
|---|---|---|---|---|---|---|---|---|---|---|
| Day <sup>h</sup> | -30 to 0 | 1 | 1 | 8 | 15 | 22 | 22 | 29 | 50 ° | 184 |
| Days to last dose <sup>h</sup> | | 0 | 0 | 7 | 14 | 21 | 0 | 7 | 28 | 162 |
| Stool collection <sup>p</sup> | | X | | Х | Х | X | | X | | |
| Subject hotline availability | Start | => | => | => | => | => | => | => | => | End |
| Issue subject diaries | | X | | | | X | | | | |
| Collect subject diaries | | | | Х | | | | X | X | |
| Record AEs since last visit | | Х | | Х | | X | | Х | Х | Χİ |
| Local reaction assessment/systemic events | | | X p | Х | | | X b | Х | Х | |
| Concomitant medication <sup>q</sup> | Х | Х | | Х | | Х | | X | Х | Х |

- Brief (symptom-directed) physical examination; no height measurement.
- b) At 1, 3, and 6 h (±15 min) after immunization.
- c) Vital signs: systolic/diastolic blood pressure, pulse rate, respiratory rate, and body temperature; body weight only at Visit 0.
- d) Urine screening for drugs of abuse (amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, tricyclic antidepressants).
- e) Dipstick urine analysis: glucose, bilirubin, ketone, specific gravity, blood, pH, protein, urobilinogen, nitrite, and leukocytes. Microscopic urinalysis: if warranted by dipstick results, urine sediment will be microscopically examined for the presence of red blood cells, white blood cells, casts, crystals, epithelial cells, and bacteria.
- f) Clinical laboratory tests: (Chemistry) alkaline phosphatase, creatinine, ferritin, C-reactive protein, albumin, alanine aminotransferase, amylase, aspartate aminotransferase, gamma glutamyl transpeptidase, total bilirubin, blood urea nitrogen, glucose, lipase, sodium, potassium, calcium; (Hematology) hemoglobin, hematocrit, red blood cell count, white blood cell count and differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count. Only in women who are not WOCBP (to confirm postmenopausal status): follicle stimulating hormone at Visit 0.
- q) Viral screening for human immunodeficiency virus (HIV) 1 or 2, hepatitis B, hepatitis C.
- h) Flexibility for visit days: Visit 3 Day 8±1 d; Visit 3a Day 15±2 d; Visit 4 Day 22±2 d; Visit 5 Day 29±3 d; Visit 7 Day 50±4 d; Visit 9 Day 184±9 d.
- i) Visit 9, only IMP-related AEs and any SAEs. Proven COVID-19 cases which have to be reported regardless on severity and relatedness to the trial drug until the last scheduled FU Visit as described in Section 10.3.1.9.
- Blood draw for anti-SARS-CoV-2 antibodies.
- k) Oral swipe for SARS-CoV-2 testing either on Day -1 or at the Visit 1 on Day 1.
- 1) The timing of the listed blood draw days may be adapted, as long as the total volume drawn does not change, if justified by the collected data. Leftover blood after completion of the immunogenicity assessments may be used for additional analyses as described in Section 8.7 (Genetics) and/or Sections 8.8 and 8.9 (Biomarkers).
- m) If HLA typing using the blood sample collected with Lithium Heparin is not conclusive, EDTA-blood will be drawn for HLA testing.
- n) For subjects who have given consent, one aliquot of the blood sample drawn for analysis of CMI or biomarkers (B cells) may be used for HLA typing to allow additional analysis of T-cell receptor repertoire and/or phenotypic characterization of T cells specific to vaccine-encoded antigens.
- b) When entering the follow-up phase, i.e., after completing the EoT Visit, subjects are allowed to participate in other clinical trials not investigating COVID-19 vaccines or treatments (including immunosuppressants) except COVID-19 vaccine trials with booster BNT162b2 vaccines (i.e., where they are allowed).
- p) Flexibility for stool sample collection is the specified visit day ±48 h, with the possibility of collection at home by providing subjects with sample tubes.

### Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


q) Record any medications that trial subjects receive during the trial in the CRF starting after Visit 0 and until the respective EoT Visit; record any vaccination, including SARS-CoV-2 vaccination, that subjects receive after the EoT Visit until the last FU Visit in the CRF.

Note: If a second dose of SARS-CoV-2 vaccine is not administered or if trial subjects permanently discontinue from IMP administration, subjects will be asked to complete all assessments listed in the SoA.

AE = adverse event; CMI = cell-mediated immune testing; CRF = case report form; D or d = day; EDTA = ethylenediamine tetraacetic acid; EoT = end of treatment (Visit); h = hour(s); FU = follow-up (visit); HLA = human leukocyte antigen; Day 0 = one day before Day 1; IMP = investigational medicinal product; min = minute(s); SAE = serious adverse event; SARS-CoV-2 = the virus leading to COVID-19; SoA = Schedule of Activities; WOCBP = women of childbearing potential.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### **TABLE OF CONTENTS**

| 1 | PROTOCOL SUMMARY | 3 |
|--------|-------------------------------------------------------|----|
| 1.1 | Trial synopsis | 3 |
| 1.2 | Schema (graphical representation of the trial) | 19 |
| 1.3 | Schedule of activities | 21 |
| TABLE | OF CONTENTS | 33 |
| LIST O | F TABLES | 37 |
| LIST O | F FIGURES | 37 |
| TRIAL- | SPECIFIC ABBREVIATIONS/TERMS | 38 |
| 2 | INTRODUCTION | 40 |
| 2.1 | Background | 40 |
| 2.1.1 | Overview of the disease | 40 |
| 2.1.2 | Introduction to BioNTech RNA-based vaccines | 40 |
| 2.2 | Trial rationale | 41 |
| 2.3 | Benefit/risk assessment | 41 |
| 2.3.1 | Risk assessment | 42 |
| 2.3.2 | Benefit assessment | 46 |
| 2.3.3 | Overall benefit/risk conclusion | 46 |
| 3 | OBJECTIVES AND ENDPOINTS | 47 |
| 4 | TRIAL DESIGN | 50 |
| 4.1 | Overall design | 50 |
| 4.1.1 | Adaptive trial design elements | 54 |
| 4.1.2 | Planned number of trial subjects | 54 |
| 4.2 | Scientific rationale for the trial design | 54 |
| 4.3 | Justification for dose | 56 |
| 4.4 | End of treatment (EoT) and end of trial definition | 57 |
| 5 | TRIAL POPULATION | 58 |
| 5.1 | Inclusion criteria | 58 |
| 5.1.1 | Inclusion criteria Part A | 58 |
| 5.2 | Exclusion criteria | 59 |
| 5.2.1 | Exclusion criteria Part A | 59 |
| 5.3 | Lifestyle considerations | 62 |
| 5.4 | Screen failures | 63 |
| 6 | TRIAL TREATMENTS | 63 |
| 6.1 | IMP administered | 63 |
| 6.2 | Preparation/handling/storage/accountability | 63 |
| 6.3 | Measures to minimize bias: randomization and blinding | 64 |

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| 6.4 | Trial treatment compliance | 64 |
|---|---|---|
| 6.5 | Concomitant therapy | 64 |
| 6.5.1 | Premedication | 65 |
| 6.5.2 | Rescue medication | 65 |
| 6.6 | Dose modifications | 65 |
| 6.6.1 | Dose limiting toxicity | 65 |
| 6.6.2 | Dose modification guidance/rules | 66 |
| 6.6.3 | Mitigation plans for specific AEs | 67 |
| 6.6.4 | Safety stopping criteria | 67 |
| 6.7 | Treatment after the end of the trial | 67 |
| 7 | DISCONTINUATION OF TRIAL TREATMENT AND TRIAL SUBJECT DISCONTINUATION/WITHDRAWAL | 68 |
| 7.1 | Discontinuation of trial treatment | 68 |
| 7.1.1 | Temporary discontinuation | 68 |
| 7.1.2 | Rechallenge | 68 |
| 7.2 | Trial subject discontinuation/withdrawal from the trial | 68 |
| 7.3 | Lost to follow-up | 69 |
| 7.4 | Replacement of permanently discontinued trial subjects | 69 |
| 8 | TRIAL ASSESSMENTS AND PROCEDURES | 69 |
| 8.1 | Efficacy assessments | 70 |
| 8.2 | Safety assessments | 70 |
| 8.2.1 | Physical examinations | 70 |
| 8.2.2 | Vital signs | 70 |
| 8.2.3 | Electrocardiograms | 71 |
| 8.2.4 | Clinical laboratory tests | 71 |
| 8.2.5 | Drugs of abuse screening | 71 |
| 8.2.6 | Testing for alcohol use | 71 |
| 8.2.7 | Viral screening (for blood-borne viruses) | 71 |
| 8.2.8 | Subject diaries | 72 |
| 8.2.9 | Assessment of local reactions | 72 |
| 8.2.10 | SARS-CoV-2 testing | 72 |
| 8.2.11 | Subject hotline | 73 |
| 8.2.12 | Subject wellbeing questioning | 73 |
| 8.2.13 | Assessment of systemic reactions | 73 |
| 8.3 | Adverse events and serious adverse events | 74 |
| 8.3.1 | Time period and frequency for collecting AE and SAE information | 74 |
| 8.3.2 | Method of detecting AEs and SAEs | 74 |
| 8.3.3 | Follow-up of AEs and SAEs | 74 |

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| 8.3.4 | Regulatory reporting requirements for SAEs | 75 |
|---|---|---|
| 8.3.5 | Pregnancy | 75 |
| 8.3.6 | Death events | 76 |
| 8.3.7 | Disease-related events and/or disease-related outcomes not qualifying or SAEs | as AEs<br>76 |
| 8.3.8 | Adverse events of special interest | 76 |
| 8.4 | Treatment of overdose | 76 |
| 8.5 | Pharmacokinetics | 77 |
| 8.6 | Pharmacodynamics | 77 |
| 8.7 | Genetics | 77 |
| 8.8 | Biomarkers (CMI responses, explorative biomarker, immunogenicity repurposes) | search<br>77 |
| 8.9 | Biomarkers (B cells) | 78 |
| 8.10 | Immunogenicity assessments | 79 |
| 8.11 | Blood collection | 80 |
| 8.12 | Saliva and stool collection | 80 |
| 9 | STATISTICAL CONSIDERATIONS | 81 |
| 9.1 | Statistical hypotheses | 81 |
| 9.2 | Sample size determination | 81 |
| 9.3 | Analysis sets | 81 |
| 9.4 | Statistical analyses | 81 |
| 9.4.1 | General considerations | 82 |
| 9.4.2 | Primary endpoints | 82 |
| 9.4.3 | Secondary endpoints | 83 |
| 9.4.4 | Exploratory endpoints | 83 |
| 9.4.5 | Other safety analyses | 83 |
| 9.4.6 | Other analyses | 84 |
| 9.5 | Interim analyses | 84 |
| 9.6 | Data Monitoring Committee | 85 |
| 10 | SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDER | ATIONS<br>85 |
| 10.1 | Regulatory, ethical, and trial oversight considerations | 85 |
| 10.1.1 | Regulatory and ethical considerations | 85 |
| 10.1.2 | Financial disclosure | 86 |
| 10.1.3 | Informed consent process | 86 |
| 10.1.4 | Data protection | 86 |
| 10.1.5 | Committees - SRC | 87 |
| 10.1.6 | Dissemination of clinical trial data | 87 |
| 10.1.7 | Data quality assurance | 87 |

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| 10.1.8 | Source documents | 88 |
|---|---|---|
| 10.1.9 | Trial and site start and closure | 88 |
| 10.1.10 | Publication policy | 89 |
| 10.1.11 | Protocol preparation and approval | 89 |
| 10.2 | Clinical laboratory tests | 89 |
| 10.3 | Adverse events: Definitions and procedures for recording, evaluating and reporting | ı, follow-up,<br>90 |
| 10.3.1 | Definition of AE and TEAE | 90 |
| 10.3.1 | Contraceptive guidance and collection of pregnancy information | 102 |
| 10.4.1 | Definitions | 102 |
| 10.4.1 | Contraception guidance | 102 |
| 10.4.3 | Collection of pregnancy Information | 103 |
| 10.4.4 | Sperm donation | 104 |
| 10.5 | Genetics | 104 |
| 10.6 | Liver safety: Suggested actions and follow-up assessments | 104 |
| 10.7 | Investigators and trial administrative structure | 104 |
| 10.7.1 | Investigators and trial site personnel | 104 |
| 10.7.2 | Trial site personnel assigned trial-related duties | 104 |
| 10.7.3 | Contract research organizations | 105 |
| 10.7.4 | The sponsor and sponsor's personnel | 105 |
| 10.8 | Country-specific requirements | 105 |
| 10.9 | Other standard abbreviations and definitions | 106 |
| 10.10 | Protocol amendments and version updates | 107 |
| 10.10.1 | Protocol amendment no. 01 | 107 |
| 10.10.2 | Protocol amendment no. 02 | 107 |
| 10.10.3 | Protocol amendment no. 03 | 107 |
| 10.10.4 | Protocol amendment no. 04 | 108 |
| 10.10.5 | Protocol amendment no. 05 | 108 |
| 10.10.6 | Protocol amendment no. 06 | 108 |
| 10.10.7 | Protocol amendment no. 06 (protocol version 10.0) | 110 |
| 10.10.8 | Protocol amendment no. 07 (protocol version 11.0) | 110 |
| 10.10.9 | Protocol amendment no. 08 (protocol version 12.0) | 110 |
| 10.10.10 | Protocol amendment no. 09 (protocol version 13.0) | 111 |
| 10.11 | Data collection and management | 111 |
| 10.11.1 | Case report forms | 111 |
| 10.11.2 | Trial subject reported outcomes | 111 |
| 10.11.3 | Data management | 111 |
| 10.11.4 | Investigator's Site File and the Trial Master File | 112 |
 Clinical Trial Protocol BioNTech SE including Amendments Nos. 01 to 09 Version: 13.0 Confidential BNT162-01 Date: 12 JAN 2022 10.12 Other data 112 10.12.1 Demographic data 112 Medical history 112 10.12.2 11 **REFERENCES** 112 LIST OF TABLES Table 1: Dose ranging: vaccine dose regimens for younger adults aged 18 to 55 years in Part A (Cohorts 1 to 7) 11 Dose ranging: vaccine dose regimens for older adults aged 56 to 85 years in Table 2: Part A (Cohorts 8 to 10) 12 Table 3: Expansion cohorts for BNT162b2 (ages 18 to 85 years) in Part A (Cohorts 11 to 13) 13 Table 4: Cohort 14 for BNT162b2 (ages 18 to 85 years) in Part A 13 Table 5: Overview of the total number of subjects for each vaccine in Part A 14 Table 6: Schedule of trial procedures and assessments – BNT162a1, BNT162b1, BNT162b2, and BNT162c2 when tested P/B (excluding Cohorts 11 to 14) 21 Table 7: Schedule of trial procedures and assessments – BNT162c2 (SD) 24 Schedule of trial procedures and assessments – Cohorts 11 to 13 (Expansion Table 8: cohorts only) 27 Schedule of trial procedures and assessments – BNT162b2 and B cell immunity Table 9: (Cohort 14) 30 Table 10: Probability to observe a particular TEAE at least once 81 Table 11: Local reaction grading scale 99 Table 12: Systemic reaction grading scale 100 Table 13: Fever grading scale 100 Table 14: Laboratory abnormality grading scale 101 LIST OF FIGURES Figure 1: Graphical depiction of the dose-finding and expansion process in Part A 20

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


## TRIAL-SPECIFIC ABBREVIATIONS/TERMS

| Abbreviation/Term | Explanation |
|---|---|
| Allocated subject | Enrolled subjects who are allocated to IMP |
| BNT162-02 | C4591001 according to the Pfizer trial code |
| BNT162a | BNT162 RNA-LNP vaccine utilizing uRNA (the variant BNT162a1 will be tested in this trial) |
| BNT162b | BNT162 RNA-LNP vaccine utilizing nucleoside modified mRNA (the variants BNT162b1 and BNT162b2 will be tested in this trial) |
| BNT162c | BNT162 RNA-LNP vaccine utilizing self-amplifying mRNA (the variant BNT162c2 will be tested in this trial) |
| C4591001 | BNT162-02 according to the BioNTech trial code |
| CMI | Cell-mediated immunity/immune |
| COVID-19 | Coronavirus Disease 2019 |
| DRFZ | Deutsches Rheuma-Forschungszentrum Berlin |
| ECG | Electrocardiogram |
| Elderly (adults) | As defined in ICH E7, individuals aged 65 years or older |
| ELISA | Enzyme-Linked Immunosorbent Assay |
| ELISpot | Enzyme-Linked Immunosorbent Spot |
| Enrolled subjects | Subjects who signed an informed consent form, i.e., who gave informed consent |
| FIH | First-in-human |
| HLA | Human leukocyte antigen |
| IM | Intramuscular(ly) |
| IV | Intravenous(ly) |
| modRNA | Nucleoside modified messenger RNA |
| mRNA | Messenger RNA |
| Older (adults) | Defined in this document to be individuals aged 56 to 85 years |
| P/B | Prime/Boost: a dosing regimen, comprising a priming immunization and a boost immunization |
| PBMC | Peripheral blood mononuclear cell |
| PEI | (German) Paul-Ehrlich-Institut |
| RNA-LNP | RNA lipid nanoparticle |
| saRNA | Self-amplifying messenger RNA |
| SARS-CoV-2 | Severe Acute Respiratory Syndrome Coronavirus 2, the virus leading to COVID-19 |
| SD | Single dose (also referred to as "single priming dose" or "single immunization") |
| uRNA | Non-modified uridine containing mRNA |
| VNT | Virus neutralization test |
| Younger (adults) | Defined in this document to be individuals aged 18 to 55 years |

For standard abbreviations, see Section 10.9.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### **NOTES FOR THE READER**

When the term "must" is used, the action/item is always mandatory. Non-compliance with this instruction constitutes a protocol deviation. When the term "should" is used, the action/item is recommended but not mandatory. Non-compliance with this instruction does not constitute a protocol deviation.


### 2 INTRODUCTION

## 2.1 Background

#### 2.1.1 Overview of the disease

Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infections and the caused disease Coronavirus Disease 2019 (COVID-19) are increasing every day and spreading globally, affecting more and more countries.

On March 11<sup>th</sup>, 2020 the World Health Organization (WHO) characterized the COVID-19 outbreak as pandemic.

The WHO Situation Update Report dated April 15<sup>th</sup>, 2020 noted 1,914,916 confirmed cases with 123,010 deaths globally, including 977,596 confirmed cases with 84,607 deaths in the European region (WHO Situation Report Nr. 85).

### 2.1.2 Introduction to BioNTech RNA-based vaccines

An LNP-formulated RNA-based vaccine would provide one of the most flexible, scalable and fastest approaches to provide protection against the emerging viruses like SARS-CoV-2 (Rauch et al. 2018; Sahin et al. 2014).

The development of an RNA-based vaccine encoding a viral antigen that is translated to protein by the vaccinated organism to induce a protective immune response provides significant advantages over more conventional vaccine approaches. Unlike live attenuated vaccines, RNA vaccines do not carry the risks associated with infection and may be given to people who cannot be administered live virus (such as pregnant women and immunocompromised persons). RNA-based vaccines are manufactured via a cell-free *in vitro* transcription process, which allows an easy and rapid production, and the prospect of producing high numbers of vaccination doses within a shorter time period than achieved with conventional vaccine approaches. This capability is pivotal to enable the most effective response in outbreak scenarios.

The development of *in vitro* transcribed RNA as an active platform for the use in infectious disease vaccines is based on the extensive knowledge of the company in RNA technology, which has been gained over the last decade. The core innovation is based on *in vivo* delivery of a pharmacologically optimized, antigen-encoding RNA to induce robust neutralizing antibodies and a concomitant T-cell response to achieve protective immunization with minimal vaccine doses (Vogel et al. 2018; Moyo et al. 2018; Pardi et al. 2017).

At BioNTech, there are three different RNA platforms under development, namely non-modified uridine containing mRNA (uRNA, BNT162a), nucleoside modified mRNA (modRNA, BNT162b), and self-amplifying mRNA (saRNA, BNT162c).

All three RNA platforms have been tested in more than a dozen non-clinical GLP safety studies and, for uRNA and modRNA, there is pre-existing clinical safety data (see the BNT162 investigator's brochure [IB]). These data have been obtained primarily with RNAs

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


formulated with liposomes which are related, but not identical, to those to be used in this trial.

The non-clinical toxicity data generated by BioNTech suggest a favorable safety profile for uRNA and modRNA, as well as saRNA formulated with different nanoparticles for various administration routes, including intravenous (IV) injection. The favorable safety profile after IV dosing is notable because it results in a higher systemic exposure than the planned IM dosing in this trial. Overall, the findings were mild and mostly related to the mode-of-action and the RNA-intrinsic stimulation of innate immune sensors. No unsuspected target organs of toxicity were identified. The non-clinical safety profile of uRNA and modRNA in rodents was predictive for clinical safety. For further details, see the BNT162 IB.

The safety and toxicity of the lipid nanoparticle enveloped uRNA, modRNA, and saRNA vaccines encoding coronavirus antigens is currently being analyzed in a GLP-compliant repeated-dose toxicity study.

A recently published clinical trial using an influenza vaccine based on modRNA encapsulated in LNPs highly related to those used in this trial and also administered IM reported good safety and well tolerability (Feldman et al. 2019).

### 2.2 Trial rationale

SARS-CoV-2 infections and the caused disease COVID-19 are increasing every day and spreading globally, affecting more and more countries, and carrying a high risk of rapidly becoming pandemic (for more details, see Section 2.1.1). There are currently no vaccines or antiviral drugs to treat these infections or its caused disease COVID-19. Therefore, there is an unmet need for the rapid development of effective prophylactic vaccines.

BioNTech has developed a technology platform of RNA-based vaccines which enables the rapid development of vaccines against emerging viral diseases (for more details, see Section 2.1.2). This technology platform is especially attractive because it has the ability to deliver high numbers of vaccine doses rapidly in a single production campaign.

This trial investigates the potential safety and immunogenicity of four prophylactic BNT162 vaccines against SARS-CoV-2, BNT162a1, BNT162b1, BNT162b2, and BNT162c2. The two variants of the BNT162b vaccines, BNT162b1 and BNT162b2, differ in the encoded antigen.

Some of the prophylactic BNT162 vaccines against SARS-CoV-2 investigated in this trial are under investigation in other ongoing trials. For the design, status, and a summary of the available results of the ongoing clinical trials, see the BNT162 IB.

### 2.3 Benefit/risk assessment

More detailed information about the known and expected benefits and risks and reasonably expected TEAEs for this trial are given in the BNT162 IB.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


#### 2.3.1 Risk assessment

The risks linked to the trial-specific procedures and connected mitigations are as follows:

- The volume of blood drawn will be kept to a minimum and will remain less than that drawn when donating blood:
  - For subjects in Cohorts 1 to 10, up to approximately 592 mL blood will be drawn per subject over the complete trial, i.e., over approximately 223 d.
  - For subjects in Cohorts 11 to 13, up to approximately 1,025 mL blood will be drawn per subject over the complete trial, i.e., over approximately 760 d.
  - For subjects in Cohort 14, up to approximately 477 mL blood will be drawn per subject over the complete trial, i.e., over approximately 223 d.
- All trial-specific procedures will be performed by qualified trial site personnel.
- Immunization will be done by a physician.
- Human experience with BNT162 vaccines was not available prior to this trial.
  However, clinical data was available for RNAs formulated with related but not
  identical liposomal compositions or non-formulated RNAs and can support risk
  assessment of the BNT162 vaccines.

Based on such data, the risks linked to the immunization with the BNT162 vaccines are as follows:

- Due to the IM route of administration, there is the risk of local reactions at the injection site, e.g., erythema, pruritus, pain, tenderness, swelling, sweating.
- Due to their immune-modulatory effect, vaccines may cause systemic flu-like reactions such as temporary headache, fatigue, loss of appetite, myalgia, arthralgia, fever. Rarely, with certain prophylactic vaccines (e.g., as seen for vaccines using attenuated viruses) severe allergic reaction or a neurological side effects, such as a seizure, were seen. Although these rare side effects are a concern, the risk of a vaccine causing serious harm or death is considered to be extremely small, in particular for BNT162 vaccines, which are molecularly defined, highly purified and based on RNA, which naturally occurs and is metabolized in the human organism.
- Due to the IM route the risk of systemic reactions is considered low.
- As with other vaccines, and with single stranded RNA being an innate immune sensor-agonist, BNT162 vaccine administration may cause temporary headache, fatigue, or loss of appetite. Rarely, with certain prophylactic vaccines (e.g., as seen for vaccines using attenuated viruses) severe allergic reactions or neurological side effects, such as seizures, were seen. Although these rare side effects are a concern, the risk of a vaccine causing serious harm or death is considered to be extremely small, in particular for BNT162 vaccines, which are molecularly defined, highly purified, subunit vaccines.

The available non-clinical data of BNT162a, BNT162b, and BNT162c suggest a favorable safety profile with events that are mild and mostly related to the mode-of-action and the RNA-intrinsic stimulation of innate immune sensors.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


 Based on the available clinical and non-clinical data on the individual components (uRNA, modRNA, saRNA, the specific LNP formulation), that are combined within the BNT162 products, a favorable safety profile of BNT162 products is expected with mild and localized effects (see the BNT162 IB for details on these trials).

To date, based on available clinical experience with BNT162 vaccines in human subjects:

- Generally, good tolerability was observed. Overall, many of the reported TEAEs appear to be similar to reactogenicity events anticipated for IM-administered vaccines, typically with an onset within first 24 h post immunization. All events / reactogenicity symptoms resolved spontaneously, mostly within 24 h of onset, and were managed with simple measures (e.g., paracetamol). There were no serious adverse events (SAEs) and no unexpected toxicities. Most TEAEs were managed with simple measures and resolved spontaneously.
- The adverse reactions (AEs for which there is a reason to conclude that the vaccine caused the events) identified for BNT162 vaccines at this time are: injection site pain, fever, fatigue, headache, chills, and muscle pain.
- While the general risk of effects potentially associated with the innate immune
  activation and transient secretion of associated cytokines are defined above based
  on the described data, the dose response-relationship, and thus the tolerability for
  the BNT162 vaccine candidates will only be defined by the ongoing trials (for a
  summary of the ongoing trials, see the BNT162 IB).
- The clinical experience after P/B dosing with BNT162b1 at 10, 20, and 30 μg and single doses of BNT162b2 at 10, 20, and 30 μg, in healthy elderly adults aged 65 to 85 years is summarized in the BNT162 IB.
- The local tolerability of BNT162b1 and BNT162b2 in elderly adults seemed comparable to that recorded in younger adults aged 18 to 55 years. Likewise, the pattern of systemic reactogenicity appeared similar between the 2 age groups, possibly with a lower overall incidence in the elderly adults in comparison to the younger adults at equal doses (for details, see the BNT162 IB).
- Preliminary data in elderly adults, show lower but measurable antibody responses in older adults than in younger adults (for details, see the BNT162 IB). The investigation of higher dose range in older adults in this trial may therefore be required to support the Phase III program planned to support marketing approval.
- When assessing the risk for dosing of older subjects with BNT162 vaccine candidates in this trial, the follow information is relevant:
  - Preliminary data in subjects treated in the ongoing BNT162 trials backed by non-human primate (rhesus macaque) immunogenicity data have shown that BNT162b1 in the tested dose range is immunogenic.
  - The risk that older adults may be under dosed with the vaccine doses chosen based on data for younger adults (as was observed for other vaccines).

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


 Preliminary data in elderly show a comparable to lower reactogenicity based on the observed local reactions and system events in similar doses. This observation may indicate a lower innate response in younger adults.

- In this trial, the P/B BNT162b1 and BNT162b2 doses planned in older adults (10, 20, and 30 μg) are within the range already shown to show acceptable tolerability in younger adults and in elderly adults in this trial and/or BNT162-02 trial (for details, see the BNT162 IB). This tolerability in elderly adults appears to be better than seen in younger adults at the same doses.
- Although using doses already found to show acceptable tolerability in younger adults and an even better tolerability in elderly adults, this trial implements numerous safety measures (e.g., sentinel dosing/staggering of subjects, on site observation periods after each immunization, wellbeing questioning, frequent on site visits after immunization).
- This trial includes inclusion/exclusion criteria to exclude potential risk factors relevant for all adults, but additional criteria have been included to further protect the safety of enrolled older adults.
- The listed risks can be managed using routine symptom driven standard of care as described in Section 6.6.3. Treatment of these events is dependent on the discretion of the investigators.
- Since this trial involves the first immunization of humans with the BNT162 vaccines, in the FIH cohorts and all dose escalation cohorts use a sentinel dosing/staggering of subjects (EMA 2017 guidance "Strategies to Identify and Mitigate Risks for Firstin-Human and Early Clinical Trials with Investigational Medicinal Products").

To further ensure trial subject safety during dose ranging cohorts, the trial protocol foresees that:

- On site observation periods after each immunization (i.e., 24 h for the first 6 subjects per group and 6 h for other subjects in the same group) that are much longer than used in recently completed FIH clinical trials investigating related RNAbased vaccines. For example, the 2 Moderna trials investigating mRNA vaccines against avian H10N8 and H7N9 influenza viruses in healthy adults (Feldman et al. 2019) that observed trial subjects on site for only 1 h after each immunization before discharge from the trial site.
- More frequent on site visits after immunization (i.e., on Days 2 and 8) than used in recently completed FIH clinical trials investigating with related RNA-based vaccines, e.g., the 2 Moderna trials investigating mRNA vaccines against avian H10N8 and H7N9 influenza viruses in healthy adults (Feldman et al. 2019) that used on site visits on Day 8.
- Subject wellbeing questioning by telephone at 48±2 h after each immunization (where applicable, after both the prime and boost immunizations) will be performed for the first 6 subjects per cohort. Additional subject wellbeing calls may be included at the discretion of the SRC.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- In the case that an individual experiences dose limiting toxicities or that the frequency or pattern of AEs within a sub-cohort gives cause for concern, the investigator may request an ad hoc review by the SRC before further doses of a given vaccine construct are administered.
- If the investigator considers necessary, the planned observation periods before proceeding to dose further subjects in the same group may be prolonged by 24 h.
- The SRC must assess the safety and tolerability data of the first 6 subjects before allowing progression to the next cohort, for each vaccine per cohort/dose level.
- After each assessment, the SRC may request a prolongation of the observation periods to up to Day 7 for later cohorts. Experience in this ongoing trial and in the ongoing BNT162-02 trial, has confirmed the adequacy of the implemented observations periods.
- The SRC may make recommendations on increasing observation periods and additional subject wellbeing calls may be included at the discretion of the SRC.
- To ensure trial subject safety during the trial, their safety will be monitored from Visit 0 (screening) until approximately 6 months after the last immunization.

#### For the expansion cohorts:

- Due to the extensive experience and exposure already achieved with BNT162b2 at 30 μg in the ongoing global Phase I/II/III trial (from which frequent, rolling safety data submissions to health authorities are being made) the measures implemented for dose ranging cohorts are deemed unnecessary for the expansion cohorts (by 20 JAN 2021, more than 25,000 trial subjects have been dosed at least once with BNT162b2).
- Immunocompromised individuals are considered at increased risk from infection
  with SARS-CoV-2 and of infections in general. Risk minimization measures already
  in place for the protection of all subjects in this trial are also considered sufficient to
  protect this increased risk group, who are generally regarded as ambulatory in
  nature. Care should however be taken to avoid unnecessary extension of on site
  time and site visits for these subjects, to minimize their risk of exposure to high risk
  pathogens.

Vaccine-related enhanced disease has been reported in the literature from non-clinical studies investigating different vaccine formulations tested to prevent various coronavirus-induced diseases. Such effects have not been documented so far for SARS-CoV-2. No data are currently available to exclude that BNT162 may cause enhanced disease in vaccinated subjects.

The risks linked to the pandemic COVID-19 outbreak will be managed by requiring that the trial subjects:

 Avoid contact with persons tested positive for SARS-CoV-2 antibodies or have an increased risk for infection during their participation in the trial.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- Practice social distancing and follow good practices to reduce their chances of being infected or spreading COVID-19 during their participation in the trial.
- Complete health status checks which include symptom-directed physical examinations, vital signs assessments, and clinical laboratory tests at the planned visit days.
- Use the Subject Hotline to contact the trial site during their participation in the trial should they require guidance or should they experience any symptoms of illness. The reporting of any symptoms of illness, e.g., enhanced respiratory disease or flulike symptoms, may trigger diagnostic measures at the discretion of the investigator.

To minimize the risk to trial subjects in this trial, an SRC will regularly review and evaluate the safety and immunogenicity data. For details, see Section 10.1.5.

#### 2.3.2 Benefit assessment

After participating in this trial, depending on the immunization regimen followed, some trial subjects should be immune against SARS-CoV-2 infection.

There is an urgent need for the development of new prophylactic vaccines given the threat posed by the increasing number of globally distributed outbreaks of SARS-CoV-2 infection. The BioNTech platform of RNA-based vaccines being tested in this trial is especially attractive because it has the ability to deliver high numbers of vaccine doses rapidly in a single production campaign. This platform has the added advantage of not employing live virus and could therefore potentially be used for immuno-compromised populations.

By participating in this trial, the trial subjects will support the development of one or more prophylactic vaccines against SARS-CoV-2 infection.

#### 2.3.3 Overall benefit/risk conclusion

Overall, the sponsor considers the benefit/risk ratio to be acceptable for a trial of this type.


#### 3 OBJECTIVES AND ENDPOINTS

#### Objectives Endpoints a Primary objective (All cohorts) Solicited local reactions at the injection site (pain, tenderness, erythema/redness, induration/swelling) recorded up to 7 d after each To describe the safety immunization (trial days 8 and 29). and tolerability profiles of prophylactic BNT162 Solicited systemic reactions (nausea, vomiting, diarrhea, headache, vaccines in healthy fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and fever) adults after single dose recorded up to 7 d after each immunization (trial days 8 and 29). (SD; prime only) or The proportion of subjects with at least 1 unsolicited treatmentprime/boost (P/B) emergent adverse event (TEAE): immunization. For BNT162a1, BNT162b1, BNT162b2, and BNT162c2 (P/B): occurring up to 21 d after the prime immunization (trial day 22) and 28 d after the boost immunization (trial day 50). For BNT162c2 (SD): The proportion of subjects with at least 1 unsolicited TEAE occurring up to 28 d after the immunization (trial day 29).

#### Secondary objectives

#### (All cohorts)

To describe the immune response in healthy adults after SD or P/B immunization measured by a functional antibody titer, e.g., virus neutralization test (VNT) or an equivalent assay available by the time of trial conduct.

#### For BNT162a1, BNT162b1, BNT162b2, and BNT162c2 (P/B)

As compared to baseline at 7 and 21 d after primary immunization (trial days 8 and 22) and at 7, 14 b, 21, 28, 63, and 162 d after the boost immunization (trial days 29 to 184):

- · Functional antibody responses (titers).
- Fold increase in functional antibody titers.
- Number of subjects with seroconversion defined as a minimum of 4-fold increase of functional antibody titers as compared to baseline.

#### For BNT162c2 (SD)

As compared to baseline at 7, 21, 28, 42, 84, and 183 d after the primary immunization (trial days 8 to 184):

- Functional antibody responses (titers).
- Fold increase in functional antibody titers.
- Number of subjects with seroconversion defined as a minimum of 4-fold increase of functional antibody titers as compared to baseline.

#### For Cohort 14 with BNT162b2

As compared to baseline at 7, 14, and 21 d after primary immunization (trial days 8, 15, and 22) and at 7, 28, and 162 d after the boost immunization (trial days 29, 50, and 184):

- · Functional antibody responses (titers).
- Fold increase in functional antibody titers.
- Number of subjects with seroconversion defined as a minimum of 4-fold increase of functional antibody titers as compared to baseline.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Objectives Endpoints <sup>a</sup> **Exploratory objectives** 

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01





### 4 TRIAL DESIGN

## 4.1 Overall design

This trial has two parts. Part A and Part B. Due to changes in the overall clinical development plan, Part B will no longer be conducted. The objectives originally described for Part B have been implemented in the ongoing development via a pivotal Phase I/II/III trial BNT162-02/C4591001 (NCT04368728).

Part A is for dose ranging of four different vaccines (BNT162a1, BNT162b1, BNT162b2, and BNT162c2) will be undertaken with dose escalation and de-escalation plus the evaluation of interim dose levels. It also includes dose ranging in older subjects.

The vaccines BNT162a1, BNT162b1, BNT162b2, and BNT162c2 will be administered using a P/B regimen. The vaccine BNT162c2 will also be administered using a SD regimen.

BNT162b2, for which the dose regimen has been determined in the dose ranging in Part A of this trial, has now entered efficacy evaluation in the ongoing development via a pivotal Phase I/II/III trial BNT162-02/C4591001 (NCT04368728). Therefore, for BNT162b2, amendment 06 of this trial introduced expansion cohorts designed to expand the existing safety profiling to a broader population and to enable detailed characterization of the adaptive immune responses, including determine factors that impact them. These cohorts will involve healthy and immunocompromised populations treated according to the selected dosing posology and exploring an alternative posology.

The chosen trial design reflects discussion and advice from the PEI obtained in scientific advice meetings held in February, March, and June 2020 in response to a fast-changing situation.

For a summary of the trial as a flow diagram, see the Schema in Section 1.2. For the planned assessments and visits, see the Schedule of Activities (SoA) in Section 1.3.

#### Part A

The first part of the trial (Part A) will follow a dose escalation design. Discretionary dose de-escalation and refinement is also planned. Part A will consist of a screening/treatment phase and a follow-up phase.

### **Dose ranging cohorts:**

Trial subjects with the FIH immunization will be immunized using a sentinel dosing/subject staggering (EMA 2017 guidance "Strategies to Identify and Mitigate Risks for First-in-Human and Early Clinical Trials with Investigational Medicinal Products"). The FIH starting dose and the planned escalation/de-escalation doses are given in Table 1. Dose escalation rules have been defined in this protocol to guide dose escalation.

For all cohorts, if the investigator considers necessary, the planned observation periods before proceeding to dose further subjects in the same group may be prolonged by 24 h.

Dose de-escalation in the case of possible vaccine-related toxicities will be guided by the Safety Review Committee (SRC), as required.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


In Cohort 1, the sentinel dosing/subject staggering process will be as follows:

- One sentinel subject will be dosed on one day.
- If the dosing in this subject was considered to be safe and well tolerated by the investigator after 24±2 h observation on site, a 5 further subjects will be dosed (with intervals of at least 1 h between subjects).
- If the dosing in these 5 subjects was considered to be safe and well tolerated by the investigator based on 48 h data (24±2 h observation on site and phone interview for assessment 48±2 h after immunization; in addition to the available 48±2 h data from the sentinel subject):
  - The remaining 6 subjects in the group will be dosed (with intervals of at least 30 min between subjects).
  - o If approved by the SRC, the next planned escalation dose (see Table 1) will be initiated. The data assessed by the SRC comprises 48 h data for 6 subjects including observation on site, short summary of phone interview (including statement about diary reports), vital signs, investigator reported local and systemic reactions, TEAEs, solicited local & systemic reactions, blood/clinical laboratory data, and brief physical examination outcome.
  - If approved by the SRC, the planned de-escalation dose in Cohort 3 will be initiated.

For any subsequent dose escalation cohorts (to doses higher than the maximum already tested for a vaccine candidate), the sentinel/subject staggering process will be as follows:

- Two sentinel subjects will be dosed on one day (with intervals of at least 30 min between subjects).
- If the dosing in these subjects was considered to be safe and well tolerated by the investigator after 24±2 h observation on site, a 4 further subjects will be dosed (with intervals of at least 30 min between subjects).
- If the dosing in these 4 subjects was considered to be safe and well tolerated by the investigator based on 48 h data (24±2 h observation on site and phone interview for assessment 48±2 h after immunization; in addition to the available 48 h data from the sentinel subjects):
  - The remaining 6 subjects in the group will be dosed (with intervals of at least 30 min between subjects).
  - o If approved by the SRC, the next planned escalation dose (see Table 1) will be initiated. The data assessed by the SRC comprises 48 h data for 6 subjects including observation on site, short summary of phone interview (including statement about diary reports), vital signs, investigator reported local and systemic reactions, TEAEs, solicited local & systemic reactions, blood/clinical laboratory data, and brief physical examination outcome.

The maximum allowed dose for each vaccine candidate is defined in Table 1.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


For the planned dose de-escalation cohorts, 12 subjects may be dosed on one day (with intervals of at least 30 min between subjects). The doses in these cohorts in younger adults must be lower than doses that have shown acceptable tolerability in younger adults (based on the data from 12 subjects up until 48 h after the first dose). The same dose will not be administered twice, i.e., in two cohorts.

For BNT162b1 and BNT162b2, administration of the planned 10 µg dose in older subjects (Cohort 8) may start once at least a 30 µg dose has shown acceptable tolerability in younger adults (based on the data from 12 subjects up until 48 h after the boost dose).

The dose in Cohort 8 must also be confirmed by the SRC. In Cohort 8, 12 subjects will be dosed using a sentinel dosing/subject staggering (2-4-6) process with intervals of at least 1 h between the first 6 subjects and then at least 30 min intervals for the remaining 6 subjects.

For BNT162b1 and BNT162b2, administration of the planned dose escalation cohorts in older adults (Cohorts 9 and 10), 12 subjects will be dosed using a sentinel dosing/subject staggering (2-4-6) process with intervals of at least 30 min between subjects. The doses planned in these cohorts will only be administered if the dose is confirmed by the SRC.

The doses planned for Cohorts 8 to 10 are defined in Table 2.

For the unplanned dose de-escalation cohorts, i.e., where the SRC requests the use of a reduced dose for safety reasons, 12 subjects may be dosed on one day with intervals of at least 30 min between subjects (as for planned de-escalation cohorts).

Note: BNT162b1 and BNT162b2 are nucleoside modified RNAs, while BNT162a1 and BNT162c2 are both non-modified uridine containing RNAs. RNA modification is known to impact the extent of innate immune activation at a given dose level, and thus potentially the extent of reactogenicity. Therefore, tolerability data obtained with one of the vaccine variants of each of these pairs may be potentially informative for the respective other one and should be taken in consideration by the SRC for recommendations of lower or interim doses.

In the case that an individual experiences dose limiting toxicities or that the frequency or pattern of AEs within a sub-cohort gives cause for concern, the investigator may request by phone an ad hoc review by the SRC, at any time, before further doses of a given vaccine construct are administered.

#### Expansion cohorts:

Protocol amendment 6.0 implemented three additional cohorts (Cohorts 11, 12, and 13) comprising additional 150 trial subjects aged from 18 to 85 years receiving BNT162b2 only.

BNT162b2 has entered a Phase II/III evaluation of efficacy, with the intent to support an application for marketing authorization. The dosing regimen under investigation is two 30 µg BNT162b2 doses given ~21 d apart.

The expansion cohorts are intended to provide a more in-depth characterization of the adaptive immune responses induced by BNT162b2, associated vaccine safety, and the impact of factors such as subject disposition and dosing posology on humoral and cell-

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


mediated immunity. These cohorts will extend the safety data of BNT162b2 to a broader trial population and thus closer to the vaccine target population.



The planned dose of BNT162b2, two 30 µg BNT162b2 doses given 21 d apart, is the same regimen that has already been tested in the dose escalation phase of this trial and in more than 25,000 trial subjects (status 20 JAN 2021), including those with acute and chronic illnesses, in the ongoing global Phase I/II/III trial BNT162-02/C4591001 (NCT04368728). As such, all trial subjects in the three expansion cohorts can be treated in parallel.

For Cohort 13, the interval between the trial subjects for the prime and boost immunizations will be at least 30 min. For Cohorts 11 and 12, the interval between the trial subjects will be at least 15 min for the prime immunizations and at least 5 min for boost immunizations.

The three expansion cohorts (with comparable numbers of male and female subjects for each of the defined age groups, see the section Population) are as follows:

- Cohort 11: Alternative posology cohort with 30 healthy adults who will receive BNT162b2 using one 3 μg prime dose and one 30 μg boost dose of BNT162b2 given approximately 21 d apart (P/B regimen).
- Cohort 12: Adaptive immune response cohort (including safety and long term immune response) with 90 healthy adults who will receive two 30 μg BNT162b2 doses given approximately 21 d apart (P/B regimen).
- Cohort 13: Population expansion cohort (including safety and long term immune response) with 30 immunocompromised adults who will receive of two 30 μg BNT162b2 doses given approximately 21 d apart (P/B regimen).

For the scientific rationale for the expansion cohorts, see Section 4.2.

All trial site visits for subjects in the expansion cohorts will be conducted on an outpatient basis, with the clinical judgment of the investigator determining whether a period of observation beyond that required for completion of study procedures is required, on a case by case basis. Standard measures to avoid cross-contamination of immunocompromised individuals with high risk pathogens should be followed for 24 months after the primary immunization.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### Biomarker (in-depth B cell immunity to SARS-CoV-2) Cohort 14:

Protocol amendment 8.0 implements an additional cohort (Cohort 14) comprising an additional 20 healthy subjects aged from 18 to 85 years receiving BNT162b2 only. Two 30 µg BNT162b2 doses will be given approximately 21 d apart (P/B regimen).

Cohort 14 is intended to provide for additional characterization of B cell immune responses induced by BNT162b2. The planned dose of BNT162b2, two 30 µg BNT162b2 doses given 21 d apart, is the same regimen that has already been tested in the dose escalation phase of this trial and in more than 25,000 trial subjects (status 20 JAN 2021) in the ongoing global Phase I/II/III trial BNT162-02/C4591001 (NCT04368728).

For the scientific rationale for Cohort 14, see Section 4.2.

#### Part B

Due to changes in the overall clinical development plan, Part B will no longer be conducted.

### 4.1.1 Adaptive trial design elements

Dose de-escalation and escalation rules have been defined in this protocol (see Section 6.6.2).

### 4.1.2 Planned number of trial subjects

See Table 5.

## 4.2 Scientific rationale for the trial design

The trial design is based on the sponsor's experience with trials of this type and other published trials for vaccine development.

The chosen trial design reflects discussion and advice from the PEI obtained in two scientific advice meetings held in February and March 2020. At these meetings, the PEI supported the high-level design of this trial, specifically the staggered approach, single dose (single immunization dose) and P/B testing, conditional to performance of lower dose exploration if appropriate and re-consideration of the dose regimens for Part B if appropriate.

Part A of the trial is designed as a classical dose escalation, investigating the dose range which is most likely to be well tolerated and induce a virus neutralizing response. To ensure trial subject safety, a staggered approach has been chosen starting with a defined low standard dose. Use of the overlapping escalating doses in Cohorts 1 to 3, i.e., progression to initiation of dosing at the next higher dose when data is available for 6 of 12 trial subjects per group, allows a faster dose escalation while ensuring trial subject safety.

Trial subjects in Cohort 1 (with the FIH immunization), will be immunized using a sentinel dosing/staggering of subjects (EMA 2017 guidance "Strategies to Identify and Mitigate Risks for First-in-Human and Early Clinical Trials with Investigational Medicinal Products").

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


The expansion cohorts (Cohorts 11 to 13) are designed to be complementary to the ongoing global Phase I/II/III trial BNT162-02/C4591001 (NCT04368728), to demonstrate clinical efficacy and safety for two 30 µg BNT162b2 doses given ~21 d apart, which enrolled over 40,000 subjects. This Phase I/II/III trial does not include the detailed immunogenicity assessments needed to better understand the mode-of-action of the vaccine and approaches for potential improvements, e.g., in defined populations (by age, gender, immunocompromised status, certain ethnicity-associated HLA, etc.). This trial will therefore include such immunogenicity assessments, including detailed characterization of immune responses to BNT162b2 in respect of binding antibodies, neutralizing antibodies, and cell-mediated immunity (CMI), including evaluation of CD4 and CD8 T-cell responses.

Cohort 11 aims to determine whether a lower prime dose may further improve vaccine tolerability (reactogenicity), without compromising immunogenicity while exploring whether this alternative posology promotes a more favorable pattern of composite immune response modulation. A lower prime dose may further improve reactogenicity and may modulate the pattern of the composite immune response towards a more pronounced B-cell response. This alternative posology, if proven effective, could support future ring-vaccination strategies and substantial dose efficiencies. The latter could be important during the scale-up phase at the beginning of a pandemic. It has previously been demonstrated for non-RNA vaccines that an asymmetric prime-boost strategy does not adversely impact the resulting immunogenicity. The use of a lower prime dose may enable optimization of the initial CMI response, when it is most beneficial for acute patient protection, without compromising the overall humoral response. This cohort will include long term monitoring of the immune response and immune defense.

Cohort 12 is intended to complement the ongoing Phase II/III evaluation of efficacy by including assessment of the immune mechanisms induced by this unique class of vaccine. The data from this cohort addresses the expected dynamic range of inter-individual variability and could provide insights into treatment success factors and/or development strategies for future vaccine candidate design/selection for the current pandemic and future COVID-19 outbreaks. This cohort will include long term monitoring of the immune response and immune defense.

Cohort 13 will comprise immunocompromised adults, a population that has a particular risk in the current pandemic for contracting COVID-19 and for severe complications. The reactogenicity but also the immune response to BNT162b2 may be dampened in immunocompromised individuals. This cohort will show whether the immune response is indeed compromised and if yes to which extent and in which of its components and thus allow rational approaches to also serve this population of subjects. It is crucial that the priority vaccination of high risk populations is supported by data demonstrating that vaccination will be well tolerated and clinically beneficial.

BNT162b2 was selected for Phase II/III evaluation of efficacy, in part, due to its superior performance in elderly subjects, who typically demonstrate lower reactogenicity than younger subjects, but also lower levels of immunogenicity than younger subjects. The objective of Cohort 13 is to characterize the immune responses in a population with both the age-related lower immunogenicity and the lower immunogenicity linked to being immunocompromised. This knowledge could help guide future treatment optimization

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


strategies. This cohort will include long term monitoring of the immune response and immune defense.

Cohort 14 will characterize B cell and plasma cell immunity to SARS-CoV-2 after vaccination with BNT162b2. Non-clinical *in vivo* studies with BNT162b2 have indicated increased cellularity of follicular germinal centers with increased plasma cells (plasmacytosis) in regional lymph nodes after vaccination. At the onset of the COVID-19 pandemic, longitudinal studies at the DRFZ Berlin assessed the adaptive immune response of patients with severe COVID-19, using single cell transcriptomics of plasmablasts and SARS-CoV-2-specific T cells. In brief, patients with severe COVID-19 showed an immune response reflected by a continuous egress of plasmablasts into the blood. This response was driven by transforming growth factor beta (TGF- $\beta$ ), which drives B cells to produce IgA2 antibodies. None of the analyzed antibodies recombinantly produced from the plasmablasts were specific for the SARS-CoV-2 S protein, RBD, or nucleocapsid phosphoprotein.

These results suggest the immune response is initially triggered by SARS-CoV-2 but later evolved away from viral-directed immune responses, resulting in a chronic immune response producing antibodies of unknown specificity. One question is how the adaptive immune response in patients with severe COVID-19 differs from individuals in whom a productive adaptive immune response is induced by vaccination. Plasmablasts and T cells are excellent biomarkers in this context, since they can be genetically traced by their immune receptor. In addition, interactions between plasmablasts and T cells as well as the cytokine environment during their activation are reflected in gene expression at the single cell level.

Characterization of B cell and plasma cell immune responses to BNT162b2 will complement the data on T cell-mediated immunity and immunogenicity. The results may help to better understand COVID-19 as well as characterize the mode-of-action of the vaccine.

Part B of the trial will no longer be conducted due to changes in the global clinical development plan in a rapidly evolving situation.

#### 4.3 Justification for dose

Given that BioNTech proposes a rapid response scenario to a newly emerged pandemic outbreak, sufficient data is currently not available to experimentally validate the dose selection and initial starting dose. Therefore, BioNTech proposed a starting dose of 0.1  $\mu$ g (for BNT162c2), 3  $\mu$ g (for BNT162a1), and 10  $\mu$ g (for BNT162b1 and BNT162b2) in this trial based on non-clinical experience with the same RNAs encoding other viral antigens (such as influenza and HIV antigens). Based on preliminary data from this trial, as explained below, the planned doses for the BNT162a1 and BNT162c2 vaccine candidates were reduced (see Table 1).

The general safety and effectiveness of uRNA and modRNA platforms have been demonstrated in oncological clinical trials with different administration routes (RB\_0003-01 [NCT02410733], SAR441000 [NCT03871348]). Doses of up to 400 µg total uRNA administered IV as RNA lipoplex (RNA-LPX) and doses of up to 1,000 µg total naked

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


modRNA administered intratumorally, have not demonstrated signs of unpredictable overstimulation of the immune system.

The BNT162 vaccines will be administered IM as this route has been demonstrated to lead to efficient induction of antigen-specific cellular and humoral immunity and *in vivo* protein expression of comparable drug products (as shown by other companies, i.e., Moderna and CureVAC).

The doses planned in this trial were discussed with the PEI in a Scientific Advice Meeting on February 6<sup>th</sup>, 2020. At this meeting, the PEI supported the high-level design of this trial, conditional to dose exploration and, if appropriate, re-consideration of the dose regimens for Part B. This protocol reflects this advice.

As discussed in Section 2.3.1, to date, there is very limited clinical experience with BNT162 vaccines in human subjects. Reactogenicity is anticipated and considered to contribute to the mode-of-action of inducing vaccine immune responses. Initial dose ranging studies have suggested AE profiles consistent with previous usage of similar constructs in cancer patients, with AEs generally dividing into 2 groups: local injection site reactions and systemic flu-like illness.

As summarized in the BNT162 IB, to date most of the AEs reported after immunization with BNT162 vaccine candidates have been mild to moderate in intensity and no SAEs have been reported. Fever of severe intensity has been reported. Most AEs were managed with simple measures and resolved spontaneously.

Based on the available clinical and non-clinical data experience, the sponsor expects the planned maximal doses (see Table 1) to be safe.

The doses planned in this trial for older adults (i.e., adults aged between 56 and 85 years) reflect clinical data from the ongoing BNT162-01 and BNT162-02 trials with the vaccine candidates BNT162b1 and BNT162b2 in younger adults and elderly (adults aged between 65 and 85 years). After P/B dosing, these doses (10, 20, and 30 µg) showed acceptable tolerability in younger adults and in elderly adults. For details, see the BNT162 IB.

The dosing regimen planned in this trial for the expansion cohorts (Cohort 12 and 13) and Cohort 14, two 30  $\mu$ g BNT162b2 doses given ~21 d apart (P/B regimen), is the dosing regimen tested in the ongoing global Phase I/II/III trial BNT162-02. Status 20 JAN 2021, more than 25,000 trial subjects have been dosed with 30  $\mu$ g BNT162b2 P/B.

Cohort 11 will explore an alternative posology with low-dose prime (3  $\mu$ g) and standard dose boost (30  $\mu$ g) as described elsewhere.

Taken together, the planned starting doses in this trial are considered to be safe, but still sufficient to induce an antiviral immune response.

## 4.4 End of treatment (EoT) and end of trial definition

A trial subject is considered to have completed the trial if they have completed all planned visits as listed in the SoA, including all follow-up visits (see Section 1.3).

The EoT is defined as the date the last subject completed the EoT Visit (for BNT162c2 given SD Visit 6, for all cohorts with P/B dosing Visit 7).

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


The end of trial is defined as the date when the last subject completed the last planned visit given in the SoA (see Section 1.3). The trial may end earlier if there are no remaining subjects from Cohorts 11 to 13 for the 2-year follow-up period (see Table 8); subjects who receive non-trial SARS-CoV-2 vaccinations will be discontinued.

#### 5 TRIAL POPULATION

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1 Inclusion criteria

#### 5.1.1 Inclusion criteria Part A

Volunteers are only eligible to be enrolled in the trial if they meet all of the following criteria:

- 1. Have given informed consent by signing the informed consent form (ICF) before initiation of any trial-specific procedures.
- 2. They must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions (e.g., to practice social distancing and to follow good practices to reduce their chances of being infected or spreading COVID-19), and other requirements of the trial.
- 3. They must be able to understand and follow trial-related instructions.
- 4. For younger adult cohorts, volunteers must be aged 18 to 55 years, have a BMI over 19 kg/m² and under 30 kg/m², and weigh at least 50 kg at Visit 0.

OR

For older adult cohorts, volunteers must be aged 56 to 85 years, have a BMI over  $19 \text{ kg/m}^2$  and under  $30 \text{ kg/m}^2$ , and weigh at least 50 kg at Visit 0.

OR

For the immunocompromised adult cohort (Cohort 13), volunteers must be aged 18 to 85 years, have a BMI over 19 kg/m<sup>2</sup> and under 30 kg/m<sup>2</sup>, and weigh at least 50 kg at Visit 0.

5. They must be healthy, in the clinical judgment of the investigator, based on medical history, physical examination, 12-lead ECG, vital signs (systolic/diastolic blood pressure, pulse rate, body temperature, respiratory rate), and clinical laboratory tests (blood chemistry, hematology, and urine chemistry) at Visit 0.

Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 wks before enrollment, can be included.

OR

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


For the immunocompromised cohort (Cohort 13); volunteers who have previously received solid organ transplant, or peripheral blood stem cell transplantation ≥6 months after transplantation, or individuals with HIV infection with a CD4<sup>+</sup> T-cell count of ≥200 x 10<sup>6</sup>/L at Visit 0. Individuals with lower T-cell counts will be excluded from the trial on the basis that this represents a significant medical complication. In the clinical judgment of the investigator, volunteers must be immunocompromised but otherwise healthy. After consultation with the Medical Monitor, this may include individuals receiving immunosuppressant therapy due to another confounding disease at least 2 wks prior to enrollment and/or at least 6 wks following immunization with BNT162b2, and/or individuals with immunosuppressive treatment of an autoimmune disease if the disease is stable.

- 6. WOCBP must have a negative beta-human chorionic gonadotropin urine test at Visit 0 and Visit 1. Women that are postmenopausal or permanently sterilized will be considered as not having reproductive potential.
- 7. WOCBP must agree to practice a highly effective form of contraception during the trial, starting after Visit 0 and continuously until 60 d after receiving the last immunization. WOCBP must agree to require their male partners to use condoms during sexual contact (unless male partners are sterilized or infertile).
- 8. WOCBP must confirm that they practiced at least one highly effective form of contraception for the 14 d prior to Visit 0.
- 9. WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting after Visit 0 and continuously until 60 d after receiving the last immunization.
- 10. Men who are sexually active with a WOCBP and have not had a vasectomy must agree to practice a highly effective form of contraception with their female partner of childbearing potential during the trial, starting after Visit 0 and continuously until 60 d after receiving the last immunization.
- 11. Men must be willing to refrain from sperm donation, starting after Visit 0 and continuously until 60 d after receiving the last immunization.
- 12. They must have confirmation of their health insurance coverage prior to Visit 0.
- 13. They must agree to not be vaccinated during the trial, starting after Visit 0 and continuously until 28 d after receiving the last immunization.

#### 5.2 Exclusion criteria

#### 5.2.1 Exclusion criteria Part A

Volunteers are excluded from the trial if they meet or present any of the following criteria:

1. Have had any acute illness, as determined by the investigator, with or without fever, within 72 h prior to the first immunization. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the investigator, the residual symptoms will not compromise their wellbeing if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


2. Are breastfeeding on the day of Visit 0 or who plan to breastfeed during the trial, starting after Visit 0 and continuously until at least 90 d after receiving the last immunization.

- 3. Have a known allergy, hypersensitivity, or intolerance to the planned IMP including any excipients of the IMP.
- 4. Had any medical condition or any major surgery (e.g., requiring general anesthesia) within the past 5 years which, in the opinion of the investigator, could compromise their wellbeing if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments. See the inclusion criteria 5 for non-excluded medical conditions for Cohort 13.
- 5. Have any surgery planned during the trial, starting after Visit 0 and continuously until at least 90 d after receiving the last immunization.
- 6. Had any chronic use (more than 21 continuous days) of any systemic medications, including immunosuppressants or other immune-modifying drugs (except for Cohort 13) within the 6 months prior to Visit 0, unless in the opinion of the investigator the medication would not prevent, limit, or confound the protocol-specified assessments or could compromise subject safety.
  Note: Healthy volunteers with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 wks before enrollment, can be included.
- 7. Had any vaccination within the 28 d prior to Visit 0.
- 8. Had administration of any immunoglobulins and/or any blood products within the 3 months prior to Visit 0.
- 9. Had administration of another investigational medicinal product including vaccines within 60 d or 5 half-lives (whichever is longer), prior to Visit 0.
- 10. Have a known history of active or ongoing hepatitis B or hepatitis C infection; or except for Cohort 13: HIV-1 or HIV-2 infection within the 30 d prior to Visit 0.
- 11. Have a positive PCR-based test for SARS-CoV-2 within the 30 d prior to Visit 1.
- 12. Have a positive drugs of abuse (for amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, and tricyclic antidepressants) result at Visit 0 or Visit 1.
- 13. Have a positive breath alcohol test at Visit 0 or Visit 1.
- 14. Previously participated in an investigational trial involving lipid nanoparticles.
- 15. Are subject to exclusion periods from other investigational trials or simultaneous participation in another clinical trial. When entering the follow-up phase, i.e., after completing the EoT visit, subjects are allowed to participate in other clinical trials not investigating COVID-19 vaccines or treatments; subjects immunized with BNT162 vaccines in this clinical trial are allowed to participate in other clinical trials involving immunization with BNT162b2.
- 16. Have any affiliation with the trial site (e.g., are close relative of the investigator or dependent person, such as an employee or student of the trial site).

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- 17. Have a history (within the past 5 years) of substance abuse or known medical, psychological, or social conditions which, in the opinion of the investigator, could compromise their wellbeing if they participate as trial subjects in the trial, or that could prevent, limit, or confound the protocol-specified assessments.
- 18. Have a history of hypersensitivity or serious reactions to previous vaccinations.
- 19. Have a history of Guillain-Barré syndrome within 6 wks following a previous vaccination.
- 20. Have a history of narcolepsy.
- 21. Have history of alcohol abuse or drug addiction within 1 year before Visit 0.
- 22. (Except for Cohort 13) Have a history of or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination at Visit 0.
- 23. Have any abnormality or permanent body art (e.g., tattoo) that, in the opinion of the investigator, would obstruct the ability to observe local reactions at the injection site.
- 24. Have had any blood loss >450 mL, e.g., due to donation of blood or blood products or injury, within the 7 d prior to Visit 0 or plan to donate blood during the trial, starting after Visit 0 and continuously until at least 7 d after receiving the last immunization.
- 25. Have symptoms of COVID-19, e.g., respiratory symptoms, fever, cough, shortness of breath and breathing difficulties.
- 26. Have had contact with persons diagnosed with COVID-19 or who tested positive for SARS-CoV-2 by any diagnostic test within the 30 d prior to Visit 1.
- 27. Are soldiers, volunteers in detention, CRO or sponsor staff or their family members.
- 28. Regular receipt of inhaled/nebulized corticosteroids (except for Cohort 13).
- 29. For older volunteers and for Cohort 13 only: Have a condition known to put them at high risk for severe COVID-19, including those with any of the following risk factors:
  - Uncontrolled hypertension.
  - Diabetes mellitus (HbA1c >8.5% ≥3 months, according to the medical history reported by the subject).
  - Chronic obstructive pulmonary disease.
  - Asthma.
  - Chronic liver disease.
  - Known Stage 3 or worse chronic kidney disease (GFR <60 mL/min/1.73 m²);</li>
     Except for post-renal transplant patients who should have (estimated)
     GFR ≥40 mL/min/1.73 m².
  - Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies.
  - Sickle cell disease.
  - Cancer (except for Cohort 13).

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- Are immune compromised due to stem cell or organ-transplantation with significant medical complications such as acute or chronic graft rejection or graft versus host disease requiring intensive immunosuppressive treatment, transplant failure, or infectious complications or other conditions that would be considered a contraindication for vaccination.
- Are immune compromised due to HIV infection with a CD4<sup>+</sup> count of <200 x 10<sup>6</sup>/L at screening or significant medical complications such as opportunistic infections, malignant complications (e.g., lymphoma, Kaposi sarcoma), other organ manifestations consistent with advanced acquired immunodeficiency syndrome (AIDS) or other conditions that would be considered a contraindication for vaccination.
- Resident in a long term facility.
- Current vaping or smoking (occasional smoking is acceptable).
- History of chronic smoking within the prior year.

## 5.3 Lifestyle considerations

Strenuous physical activity will not be allowed on visit days. When at the trial site, trial subjects will not be allowed to smoke or to drink alcohol.

Trial subjects will be required to practice social distancing and to follow good practices to reduce their chances of being infected or spreading COVID-19, e.g., as described in the WHO guidance "Protection measures for persons who are in or have recently visited (past 14 days) areas where COVID-19 is spreading" or regional equivalents.

Trial subjects will be warned to avoid contact with persons tested positive for SARS-CoV-2 antibodies or those who have an increased risk for infection.

#### Dose ranging (Cohorts 1 to 10)

For Cohort 1 and any subsequent dose escalation cohort (in younger adults or older adults), the first 6 subjects dosed in each group will be required to remain at the site for approximately 24 h after the first immunization. The remaining trial subjects in these cohorts will be required to remain at the site for approximately 6 h after the first immunization.

For any dose de-escalation or dose-refinement cohorts, i.e., cohorts with doses lower than previously tested and found to be acceptable, trial subjects will be required to remain at the site for approximately 6 h after the first immunization.

For all cohorts with P/B dosing (irrespective of whether dose escalation, dose deescalation, or dose-refinement cohorts), all trial subjects will be required to remain at the site for approximately 6 h after the boost immunization.

#### Expansion for BNT162b2 (Cohorts 11 to 13) and Cohort 14

For Cohorts 11 to 14, all trial subjects will not be required to remain at the site beyond the time required for all trial-visit-related procedures to be completed. Care should be taken with Cohort 13 subjects (immunocompromised) to minimize the duration of site visits.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### 5.4 Screen failures

Screen failures are defined as individuals who consent to participate in the trial but who are not subsequently assigned to IMP.

A minimal set of screen failure information is required to ensure transparent reporting of screening failures to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, date the ICF was signed, the reasons for screen failures, and any serious AEs (SAEs), if applicable.

### 6 TRIAL TREATMENTS

Trial treatment is defined as any IMP intended to be administered to a trial subject according to the trial protocol. Trial treatment must be administered a physician.

#### 6.1 IMP administered

**IMP name:** BNT162 vaccines - Antiviral RNA vaccines for active immunization against COVID-19

Type: RNA-LNP vaccines utilizing different BioNTech RNA formats, i.e., uRNA (product code

BNT162a1), modRNA (two variants, product codes BNT162b1 and BNT162b2),

saRNA (product code BNT162c2)

**Dosage levels:** See Table 1, Table 2, Table 3, and Table 4. The planned dose per vaccine candidate

will not exceed the pre-defined maximum dose (see Table 1 and Table 2). The planned dose per vaccine candidate will not exceed the listed pre-defined maximum doses.

Dosage frequency:

One injection or two injections 21 d apart. Injection volumes will be up to 1.5 mL

irequericy.

**Administration** Intramuscular (IM); upper arm, musculus deltoideus. For the P/B regimens the same

**route:** arm may be used for both immunizations. The non-dominant arm is preferred.

## 6.2 Preparation/handling/storage/accountability

The preparation of solution for injection will be performed by aseptic handling procedures by pharmaceutical personnel or other trained personnel at the trial site.

For instructions on IMP (BNT162 vaccine) preparation, handling, and storage, see the Pharmacy Manual.

The investigator or a physician must confirm appropriate temperature conditions have been maintained during transit for all trial intervention received and any discrepancies are reported and resolved before use of the trial intervention.

Only trial subjects enrolled in the trial may receive IMP and only authorized site personnel may administer IMP. All IMP (and any components thereof) must be stored in a secure, environmentally controlled, and monitored (manual or automated) area in accordance with the labeled storage conditions with access limited to the investigator and authorized trial site personnel.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


The investigator, nominated site personnel, or the head of the site (where applicable) is responsible for IMP (and any components thereof) accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).

Further guidance and information for the final disposition of unused IMP (and any components thereof) is provided in the Pharmacy Manual.

## 6.3 Measures to minimize bias: randomization and blinding

Not applicable.

## 6.4 Trial treatment compliance

Trial subjects will be immunized by a physician.

The date and time of each immunization must be recorded in the source documents and recorded in the case report form (CRF). The IMP dose and trial subject identification will be confirmed at the time of administration by a member of the trial site personnel other than the person administering the IMP.

## 6.5 Concomitant therapy

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements, or other specific categories of interest) that the trial subject receives during the trial, i.e., starting after Visit 0 and until the respective EoT Visit, must be recorded along with the:

- Reason for use
- Dates of administration including start and end dates
- Dosage information including dose and frequency

Record any vaccination, including SARS-CoV-2 vaccination, received after the EoT Visit until the last FU Visit in the CRF.

The sponsor's Medical Monitor should be contacted if there are any questions regarding concomitant or prior therapy.

Trial subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), unless, in the opinion of the investigator and sponsor, the medication will not compromise their wellbeing, or could prevent, limit, or confound the protocol-specified assessments.

Trial subjects are required to agree to not be vaccinated during the trial, starting after Visit 0 and continuously until 28 d after receiving the last immunization (see the inclusion criterion 13).

Trial subjects who receive non-trial SARS-CoV-2 vaccinations will be discontinued from the BNT162-01 trial (see Section 7.2).

Nonsteroidal anti-inflammatory drugs (NSAIDs), e.g., paracetamol/acetaminophen at doses of up to 4 g/day is permitted for use any time during the trial. Other concomitant

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


medication may be considered on a case by case basis by the investigator, if required after consultation with the sponsor's Medical Monitor.

### 6.5.1 Premedication

Not applicable.

#### 6.5.2 Rescue medication

Not applicable.

#### 6.6 Dose modifications

The trial design allows for a flexible dosing which allows a better evaluation on the optimal dose range. For details, see Section 4.1.

The decision to make dose adaptions or to initiate a cohort for each vaccine will be made by the SRC (for details, see Section 10.1.5). Dose de-escalation and escalation rules have been defined in this protocol (see Section 6.6.2).

### 6.6.1 Dose limiting toxicity

#### Applicable to dose ranging cohorts only

During the time of enrollment into a given dose escalation cohort in Part A, if any of the following events occur, it will be considered an individual dose limiting toxicity and further dosing in that cohort will be stopped:

- Anaphylactic reaction considered related.
- Generalized urticaria considered related.
- Four trial subjects in that cohort with any severe unsolicited local event, if considered related and not manageable with simple measures (e.g., cooling, analgesia, nonsteroidal anti-inflammatory drugs [NSAIDs]).
- AEs within 7 d of vaccination assessed by the investigator to be potentially lifethreatening (Grade 4) and that are possibly related, or for which there is no alternative, plausible, attributable cause.
- Any systemic SAE within 7 d of vaccination that is assessed by the investigator as possibly related, or for which there is no alternative, plausible, attributable cause.
- Any fever >40.0°C (>104.0°F) within 7 d of vaccination considered related and confirmed by an investigator or medically qualified person.
- Two trial subjects (at any dose level) with the same or similar severe (Grade 3 or higher) AE (including reactogenicity reported as AEs and clinically significant laboratory abnormalities) within 7 d of vaccination, considered related, or for which there is no alternative, plausible, attributable cause (for severity grading of AEs see Section 10.3.1.7).

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


For the cohorts with BNT162c2 P/B dosing, dosing with the boost dose will only start after SRC assessment of Day 28 safety data (solicited and unsolicited) for the cohort testing BNT162c2 (SD).

Approval from the SRC will be required prior to any further dosing in the affected cohort. The SRC may call for the opening of a lower dose level cohort.

The same events will prompt IMP discontinuation for individual subjects as described in Section 6.6.4. Tasks connected to the discontinuation of IMP are described in Section 7.1.

The above guidance regulates how potential dose limiting toxicities may influence the decisions to further enroll trial subjects in any cohort. These decisions are taken by the SRC based on the 48 h safety data from the first 6 subjects of each cohort (see Section 4.1). Due to the staggered sentinel dosing design, subjects will have been followed for 4 d for the sentinel subjects when this SRC decision is made.

The above guidance also regulates how potential dose limiting toxicities may influence the decisions to enroll subjects into the next cohort for that vaccine, i.e., to progress to the next cohort. These decisions are taken by the SRC based on the 48 h safety data from all 12 subjects of each cohort (see Section 4.1). Due to the staggered sentinel dosing design, subjects will have been followed for 6 d for the sentinel subjects when this SRC decision is made.

The sum of the above events occurring at any time during the trial conduct (i.e., not just with 7 d of vaccination) will be used for the overall assessment of the candidate vaccine safety profile, i.e., to assess whether any of the observed side effects are possibly linked to vaccination.

The assessment of dose limiting toxicity should be done consistently for all subjects treated with the same treatment and dose.

In addition to data entry in the CRF, dose limiting toxicities (DLTs) will be reported within 24 h via a SAE Report Form as described in Section 10.3.1.10 and forwarded to the safety contacts listed in the same section.

## 6.6.2 Dose modification guidance/rules

#### Part A

See Section 10.1.5 for the data set upon which SRC decisions described below for Part A are made.

- The decision to test reduced or intermediate doses will be made for each vaccine independently.
- Any proposal to alter the planned escalation dose, or to test an additional deescalation dose, must be approved by the SRC.

#### Dose escalation:

 Dose escalation will only continue if the previous dose was considered safe and well tolerated by the SRC.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Any proposal to alter the planned escalation doses must be approved by the SRC.

### 6.6.3 Mitigation plans for specific AEs

Based on experience with other BioNTech RNA-based vaccines and published data from other RNA-based vaccines, it is anticipated that subjects may experience TEAEs of flu-like symptomatology following the administration of RNA vaccines due to the mechanism of action of RNA vaccines. This may include fever, chills, rigors, tachycardia, arthralgia, myalgia, headache, nausea. Treatment of these events is dependent on the discretion of the investigators; however, the following management suggestions are provided:

- Treat fever with acetaminophen or NSAIDs with a dose per trial site recommendation.
- After the first occurrence of flu-like symptomatology, subjects can be treated with standard therapeutic dose of acetaminophen, or NSAIDs, starting at least 2 h after the immunization.
- Corticosteroids should be avoided as either prophylaxis or treatment as it counteracts the effects of immunization.
- Ensure adequate hydration of trial subjects on the day of immunization. Consider administering fluids (e.g., water for drinking, 0.5 to 1.0 L) within approximately 2 h following the immunization per trial site standard.

If subjects experience enhanced respiratory disease or progression of flu-like symptomatology, such as non-resolution of the symptoms after 7 d, symptom kinetics that are inconsistent with a relationship to RNA immunization, additional diagnostic measures should be considered and the Medical Monitor should be informed.

### 6.6.4 Safety stopping criteria

See Section 6.6.1 for the list of events that must prompt discontinuation for the individual subjects.

The SRC will review and evaluate the collected safety data periodically during the trial (see Section 10.1.5 for details). A decision to stop treatment for an individual subject or to terminate the trial may be taken if safety concerns are identified by the SRC.

Suspected unexpected serious adverse reactions (SUSARs) will immediately be reviewed by the SRC. They will trigger a temporary stop of IMP administration to new subjects in the respective dose level cohort for that vaccine until the SRC recommendation to continue or to permanently stop IMP administration of new subjects in the respective dose level cohort for that vaccine.

Guidance for discontinuation of trial treatment is provided in Section 7.1.

#### 6.7 Treatment after the end of the trial

Not applicable.

7

DISCONTINUATION OF TRIAL TREATMENT AND TRIAL SUBJECT DISCONTINUATION/WITHDRAWAL


Version: 13.0

Date: 12 JAN 2022

#### 7.1 Discontinuation of trial treatment

In rare instances, it may be necessary for a trial subject to permanently discontinue IMP administration (i.e., to not receive the boost dose for groups with P/B regimens). If IMP administration is definitively discontinued, the trial subject will remain in the trial to be evaluated for safety, i.e., subjects should still complete all assessments planned in the SoA (Section 1.3).

IMP administration must be stopped if dose limiting toxicities described in Section 6.6.1 are observed.

If any of the above are observed, an unscheduled safety analysis by the SRC will be required. Trial subjects who tolerated initial vaccinations will be allowed to receive a second vaccination during this time.

In the event of discontinuation of trial treatment, it must be documented on the appropriate CRF/in the medical records whether the participant is discontinuing further receipt of trial treatment or also from trial procedures, post-treatment follow-up, and/or future collection of additional information.

### 7.1.1 Temporary discontinuation

For the Cohorts 11 to 14 (inclusive), temporary delays to the boost doses due to intercurrent illness (i.e., immunization with the boost dose within 1 wk of the scheduled day) are allowed.

### 7.1.2 Rechallenge

Not applicable.

## 7.2 Trial subject discontinuation/withdrawal from the trial

A trial subject may withdraw from the trial at any time at his/her own request, or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons.

A trial subject in Cohort 11, 12, or 13 who receives a non-trial SARS-CoV-2 vaccination will be withdrawn from follow-up and discontinued from the BNT162-01 trial.

If the trial subject withdraws consent for data processing, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.

If a trial subject withdraws from the trial, he/she may request destruction of any samples taken and not tested, and the investigator must document sample destruction in the Investigator's Site File (ISF).

If the trial subject withdraws consent or is permanently discontinued from the trial, the trial subject will be permanently discontinued both from IMP administration and from the trial at that time.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


#### If possible, permanently discontinued trial subjects will:

- Complete all assessments planned for that visit and for the EoT Visit, if discontinued on a visit day.
- Complete all assessments planned for the EoT Visit, if not discontinued on a visit day.
- Subjects permanently discontinued after the EoT Visit will be asked to complete all assessments planned for the last planned visit for that cohort as per the SoA (see Section 1.3).

## 7.3 Lost to follow-up

A trial subject will be considered lost to follow-up if they repeatedly fail to return for scheduled visits and is unable to be contacted by the trial site.

The following actions must be taken if a trial subject fails to return to the trial site for a required trial visit:

- The trial site must attempt to contact the trial subject and reschedule the missed visit as soon as possible and counsel the trial subject on the importance of maintaining the assigned visit schedule and ascertain whether or not the trial subject wishes to and/or should continue in the trial.
- Before a trial subject is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the trial subject (where possible, three telephone calls and, if necessary, a certified letter to the trial subject's last known mailing address or local equivalent methods). These contact attempts should be documented in the trial subject's medical record.
- If the trial subject continues to be unreachable, they will be considered to have withdrawn from the trial.

## 7.4 Replacement of permanently discontinued trial subjects

Permanently discontinued trial subjects will be replaced to ensure that the 12 subjects complete the trial as planned up to Visit 3 for each group unless permanently discontinued due to safety issues; in the latter cases, the SRC will decide whether to replace the discontinued trial subjects. Trial subjects permanently discontinued after Visit 3 will not be replaced.

#### 8 TRIAL ASSESSMENTS AND PROCEDURES

See the SoA (Section 1.3) for all planned time points for assessments.

Protocol waivers or exemptions are not allowed.

Immediate safety concerns should be discussed with the sponsor immediately upon occurrence or awareness to determine if the trial subject should continue or discontinue IMP administration (i.e., to administer the boost administration for groups with the P/B regimen).

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Adherence to the trial protocol requirements, including those specified in the SoA, is essential and required for trial conduct.

All screening evaluations must be completed and reviewed to confirm that potential trial subjects meet all eligibility criteria. The investigator will maintain a screening log to record details of all trial subjects screened and to confirm eligibility or record reasons for screening failure, as applicable.

For the baseline assessments (demographics, medical history), see Section 10.12.

The listed trial assessments and procedures will be updated to reflect the needs of Part B in the planned protocol amendment.

### 8.1 Efficacy assessments

Not applicable.

## 8.2 Safety assessments

Planned time points for all safety assessments are provided in the SoA (Section 1.3).

### 8.2.1 Physical examinations

Complete physical examinations will be performed at screening. Brief physical examinations will be performed at later time points including prior boost immunizations (see the SoA in Section 1.3).

- A complete physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal, and neurological systems. Height (in cm) will also be measured and recorded during complete physical examinations.
- A brief (symptom-directed) physical examination. The brief physical examination includes an overall health judgment. In-depth physical examinations are required if obvious pathological signs are visible or in the case the subject states any signs or symptoms.

### 8.2.2 Vital signs

Body temperature (in °C), pulse rate, respiratory rate, and blood pressure will be assessed at the times given in the SoA (Section 1.3). Body weight (in kg) will also be measured and recorded.

Blood pressure (systolic/diastolic, in mmHg) and pulse (in bpm) measurements will be assessed while the trial subject is in a supine position/at rest. If available, a completely automated device should be used, otherwise manual techniques can be used. The same method of measurement should be used for the trial subject during the course of the trial.

Blood pressure and pulse measurements should be preceded by at least 5 min of rest for the trial subject in a quiet setting without distractions (e.g., television, cell phones).

Vital signs should be taken before any blood collection.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### 8.2.3 Electrocardiograms

Standard 12-lead ECGs will be recorded at the times given in the SoA (Section 1.3) using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc; according to Bazett) intervals.

ECGs will be judged by the investigator as clinically significant (yes/no); only the investigator assessment and heart rate will be recorded in the CRF.

### 8.2.4 Clinical laboratory tests

See Section 10.2 for the list of clinical laboratory tests to be performed at the times given in the SoA (Section 1.3).

The investigator must review the laboratory report, document this review with signature and date, and record any clinically relevant changes occurring during the trial in the AE section of the CRF.

All laboratory tests with values considered clinically significantly abnormal during participation in the trial should be repeated until the values return to normal or baseline or are no longer considered clinically significant by the investigator or the sponsor's Medical Monitor.

If such values do not return to normal/baseline within a period of time judged reasonable by the investigator, the etiology should be identified and the sponsor notified.

All protocol-required clinical laboratory tests (see Section 10.2) must be conducted in accordance with the trial site standard.

If laboratory values from non-protocol-specified laboratory assessments performed at the laboratory require a change in trial subject management or are considered clinically significant by the investigator (e.g., SAE, AE or dose modification), then the results must be recorded in the CRF.

### 8.2.5 Drugs of abuse screening

Screening for drugs of abuse (amphetamines, benzodiazepines, barbiturates, cocaine, cannabinoids, opiates, methadone, methamphetamines, phencyclidine, and tricyclic antidepressants) will be performed using a commercially available kit at the times given in the SoA (Section 1.3).

### 8.2.6 Testing for alcohol use

Breath testing for alcohol use will be performed at the times given in the SoA (Section 1.3).

### 8.2.7 Viral screening (for blood-borne viruses)

The screen will test for: hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibodies, and HIV-1 and HIV-2 antibodies. For SARS-CoV-2 testing, see Section 8.2.10.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


## 8.2.8 Subject diaries

Trial subjects will be given subject diaries at Visit 1 and be asked to record any reactions between visits, solicited local reactions at the injection site (pain, tenderness, erythema/redness, induration/swelling) and solicited systemic reactions (nausea, vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, loss of appetite, malaise, and fever [i.e., ≥38°C]).

Subject diaries may include App-supported electronic documentation in compliance with the applicable data protection regulations.

Trial site personnel will collect subject diaries at the visits given in the SoA (Section 1.3).

### 8.2.9 Assessment of local reactions

Local reactions after IM immunization will be assessed by the investigator at the times given in the SoA (Section 1.3). This information will be used to validate the solicited assessment of local reactions in the patient diary and potentially support AE reporting.

Local reactions (both investigator assessed and solicited in the subject diaries) will be graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" for "Local Reaction to Injectable Products" (see the section "Assessment of intensity" in Section 10.3.1.11).

### 8.2.10 SARS-CoV-2 testing

SARS-CoV-2 testing (PCR-based and antibody-based) will be performed at the time points provided in the SoA (Section 1.3).

This includes PCR-based testing for SARS-CoV-2 as an eligibility criterion and blood draws for anti-SARS-CoV-2 antibody testing as baseline reference for immunogenicity analysis.

If required, this reference will allow the discrimination between vaccinated and infected subjects.

The screen for SARS-CoV-2 by PCR-based test using oral swipe sample can be performed by either a central laboratory or a "point of care" device at the trial site.

- If a central laboratory is used: Only the SARS-CoV-2 status will be tested and no further data will be generated.
- If a point of care device is used: The most commonly used devices come with predefined test panels that test for a range of pathogens and not just for SARS-CoV-2. Thus, inevitably and automatically, incidental data for the pathogens other than SARS-CoV-2 will be generated when using such devices. Since this incidental data is not required by this trial, only the results for SARS-CoV-2 will be recorded in the CRF, analyzed, and reported as described in this protocol. If a test result for SARS-CoV-2 or another pathogen must be reported to relevant authorities, this notification will be done by the trial site.
## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


The anti-SARS-CoV-2 antibody testing will be performed with a commercially available antibody test. In case this commercial antibody test can, discriminate between vaccine-specific and infection-specific antibody responses (based on the antigens used), it will be used to test subjects who may have experienced enhanced respiratory disease or progression of flu-like symptomatology, such as non-resolution of the symptoms after 7 d, symptom kinetics that are inconsistent with a relationship to RNA immunization, as might be expected with a COVID-19 disease (see Section 6.6.3).

In these cases, ad hoc anti-SARS-CoV-2 antibody testing will be performed to test for the development and presence of SARS-CoV-2-specific antibodies, ideally at approximately 14 d and 28 d after the last immunization with the BNT162 candidate vaccine. This data will be used to evaluate the development and progression of an antibody response allowing the diagnosis of a manifest infection.

In case this commercially available test cannot discriminate between vaccine-specific and infection-specific antibody responses, the same kind of analysis will be performed with a custom-made assay specifically developed by the CRO.

### 8.2.11 Subject hotline

Subjects will be provided with contact details for a Subject Hotline, which can be used to contact the trial site during their participation in the trial should they require guidance or should they experience any symptoms of illness. The reporting of any symptoms of illness, e.g., flu-like symptoms, may trigger diagnostic measures (including ad hoc site visits) at the discretion of the investigator. For guidance for specific AEs, see Section 6.6.3.

### 8.2.12 Subject wellbeing questioning

Structured non-leading subject wellbeing questioning will be performed at the times given in the SoA (Section 1.3). Subject responses may trigger more in-depth questioning on specific topics, and may trigger diagnostic measures (including ad hoc site visits) at the discretion of the investigator.

### 8.2.13 Assessment of systemic reactions

Systemic reactions after IM immunization will be assessed via daily solicited reports in the subject diaries and at the times given in the SoA (Section 1.3).

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Systemic reactions will be graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" for "Systemic reaction grading scale" (see the section "Assessment of intensity" in Section 10.3.1.11).

#### 8.3 Adverse events and serious adverse events

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible for following up all AEs and SAEs.

## 8.3.1 Time period and frequency for collecting AE and SAE information

For Cohorts 1 to 10, all AEs and SAEs will be collected from the date of subject consent until discharge from the trial only IMP-related AEs and any SAEs will be collected.

For Cohorts 11 to 13 and 14, all AEs and SAEs will be collected from the date of subject consent until Visit 7 (the EoT Visit). From Visit 7 through 9 only IMP-related AEs, SAEs, and SARS-CoV-2 infections will be collected. After Visit 9 (e.g., Visits 10, 11, and 12) until the last scheduled FU Visit (i.e., when the subject is discharged from the trial), any SARS-CoV-2 infections and SAEs will be collected.

For subjects in Cohorts 11 to 13 who receive a non-trial SARS-CoV-2 vaccination, AEs/SAEs will be collected as specified above until the date when the subject was vaccinated with the non-trial SARS-CoV-2 vaccine. The AEs expected to be captured after non-trial SARS-CoV-2 vaccination are within the frame of post-marketing safety data reporting.

All SAEs (initial and follow-up reports) will be recorded and reported to the sponsor or designee within 24 h after becoming aware of the event, as indicated in Section 10.3.1.10.

Investigators are not obligated to actively seek AEs or SAEs after conclusion of the trial participation. However, if the investigator learns of any SAE, including a death, at any time after a trial subject has been discharged from the trial, and he/she considers the event to be reasonably related to the IMP administration or trial participation, the investigator must promptly notify the sponsor.

#### 8.3.2 Method of detecting AEs and SAEs

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Section 10.3.

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the trial subject is the preferred method to inquire about AE occurrences.

## 8.3.3 Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each trial subject at subsequent visits/contacts. All AEs/SAEs/DLTs will be followed until resolution, stabilization, the event is otherwise explained, or the trial subject is lost to follow-up (as

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


defined in Section 7.3). Further information on follow-up procedures is provided in Section 10.3.1.7.

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the sponsor to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other healthcare professionals.

New or updated information will be recorded in the originally completed CRF.

The investigator will submit any updated SAE data to the sponsor within 24 h of receipt of the information as indicated in Section 10.3.1.10.

All ongoing AEs/SAEs will be followed until resolution, considered by the investigator to be stable or chronic (resolved with sequelae), the trial subject is lost to follow-up or the trial subject withdraws consent. If no final status is reached by the time of discharge from the trial, the investigator must confirm the unavailability of a final status.

## 8.3.4 Regulatory reporting requirements for SAEs

Prompt notification of an SAE by the investigator to the sponsor is essential so that legal obligations and ethical responsibilities towards the safety of trial subjects and the safety of a trial treatment under clinical investigation are met.

The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a trial treatment under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, Independent Ethics Committees (IECs), and investigators. The execution of expedited reporting to the different entities may be delegated as detailed in the trial Safety Management Plan.

Safety reports will be prepared for SUSARs according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.

For the IMP, it is the sponsor's or delegate's responsibility to perform SUSAR reporting to the regulatory authority, the IEC and the other investigators as required by national law and applicable guidelines.

An investigator who receives an investigator safety report describing an SAE or other specific safety information (e.g., summary or listing of SAEs) from the sponsor should review it and then file it together with the IB. If required by local requirements, the investigator will notify the relevant IEC.

#### 8.3.5 Pregnancy

For WOCBP, urine pregnancy tests will be performed using a commercial kit at the times given in the SoA (see Section 1.3).

Pregnancy information will only be collected after obtaining written informed consent from the pregnant female subject (or if a male subjects' partner becomes pregnant, written informed consent from both).

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Pregnancy information will be collected for pregnancies that occurred after the date of the first dose of trial treatment until 60 d after the last dose of trial treatment for pregnant subjects (or until 60 d after the last immunization of the male subject for pregnant female partners).

If a pregnancy is reported, the investigator should inform the sponsor within 24 h of learning of the pregnancy and should follow the procedures outlined in Section 10.4.

Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs.

#### 8.3.6 Death events

Any death that occurs within the observation period will be reported as an SAE.

In case of a fatal event, the event term should not be "death" but the underlying event which led to death (death = outcome). If there is more than one AE in a fatal case, only for the AE leading to death the outcome "fatal" should be selected. If the cause of death is unknown and cannot be ascertained at the time of reporting, "unexplained death" should be documented as event term.

## 8.3.7 Disease-related events and/or disease-related outcomes not qualifying as AEs or SAEs

Not applicable, this trial will only enroll healthy trial subjects.

#### 8.3.8 Adverse events of special interest

Enhanced respiratory disease or flu-like symptomatology not resolved after 7 d or with symptom kinetics that are inconsistent with a relationship to RNA immunization will be considered adverse events of special interest (AESI).

#### 8.4 Treatment of overdose

Any dose of trial treatment above the planned dose specified in this protocol will be considered an overdose.

The sponsor does not recommend specific treatment for an overdose.

In the event of an overdose, the investigator should:

- Contact the sponsor's Medical Monitor immediately.
- Closely monitor the trial subject for any AE/SAE and laboratory abnormalities (at least for 7 d).
- Document the quantity of the excess dose as well as the duration of the overdose in the CRF.

Decisions regarding dose interruptions or modifications will be made by the investigator in consultation with the sponsor's Medical Monitor based on the clinical evaluation of the trial subject.


#### 8.5 Pharmacokinetics

Not applicable.

## 8.6 Pharmacodynamics

Not applicable.

#### 8.7 Genetics



## 8.8 Biomarkers (CMI responses, explorative biomarker, immunogenicity research purposes)

Blood draws will be taken at the times listed in the SoA (Section 1.3) for explorative biomarker/immunogenicity research purposes, these will be in addition to standard trial assessments in selected dose ranging cohorts, and as core elements of the assessments of the expansion cohorts.



In addition, samples may be stored and analysis may be performed on biomarker variants thought to play a role in the mechanism of action of BNT162 to evaluate their association with observed clinical responses to BNT162. Furthermore, samples may be used for research to develop methods, assays, prognostics and/or companion diagnostics related to BNT162.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Samples for biomarker analysis will be retained for use for up to 5 years after the end of the trial. The tube with the sample will be labeled with a number (optionally also with a bar code) to keep the subject's identity confidential; the tube label will not include information that could be used to identify the subject. Results of the blood analyses will be linked to the clinical information collected during the trial using this specific number. The analysis will only be carried out on the basis of the label data and samples. Biomarker samples and all data generated using the samples, will be handled in accordance with applicable laws and regulations; this includes requirements applicable for data protection, for sample shipment outside Germany, and a potential withdrawal of consent.

Blood samples will only be used for biomarker analysis if the trial subjects have provided informed consent for this biomarker analysis.

## 8.9 Biomarkers (B cells)

Blood draws to characterize B cell and plasma cell immunity to SARS-CoV-2 will be taken at the times listed in the SoA (Section 1.3) for explorative biomarker/immunogenicity research purposes. These will be in addition to standard trial assessments already performed in selected dose ranging cohorts and the expansion cohorts.



In addition, samples may be stored and analysis may be performed on biomarker variants thought to play a role in the mechanism of action of BNT162b2 to evaluate their association with observed clinical responses to BNT162b2. Furthermore, samples may be used for research to develop methods, assays, prognostics, and/or companion diagnostics related to BNT162b2.

Samples for biomarker analysis will be retained for use for up to 5 years after the end of the trial. The tube with the sample will be labeled with a number (optionally also with a bar code) to keep the subject's identity confidential; the tube label will not include information that could be used to identify the subject. Results of the blood analyses will be linked to the clinical information collected during the trial using this specific number. The analysis will only be carried out on the basis of the label data and samples. Biomarker samples and all data generated using the samples, will be handled in accordance with applicable laws and regulations; this includes requirements applicable for data protection, for sample shipment outside Germany, and a potential withdrawal of consent.

Blood samples will only be used for biomarker analysis if the trial subjects have provided informed consent for this biomarker analysis.


## 8.10 Immunogenicity assessments

Immune responses as laid down in the trial objectives will be assessed at the times listed in the SoA (Section 1.3) using:

- 1) A functional antibody titer determined, e.g., via virus neutralization test (VNT) or an equivalent assay.
  - Seronegative is defined as titers below the starting dilution (i.e., below the limit of detection of the assay).
  - Seroconversion after immunization is defined as a 4-fold increase in titer.
    - o for seronegative pre-immunization sera: a titer ≥4 times the limit of detection.
    - for seropositive pre-immunization sera: a titer which is 4-fold higher than the measured pre-immunization titer.
- 2) An antibody binding assay, e.g., enzyme-linked immunosorbent assay (ELISA) or an equivalent assay.
  - Seroconversion after immunization is defined as a 4-fold increase in titer/antibody concentration.



## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01




Instructions on the sample collection, handling, and shipping will be provided in a Laboratory Manual. The methodology used for these assessments will be documented in the Biomarker Manual.

Leftover blood after completion of the immunogenicity assessments may be used for additional analyses as described in Section 8.7 (Genetics) and/or Section 8.8 (Biomarkers).

Blood samples will only be used for additional analyses if the trial subjects have provided informed consent for these additional analyses.

#### 8.11 Blood collection

For subjects in Cohorts 1 to 10, up to approximately 592 mL blood will be drawn per subject over the complete trial, i.e., over approximately 223 d.

For subjects in Cohorts 11 to 13, up to approximately 1,025 mL blood will be drawn per subject over the complete trial, i.e., over approximately 760 d.

For subjects in Cohort 14, up to approximately 477 mL blood will be drawn per subject over the complete trial, i.e., over approximately 223 d.

Additional blood samples may be taken, e.g., for safety assessments after AEs or SAEs.

For enrolled subjects who have not completed the EoT Visit (see the SoA in Section 1.3) before approval of protocol amendment 04, the optional additional blood draws added by protocol amendment 04 will only apply for subjects who give consent.

#### 8.12 Saliva and stool collection

For subjects in Cohort 14, saliva and stool will be collected as shown in the SoA in Section 1.3.


#### 9 STATISTICAL CONSIDERATIONS

## 9.1 Statistical hypotheses

There is no formal statistical hypothesis under test.

## 9.2 Sample size determination

No formal sample size calculations have been performed.

For Part A, the inclusion of 12 subjects per group is considered to be adequate for a safety assessment of each vaccine per dose level. The probability to observe a particular TEAE with incidence of 15% at least once in 12 subjects per group is 85.8%.

For the expansion cohorts the probability to observe a particular TEAE with incidence of 5% at least once in 30 and 90 subjects per group, respectively, is 78.5% and 99.0% respectively (see Table 10).

Table 10: Probability to observe a particular TEAE at least once

| Number of subjects | TEAE incidence | Probability to observe a particular TEAE at least once |
|---|---|---|
| 12 | 15% | 85.8% |
| 30 | 15% | 99.2% |
| | 10% | 95.8% |
| | 5% | 78.5% |
| 90 | 15% | >99.9% |
| | 10% | >99.9% |
| | 5% | 99.0% |

TEAE = treatment-emergent adverse event.

## 9.3 Analysis sets

The following analyses sets are defined:

| Analysis set | Description |
|---|---|
| Screened Set | The Screened Set is defined as all subjects who signed informed consent. |
| Safety Set | The Safety Set is defined as all subjects who received at least one dose of IMP. |

## 9.4 Statistical analyses

Statistical analyses will be performed by BioNTech or a designated CRO. All statistical analyses will be carried out using SAS®, Version 9.3 or higher, and/or other statistical software as required.

The statistical analysis plan (SAP) will be finalized prior to database snapshot for the primary analysis and it will include a more technical and detailed description of the

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


statistical analyses described in this section. Any deviations from the planned analyses described in the final SAP will be described and justified in the clinical trial report.

This section gives a summary of the planned statistical analyses of the most important endpoints including primary and key secondary endpoints.

#### 9.4.1 General considerations

In general, data will be summarized by groups and groups may be combined as appropriate.

Continuous variables will be summarized by group using the following descriptive statistics: number of subjects (n), mean, standard deviation, median, minimum, and maximum.

Categorical variables will be summarized by group presenting absolute and relative frequencies (n and %) of subjects in each category.

Baseline is defined as last available value prior to first dose of IMP.

### 9.4.2 Primary endpoints

The primary endpoints are defined in Section 3.

All AEs will be coded using the most recent version of Medical Dictionary for Regulatory Activities (MedDRA®) coding system to get a system organ class (SOC) and preferred term (PT) for each AE.

Treatment-emergent AEs (TEAEs) are defined in Section 10.3.1.1 and will be summarized using the Safety Set. In general, AEs will be analyzed by group (i.e., by type [BNT162a1, BNT162b1, BNT162b2, BNT162c2 SD, and BNT162c2 P/B] and dose level) and for each immunization, i.e., for:

- Prime immunization up to 7 d after initial immunization
- Prime immunization up to boost immunization or 28 d after initial immunization (whatever comes first)
- Boost immunization up to 7 d after boost immunization (only for P/B regimens)
- Boost immunization up to 28 d after boost immunization (only for P/B regimens)
- Prime immunization up to 28 d after boost immunization or after prime immunization (if no boost was given)

Additionally, AEs will be summarized for all dose levels combined for each type.

For each analysis, the number and percentage of subjects reporting at least one AE will be summarized by PT nested within SOC for each of the following AE types using the Safety Set:

- Any AE
- Any AE excluding AEs based on solicited reporting via subject diaries
- Related AE

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- Grade ≥3 AE
- Related Grade ≥3 AE
- Any SAE
- Related SAE

Moreover, the number and percentage of subjects with any AE will be summarized by worst grade by PT nested within SOC.

Local reactions and systemic reactions will be graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" (see Section 10.3.1.11).

For each immunization, the number and percentage of subjects reporting at least one local reaction or systemic reaction (i.e., solicited data collected using subject diaries) will be summarized for each of the following types using the Safety Set:

- Any local reactions or systemic reactions
- Grade ≥3 local reactions or systemic reactions

The analysis of local and systemic reactions will be repeated with a reduced set of terms (called the "comparability analysis"), to facilitate like-for-like comparisons between different trials in the clinical development program for BNT162 vaccines.

Moreover, the number and percentage of subjects reporting at least one local reaction will be summarized by worst grade using the Safety Set.

### 9.4.3 Secondary endpoints

The secondary endpoints are defined in Section 3.

The binary secondary endpoints will be summarized by group presenting absolute and relative frequencies (n and %) of subjects in each category for each assessment. The continuous secondary endpoints will be summarized by group using summary statistics. The scheduled time points for assessment are given in the SoA (see Section 1.3).

### 9.4.4 Exploratory endpoints

The exploratory endpoints are defined in Section 3. Exploratory analyses will be described in the SAP.

#### 9.4.5 Other safety analyses

Safety data other than AEs that will be summarized includes clinical laboratory parameters, vital signs, and ECGs. All safety analyses will be based on the Safety Set and will be summarized descriptively by group unless otherwise stated.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


## **Clinical laboratory parameters**

The clinical laboratory parameters to be summarized and assessed are listed in Section 10.2. The scheduled time points for assessment are given in the SoA (see Section 1.3).

Clinical laboratory parameters at each time point and change from baseline to each postbaseline time point will be summarized using descriptive summary statistics for each parameter by group.

Shift tables from baseline to worst intensity grade will be provided for each laboratory parameter by group.

Additionally, the occurrence of clinically significant abnormal laboratory results within a trial subject will be analyzed using descriptive summary statistics for each parameter and visit by group.

Abnormal laboratory results will be graded using criteria based on the guidance given in US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" (see Section 10.3.1.11).

Laboratory parameter results will be listed along with the normal ranges. Values that are below or above the normal ranges will be flagged.

Clinical laboratory analysis details will be described in the SAP.

### Vital signs

The vital sign parameters to be summarized and assessed are given in Section 8.2.2. The scheduled time points for assessment are given in the SoA (see Section 1.3).

Vital sign parameters at each time point and change from baseline to each post-baseline time point will be summarized using descriptive summary statistics for each parameter by group.

#### **ECG**

ECG parameters to be summarized and assessed are given in Section 8.2.3. The scheduled time points for assessment are given in the SoA (see Section 1.3).

ECGs will be judged by the investigator as clinically significant (yes/no).

#### 9.4.6 Other analyses

Other analyses will be described in the SAP.

## 9.5 Interim analyses

The final analysis will be performed once all subjects have completed the EoT Visit as defined in Section 1.3. An analysis update will be performed once all subjects will have completed the last planned visit. No formal interim statistical analysis will be performed. However, preliminary analyses based on all data collected until a pre-defined data cut-off date (snapshot analyses) may be performed for each cohort once subjects within a cohort will have been followed up for at least 7 d following each dose.

 Version: 13.0

Date: 12 JAN 2022

#### 9.6 **Data Monitoring Committee**

A DMC is not planned. An SRC is planned, for details see Section 10.1.5.

#### 10 SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

#### 10.1 Regulatory, ethical, and trial oversight considerations

This trial will be conducted in according to this protocol, the ethical principles that have their origin in the Declaration of Helsinki, Good Clinical Practice (GCP), and applicable regulatory requirements.

#### Regulatory and ethical considerations 10.1.1

This trial will be conducted in accordance with the protocol and with the following:

- Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) international ethical guidelines
- Applicable GCP guidelines
- Applicable laws and regulations

The protocol, protocol amendments, ICF, IB, and other relevant documents (e.g., advertisements) must be submitted to an IEC and reviewed and approved by the IEC before the trial is initiated.

Any amendments to the protocol will require IEC approval before implementation of changes made to the trial design, except for changes necessary to eliminate an immediate hazard to trial subjects.

The coordinating investigator or delegate will be responsible for the following:

- Providing written summaries of the status of the trial to the IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IEC.
- Notifying the IEC of SAEs or other significant safety findings as required by IEC procedures.
- Providing oversight of the conduct of the trial at the site and adherence to requirements of ICH guidelines, the IEC, European regulation 536/2014 (if applicable), and all other applicable local regulations.

The principal investigator, any investigator(s), the sponsor, or personnel at other establishments must cooperate with any inspection of the documents, facilities, records, and other resources deemed appropriate by the inspecting authorities to be related to the trial and that may be located at the trial site, at the sponsor, or at other establishments.

The sponsor must be notified as soon as possible about any upcoming regulatory authority inspection.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


#### 10.1.2 Financial disclosure

All investigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the trial and for 1 year after completion of the trial.

### 10.1.3 Informed consent process

Informed consent must be obtained before any trial-specific screening procedure is performed.

The investigator or his/her representative will explain the nature of the trial to the trial subject and answer all questions regarding the trial.

Trial subjects must be informed that their participation is voluntary.

Trial subjects will be required to sign a statement of informed consent that meets the requirements of local regulations, ICH guidelines, Health Insurance Portability and Accountability Act (HIPAA) requirements, where applicable, and the IEC or trial site.

The medical record must include a statement that written informed consent was obtained using a sponsor-approved ICF before the trial subject was enrolled in the trial and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.

Trial subjects must be re-consented to the most current version of the ICF during their participation in the trial.

Informed consent will be obtained for the use of residual biosamples collected for further explorative investigations of the immune response in healthy adults after SD or P/B immunization, e.g., using new assays that become available after completion of trial conduct.

#### 10.1.4 Data protection

Trial subjects will be assigned a unique identifier by the investigator according to the sponsor specifications on unique identifier assignment. Any trial subject records or datasets that are transferred to the sponsor will contain the identifier only; trial subject names or any information which would make the trial subject identifiable will not be transferred.

Trial subjects must be informed that his/her personal trial-related data will be used by the sponsor in accordance with local data protection laws. The level of disclosure must also be explained to the trial subject who will be required to give consent for their data to be used as described in the informed consent.

Trial subjects who withdraw consent must be informed that the data collected up until consent was withdrawn will still be used by the sponsor as described in the ICF.

Trial subjects who withdraw consent must be informed that, unless they agree otherwise, any biosamples collected will be destroyed.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Trial subjects must be informed that their medical records may be examined by sponsor Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IEC members, and by inspectors from regulatory authorities.

#### 10.1.5 Committees - SRC

For Part A, the SRC will be comprised by a sponsor medical representative, the Medical Monitor, a sponsor-independent investigator, and a site representative.

Key roles of the SRC are as follows:

- <u>Before progression to the next cohort</u>, for each vaccine per cohort/dose level, assess the data, decide whether to approve initiation of the next cohort/dose level and to confirm the planned dose or define another dose for use. The data assessed by the SRC is defined in Section 1.1.
- After completing its evaluation of the 48 h data for the first 6 subjects per group in cohort, the SRC may request a prolongation of the observation period to up to Day 7 data for later cohorts or other similar adaptions to protect subject wellbeing.
- <u>Throughout the trial</u>, assess whether to replace trial subjects permanently discontinued due to safety issues.
- <u>Throughout the trial</u>, approval from the SRC will be required prior to resuming any dosing in a "stopped" cohort (see Section 6.6.1). The SRC may call for the opening of a lower dose level cohort.
- SRC may make recommendations on increasing the length of the observation periods and additional subject wellbeing calls may be included at the discretion of the SRC.

The SRC will act according to its own written procedures described in a charter, and will prepare written minutes of its meetings.

#### 10.1.6 Dissemination of clinical trial data

A final clinical trial report integrating all trial results will be prepared by the sponsor.

This trial will be registered and trial results be posted on publicly accessible trial registries (e.g., the EU Clinical Trial Register) in accordance with the applicable regulations.

#### 10.1.7 Data quality assurance

All trial subject data relating to the trial will be recorded in a CRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by signing the CRF.

The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.

The investigator must permit trial-related monitoring, audits, IEC review, and regulatory agency inspections and provide direct access to source data documents.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Monitoring details describing strategy (e.g., risk-based initiatives in operations and quality, such as risk management and mitigation strategies and analytical risk-based monitoring), methods, responsibilities and requirements, including handling of non-compliance issues and monitoring techniques (central, remote, or on site monitoring) are provided in the Monitoring Plan.

The sponsor or designee is responsible for the data management of this trial including quality checking of the data.

The sponsor assumes accountability for actions delegated to other parties (e.g., CRO).

Trial monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of trial subjects are being protected; and that the trial is being conducted in accordance with the currently approved protocol and any other trial agreements, GCP, and all applicable regulatory requirements.

Records and documents, including signed ICFs, pertaining to the conduct of this trial must be retained by the investigator for 25 years after trial completion unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor.

#### 10.1.8 Source documents

Source documents provide evidence for the existence of the trial subject and substantiate the integrity of the data collected. Source documents are filed in the ISF.

Data entered in the CRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the trial. Also, current medical records must be available.

Source data are all information in original records and certified copies of original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Source data are contained in source documents (original records or certified copies).

Source documents are original documents, data, and records (e.g., hospital records, clinical and office charts, laboratory notes, memoranda, subject diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate copies, microfiches, photographic negatives, microfilm or magnetic media, x-rays, subject files, and records kept at the pharmacy, at the laboratories and at medico-technical departments involved in the clinical trial).

#### 10.1.9 Trial and site start and closure

The trial start date is the date on which the trial will be open for enrollment of trial subjects.

The sponsor designee reserves the right to close the trial site or terminate the trial at any time for any reason at the sole discretion of the sponsor. Trial sites will be closed upon trial

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


completion. A trial site is considered closed when all required documents and trial supplies have been collected and a trial site closure visit has been performed.

The investigator may initiate trial site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a trial site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IEC or local health authorities, the sponsor's procedures, or GCP guidelines.
- Inadequate recruitment of trial subjects by the investigator.
- Discontinuation of further trial treatment development.

If the trial is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the IECs, the regulatory authorities, and any CROs used in the trial of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the trial subject and should assure appropriate follow-up.

### 10.1.10 Publication policy

The results of this trial may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This will allow the sponsor to protect proprietary information and to provide comments.

The sponsor will comply with the requirements for the publication of trial results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multi-site trials only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors (ICMJE) authorship requirements.

## 10.1.11 Protocol preparation and approval

This protocol has been prepared, reviewed and approved, including wet ink sign-off by the sponsor's responsible person, in accordance with the sponsor's standard operating procedures. Documentation of this process is filed in the TMF.

## 10.2 Clinical laboratory tests

Blood will be drawn and urine will be collected for clinical laboratory tests at the times given in the SoA (Section 1.3).

#### Hematology

Hemoglobin, hematocrit, red blood cell count, white blood cell count and differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


## **Clinical chemistry**

Alkaline phosphatase, creatinine, ferritin, C-reactive protein, albumin, alanine aminotransferase, amylase, aspartate aminotransferase, gamma glutamyl transpeptidase, total bilirubin, blood urea nitrogen, glucose, lipase, sodium, potassium, calcium.

Follicle stimulating hormone: Only in women who are not of childbearing potential.

#### **Urinalysis**

<u>Dipstick</u>: glucose, bilirubin, ketone, specific gravity (1 mL  $\triangleq$  1 g), blood, pH, protein, urobilinogen, nitrite, and leukocytes.

<u>Microscopic urinalysis</u>: If warranted by dipstick results, urine sediment will be microscopically examined for presence of red blood cells, white blood cells, casts, crystals, epithelial cells, and bacteria.

## 10.3 Adverse events: Definitions and procedures for recording, evaluating, follow-up, and reporting

#### 10.3.1 Definition of AE and TEAE

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  - NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding that is clinically significant), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.
- Events after signing ICF and before IMP administration will be handled as AEs.
- A TEAE is defined as any AE with an onset date on or after the first administration
  of IMP (if the AE was absent before the first administration of IMP) or worsened
  after the first administration of IMP (if the AE was present before the first
  administration of IMP). AEs with an onset date more than 28 d after the last
  administration of IMP will be considered as treatment-emergent only if assessed as
  related to IMP by the investigator.

## 10.3.1.1 Events <u>meeting</u> the AE definition

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis)
  or other safety assessments (e.g., ECG, radiological scans, vital signs, physical
  examination, measurements), including those that worsen from baseline, and which
  are considered clinically significant in the medical and scientific judgment of the
  investigator, may be considered as AEs.
- Reactogenicity need only be reported as an AE if doing so provides clinically significant information not available elsewhere (such as the solicited reactions listings), e.g., severe reactogenicity lasting longer than the period of solicitation of symptoms in the subject diary. Diagnostic AEs for local and/or systemic

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


reactogenicity, e.g., "injection site reaction" or "flu-like illness", should generally be preferred over AEs reporting of individual signs and symptoms.

- New conditions or (at the discretion of the investigator) any worsening of a preexisting condition detected or diagnosed after Visit 0.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either trial treatment or a concomitant medication. Overdose *per se* will not be reported as an AE/SAE.

## 10.3.1.2 Events <u>not meeting</u> the AE definition

- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).

### 10.3.1.3 Suspected adverse reactions

All untoward and unintended responses to an IMP-related to any dose administered.

- The definition also covers medication errors and uses outside what is foreseen in the protocol, including misuse and abuse of the IMP.
- The definition implies a reasonable possibility of a causal relationship between the event and the IMP. This means that there are facts (evidence) or arguments to suggest a causal relationship.

#### 10.3.1.4 Definition of SAE

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under trial, death due to progression of disease).

An SAE is defined as any untoward medical occurrence that, at any dose:

- Results in death
- Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the trial subject was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it were more severe.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- Requires trial subject hospitalization or prolongation of existing hospitalization
  - In general, hospitalization signifies that the trial subject has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or out trial subject setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.
- Results in persistent disability/incapacity:
  - This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.
- Is a congenital anomaly or a birth defect.
- Other situations:
  - Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the trial subject or may require medical or surgical treatment to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.

## 10.3.1.5 Suspected unexpected serious adverse reactions (SUSARs)

All suspected adverse reactions related to an IMP (the tested drugs and comparators) that occur in this trial, and that are both unexpected and serious are SUSARs. SUSARs are subject to expedited reporting.

#### 10.3.1.6 Use of the terms "severe" and "serious"

Severity and seriousness need to be assessed independently for each AE recorded on the CRF.

SAEs must be reported by the investigator to the sponsor immediately (i.e., no more than 24 h after learning of the event; see Section 10.3.1.10 for reporting instructions).

### 10.3.1.7 Recording and follow-up of AE and/or SAE

#### AE and SAE recording

The investigator needs to assess and document any AE regardless of association with the use of the trial treatment during the period of observation (starting from Visit 0 until 21 d after the last immunization or trial subject discharge from the trial, whichever one is later). To ensure trial subject safety during the trial, safety will be monitored from Visit 0 (screening) until at least (approximately) 6 months after the last immunization.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- Data pertaining to AEs will be collected during each trial visit either based on the trial subject's spontaneous description or investigator's inquiry or discovered in the course of examinations done during the visit, clinical significance of any sign or symptom needs to be evaluated by the investigator.
- Clinically significant findings need to be documented as AEs in the source data and CRF. Findings that are evaluated and documented in the source data as not clinically significant (e.g., an abnormal laboratory value without any clinical manifestation), should not be documented as AE.
- The investigator will then record all relevant AE information in the CRF and perform an assessment on:
  - Intensity, see the section "Assessment of intensity" in Section 10.3.1.11 for guidance on the assessment of intensity
  - Seriousness
  - Outcome
  - Causal relationship of the AE to the trial treatment
  - Any trial treatment action and/or any other action taken
- All assessments as well as AE term (diagnosis/description), start date and time of onset, end date and time need to be documented in the CRF.
- There may be instances when copies of medical records for certain cases are requested by the sponsor. In this case, all trial subject identifiers, with the exception of the trial subject number, will be redacted on the copies of the medical records before submission to the sponsor.
- To avoid colloquial expressions, the AE should be reported in standard medical terminology. The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE. If a definitive diagnosis is not possible, the individual signs and symptoms should be recorded.

#### Assessment of AE and/or SAE intensity

For subjects in yet to be started cohorts, the assessment of AE and/or SAE intensity should be done as described in protocol version 7.0 (which includes amendment 04).

The assessment of AE and/or SAE intensity should be done consistently for all subjects treated with the same treatment and dose.

All subjects treated in completed cohorts, where the first treatment pre-dates approval of the protocol version 5.0 (i.e., including amendment 04), should continue to use the grading scheme in the earlier protocol version, such that the same grading scheme is used consistently for all subjects given the same treatment and dose.

Where applicable, retrospective re-mapping of grading from 3-point to 4-point scale will be completed prior to database lock, with definitions for mild and moderate intensity events

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


aligned and all events previously graded as severe intensity (on 3-point scale), queried to determine whether Grade 3 (severe) or 4 (potentially life-threatening) should be applied.

In case of doubt, the Medical Monitor should be consulted.

The intensity of AEs or SAEs will be graded by the investigator. For further guidance on grading of solicited reactions, please refer to guideline "US FDA Guidance for Industry. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". Where specific guidance for an adverse event term is not provided, the following general approach should be followed:

- Grade 1 Mild; does not interfere with the subject's usual function.
- Grade 2 Moderate; interferes to some extend with the subject's usual function.
- Grade 3 Severe; interferes significantly with the subject's usual function.
- Grade 4 Potentially life-threatening; life-threatening consequences, urgent intervention required.

Please also refer to the intensity tables given in the guideline for intensity of clinical and laboratory abnormalities to be reported as AEs:

• Guideline Section III.A for assessment of clinical abnormalities (local and systemic)

### Actions taken by the investigator

Actions taken by the investigator as a result of an AE must be documented.

Action(s) taken with trial treatment (IMPs) by the investigator:

- Dose not changed (= continuation of trial treatment administration according to the trial protocol)
- Dose reduced
- Drug interrupted; i.e., interruption of IMP administration during a given visit
- Drug withdrawn
- Unknown (e.g., in case the trial subject is lost to follow-up)
- Not applicable (e.g., in case treatment with trial treatment has not yet started or event starts after last trial treatment administration)

Other action(s) that may be taken by the investigator include:

- None
- Remedial drug therapy
- Other specific treatment(s) of AE (to be specified)

#### **Outcome**

The investigator has to assess the outcome of an AE (and not the trial subject's outcome) at the time of documentation based on the following criteria:

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


- Recovered/resolved\* (= complete resolution of the AE)
- Recovering/resolving (= AEs which are improving but not yet resolved completely, e.g., decrease in an intensity grade)
- Not recovered/not resolved (= AEs which are ongoing without improving or still
  present when the trial subject deceases due to another cause)
- Recovered/resolved with sequelae\* (= trial subject recuperated but retained pathological conditions resulting from the AE; the sequelae should be indicated)
- Fatal\*\* (= death due to the AE)
- Unknown (e.g., in case the trial subject is lost to follow-up)
- \* Generally, an AE is defined as recovered/resolved if all symptoms have ceased, no medication for treatment of the event is taken anymore and no other measures (e.g., hospitalization) are ongoing.

If the trial subject has developed permanent or chronic symptoms or if the event requires long term medication(s), the AE is defined as recovered/resolved with sequelae as soon as no changes of symptoms and/or medication(s) are expected anymore.

An AE that is documented as a worsening of a medical condition already known at baseline, is defined as recovered as soon as the medical condition has returned to baseline status.

\*\* In case of a fatal event, the event term should not be "death" but the underlying event which led to death (death = outcome). If there is more than one AE in a fatal case, only the AE leading to death will be attributed with the outcome "fatal". All other AEs ongoing at the time of death will be attributed with the outcome "not recovered/not resolved". A copy of an autopsy report should be submitted if available.

#### Assessment of causality

The investigator is obligated to assess the relationship between trial treatment/trial procedure and each occurrence of each AE/SAE.

The investigator will use clinical judgment to determine the relationship.

Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to trial treatment administration will be considered and investigated.

It is sufficient to document the causality in the source data and CRF as:

- Related (= there is a reasonable possibility of a causal relationship) or
- Not related (= there is <u>no reasonable possib</u>ility of a causal relationship)

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### Relationship to trial treatment

- The relationship or association of an AE or SAE to a trial treatment will be made by the investigator after having evaluated all accessible data and, if necessary, he/she will re-evaluate the case as new information becomes available.
- Events caused by the procedure of trial treatment administration should be differentiated from events caused by the trial treatment itself. Only events suspected to be caused by the IMPs itself should be documented as suspected Relationship to trial procedures.
- In this trial, it cannot be excluded that during the course of the trial some
  procedures give rise to AEs which are related to the trial procedure and not to the
  trial treatment. Procedure-related AEs can occur on the site of injection of the trial
  treatment e.g., redness, swelling, hematoma or itching or during or after trialspecific procedure, e.g., discomfort after blood drawing.
- There may be situations in which an SAE has occurred and the investigator has
  minimal information to include in the initial report to the sponsor. However, it is very
  important that the investigator always makes an assessment of causality for every
  event before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### 10.3.1.8 SAE exemptions

In general, SAEs are defined according to ICH Topic E2A (CPMP/ICH/377/95), EU Directive 2001/20/EC and ENTR/CT-3 (see Section 10.3.1.4).

In the present trial, some events are excluded from the SAE definition. The following events do not need to be reported as SAEs:

- AEs and SAEs occurring after trial subject discharge from the trial must only be reported by the investigator to the sponsor if a relationship to trial treatment or trial procedure is suspected.
- Planned hospitalizations required by the protocol (e.g., for trial treatment administration) will not be considered as reportable SAE.

#### 10.3.1.9 Documentation of particular situations

#### **AEs that are secondary to other events:**

In general, AEs that are secondary to other events (e.g., cascade events or clinical sequelae) should be identified by their primary cause, with the exception of severe or serious secondary events. A medically significant secondary AE that is separated in time

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


from the initiating event should be documented as an independent AE in source data and CRF. For example:

- If vomiting results in mild dehydration with no additional treatment in a healthy adult, only vomiting should be documented as AE.
- If vomiting results in severe dehydration, both events should be documented as AEs separately.

### Abnormal laboratory results and vital signs values:

Not every laboratory or vital signs abnormality needs to be documented as AE. For clinically significant laboratory/vital signs abnormalities the following definitions and documentation rules apply:

- If a laboratory/vital signs abnormality is a sign of a disease or syndrome, the laboratory/vital signs abnormality is clinically significant and only the diagnosis of the causing disease or syndrome needs to be documented as AE.
- If a laboratory/vital signs abnormality results in specific symptoms but no diagnosis of a disease or syndrome can be made, the laboratory/vital signs abnormality is clinically significant and only the symptoms need to be documented as AEs.
- If a laboratory/vital signs abnormality is not a sign of a disease or syndrome and does not result in specific symptoms but leads to a change in trial treatment or in a medical intervention, the laboratory/vital signs abnormality is clinically significant and must be documented as AE.
- If a laboratory/vital signs abnormality is not considered clinically significant by the investigator, then an AE does not need to be documented.

#### AEs associated with an overdose or error in drug administration:

An overdose is the accidental or intentional use of a drug in an amount (per administration or cumulatively) higher than the dose being studied (for the trial treatment) or higher than the maximum recommended dose according to the authorized product information (for approved concomitant medications). An overdose or incorrect administration of a drug is not itself an AE, but it may result in an AE.

All AEs associated with an overdose or incorrect administration should be documented as AE in source data and CRF and reported as SAE if applicable.

#### AEs of proven COVID-19 disease:

Any case of proven COVID-19 disease occurring till the last FU Visit should be reported as an SAE/AE. AEs which are rated as "moderate" or "severe" (according to the criteria provided in Section 10.3.1.7) will need to be reported as an SAE. If none of the other SAE definitions are deemed suitable, then the SAE criterion of being a "medically important event" should be applied (according to the definitions provided in Section 10.3.1.4). An SAE form should be completed, including follow-up information, as detailed in Section 10.3.1.10 such that an SAE report and narrative can be prepared and distributed.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


All mild cases of proven COVID-19 cases which do not correspond to seriousness criteria will be reported as AEs in the CRF.

### 10.3.1.10 Reporting of SAEs

All SAEs or DLTs (even if non-serious) which occur in a trial subject during the observation period, whether considered to be associated with trial medication or not, must be reported by the investigator to the sponsor within 24 h following knowledge of the event.

All SAEs occurring after the end of the period of observation only have to be reported to the sponsor if the investigator suspects a relationship to trial medication or the trial procedure.

### SAE reporting to sponsor using a paper form (SAE Report)

For the period of observation, see Section 8.3.1.

For any SAE or DLT (even if non-serious), the investigator needs to complete the paper <u>Serious Adverse Event Form</u> which must be sent to the sponsor via one of the following reporting methods:

| • | Safety Report fax no.: | +49 (0) 231 |
|---|-------------------------------|-------------|
| • | Safety Report e-mail address: | |

Information for final description and evaluation of a case report may not be available within the required time frames for reporting. Nevertheless, for regulatory purposes, initial reports should be submitted if the following minimal information is available:

- An identifiable trial subject (trial subject number)
- A suspected medicinal product
- An identifiable reporting source (investigator/trial site identification)
- An event or outcome that can be identified as serious

SAE follow-up information should be sent to the sponsor (indicating that this is a "follow-up" report using the SAE Form or the Additional Information and Follow-Up Form) without delay as described above and accompanied by appropriate anonymous supporting documentation (e.g., discharge letters, medical reports, or death certificates), until a final outcome and date are available. All confidential information (name, address, full day of birth) needs to be blackened before sending. In addition to a medical record, the investigator should complete an <u>Additional Information and Follow-Up Form</u>, which contains the SAE term and trial subject number.

A copy of the submitted SAE report must be retained on file by the investigator. If explicitly required according to national legislation, the investigator must submit copies of the SAEs to the IEC or authority and retain documentation of these submissions in the ISF.

| In case an investigator or any other trial to | am member ha | as questions on | sa <u>fety</u> | reporting |
|---|---|---|---|---|
| the sponsor may be contacted via e-mail: | | | | |

For medical questions, the sponsor's Medical Monitor for this trial should be contacted; contact details are given in the trial Safety Management Plan.


Version: 13.0

Date: 12 JAN 2022

10.3.1.11 Assessments of intensity for solicited local and systemic reactions and laboratory abnormalities

The grading of solicited local and systemic reactions, recorded in the patient diaries, will be according to the following guidance, in line with Guideline Section III.A for assessment of clinical abnormalities (local and systemic).

#### Local reactions

Redness and swelling / induration will be measured and recorded in centimeters and then categorized during analysis as absent, mild, moderate, severe, or potentially life-threatening, based on the grading scale in Table 11. Likewise, pain (perceived) and tenderness (elicited) at the injection site will be assessed by the trial subject as absent, mild, moderate, severe, or potentially life-threatening, according to the grading scale in Table 11.

Table 11: Local reaction grading scale

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially life-threatening (Grade 4) |
|---|---|---|---|---|
| Pain at the injection site | Does not interfere with activity | Interferes with activity | Prevents daily activity | Emergency room visit or hospitalization for severe pain |
| Tenderness | Mild discomfort to touch | Discomfort with movement | Significant discomfort at rest | Emergency room visit or hospitalization |
| Erythema/<br>redness <sup>a</sup> | 2.5 cm to 5.0 cm | >5.0 cm to 10.0 cm | >10 cm | Necrosis or exfoliative dermatitis |
| Induration/<br>swelling <sup>b</sup> | 2.5 cm to 5.0 cm | >5.0 cm to 10.0 cm | >10 cm | Necrosis |

a) In addition to grading the measured local reaction at the greatest single diameter, the measurement should be recorded as a continuous variable.

#### Systemic reactions (signs and symptoms)

Symptoms of vomiting, diarrhea, headache, fatigue, chills, new or worsened muscle pain, and new or worsened joint pain will be assessed by the participant as absent, mild, moderate, severe, or potentially life-threatening, according to the grading scale in Table 12.

b) Induration/swelling should be evaluated and graded using the functional scale as well as the actual measurement.


Version: 13.0

Date: 12 JAN 2022

Table 12: Systemic reaction grading scale

| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially life-threatening (Grade 4) |
|---|---|---|---|---|
| Vomiting | 1-2 times in 24 h | >2 times in 24 h | Requires IV hydration | Emergency room visit or hospitalization for hypotensive shock |
| Diarrhea | 2 to 3 loose stools in 24 h | 4 to 5 loose stools in<br>24 h | 6 or more loose stools in 24 h | Emergency room visit or hospitalization for severe diarrhea |
| Headache | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe headache |
| Fatigue/<br>tiredness | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe fatigue |
| Chills | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe chills |
| New or<br>worsened<br>muscle pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe new or worsened muscle pain |
| New or<br>worsened joint<br>pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room visit or hospitalization for severe new or worsened joint pain |

#### Fever

Fever is defined as an oral temperature of ≥38.0°C. Temperature will be measured and recorded to 1 decimal place and then categorized during analysis according to the scale shown in Table 13.

Table 13: Fever grading scale

| | Mild<br>(Grade 1) | | | Potentially life-threatening (Grade 4) |
|---|---|---|---|---|
| Fever | 38.0 to 38.4°C | 38.5 to 38.9°C | 39.0 to 40.0°C | >40.0°C |

If a fever of ≥39.0°C is recorded by a subject during the 7-day post-vaccination diary period, a telephone contact should occur to ascertain further details and determine whether a site or healthcare professional visit is clinically indicated. Only an investigator or medically qualified person is able to confirm a participant's fever as >40.0°C for recording in the trial database. If a participant experiences a confirmed fever >40.0°C, the investigator must immediately notify the sponsor and, if it is determined to be related to the administration of the trial intervention, further vaccinations will be discontinued in that participant (see Section 6.6.1).

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


### Laboratory abnormalities

Laboratory abnormalities will be graded according to the grading scheme given in Table 14.

Table 14: Laboratory abnormality grading scale

| | | | l _ | |
|---|---|---|---|---|
| Hematology | Mild | Moderate | Severe | Potentially life- |
| | (Grade 1) | (Grade 2) | (Grade 3) | threatening (Grade 4) |
| Hemoglobin (female) - g/dL | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 | <8.0 |
| Hemoglobin (female)<br>change from baseline<br>value - g/dL | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 | >5.0 |
| Hemoglobin (male) - g/dL | 12.5 – 13.5 | 10.5 – 12.4 | 8.5 – 10.4 | <8.5 |
| Hemoglobin (male)<br>change from baseline<br>value - g/dL | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 | >5.0 |
| WBC increase - cells/mm <sup>3</sup> | 10,800 – 15,000 | 15,001 – 20,000 | 20,001 - 25,000 | >25,000 |
| WBC decrease - cells/mm <sup>3</sup> | 2,500 - 3,500 | 1,500 – 2,499 | 1,000 – 1,499 | <1,000 |
| Lymphocytes decrease - cells/mm <sup>3</sup> | 750 – 1,000 | 500 – 749 | 250 – 499 | <250 |
| Neutrophils decrease - cells/mm <sup>3</sup> | 1,500 – 2,000 | 1,000 – 1,499 | 500 – 999 | <500 |
| Eosinophils - cells/mm <sup>3</sup> | 650 – 1,500 | 1,501 – 5,000 | >5,000 | Hypereosinophilic |
| Platelets decrease - cells/mm <sup>3</sup> | 125,000 - 140,000 | 100,000 - 124,000 | 25,000 - 99,000 | <25,000 |
| Chemistry | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially life-<br>threatening (Grade 4) |
| BUN - mg/dL | 23 – 26 | 27 – 31 | >31 | Requires dialysis |
| Creatinine - mg/dL | 1.5 – 1.7 | 1.8 – 2.0 | 2.1 – 2.5 | >2.5 or requires dialysis |
| Alkaline phosphatase - increase by factor | 1.1 – 2.0x ULN | 2.1 – 3.0x ULN | 3.1 – 10x ULN | >10x ULN |
| Liver function tests - ALT,<br>AST -<br>increase by factor | 1.1 – 2.5x ULN | 2.6 – 5.0x ULN | 5.1 – 10x ULN | >10x ULN |
| Bilirubin - when accompanied<br>by any increase in liver<br>function test -<br>increase by factor | 1.1 – 1.25x ULN | 1.26 – 1.5x ULN | 1.51 – 1.75x ULN | >1.75x ULN |
| Bilirubin - when liver function test is normal - increase by factor | 1.1 – 1.5x ULN | 1.6 – 2.0x ULN | 2.0 – 3.0x ULN | >3.0x ULN |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen; ULN = upper limit of normal; WBC = white blood cell.


## 10.4 Contraceptive guidance and collection of pregnancy information

#### 10.4.1 Definitions

#### **WOCBP**

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (e.g., amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before first dose of trial treatment, additional evaluation should be considered.

Women in the following categories are not considered WOCBP:

- Premenarchal
- Premenopausal female with 1 of the following:
- Documented hysterectomy
- Documented bilateral salpingectomy
- Documented bilateral oophorectomy

For trial subjects with permanent infertility due to an alternate medical cause other than the above (e.g., mullerian agenesis, androgen insensitivity), investigator discretion should be applied to determining trial entry.

Note: Documentation can come from the site personnel review of the trial subject's medical records, medical examination, or medical history interview.

#### Postmenopausal female

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

A high FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with more than one FSH measurement is required.

Females on HRT and whose menopausal status is in doubt will be required to use one of the non-estrogen hormonal highly effective contraception methods if they wish to continue their HRT during the trial. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before trial enrollment.

## 10.4.2 Contraception guidance

WOCBP must confirm that they practiced at least one highly effective form of contraception for the 14 d prior to Visit 0.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


WOCBP must practice a highly effective form of contraception during the trial, starting after Visit 0 and continuously until 60 d after receiving the last immunization. WOCBP must agree to require their male partners to use condoms during sexual contact (unless male partners are sterilized or infertile).

Men who are sexually active with a WOCBP and have not had a vasectomy must agree to practice a highly effective form of contraception with their female partner of childbearing potential during the trial, starting after Visit 0 and continuously until 60 d after receiving the last immunization.

Subjects with bilateral tubal occlusion, previous successful vasectomy or those who are truly abstinent or exclusively homosexual are deemed as being "not of reproductive potential".

The investigator or delegate should advise the subject how to achieve highly effective contraception. The following birth control methods may be considered as highly effective:

- Intrauterine device. a
- Intrauterine hormone-releasing system. <sup>a</sup>
- Combined estrogen and progestogen-based contraception: established use of oral, intravaginal, or transdermal hormonal methods of contraception.
- Progesterone-based contraception: established use of oral, injected, or implanted <sup>a</sup> hormonal methods of contraception.

## 10.4.3 Collection of pregnancy Information

Pregnancy information will only be collected after obtaining written informed consent from the pregnant female trial subject (or if a male trial subjects' partner becomes pregnant, written informed consent from both).

Pregnancy information will be collected for pregnancies that occurred after the start of trial intervention and until 60 d after the last administration of IMP for pregnant trial subjects (or until 60 d after the last administration of IMP to the male trial subject for pregnant female partners).

The initial and follow-up information must be documented on the paper-based <u>Pregnancy Reporting Form</u> and <u>submitted to the sponsor within 24 h</u> of learning of a trial subject's pregnancy/partner's pregnancy. The completed form needs to be sent to the Safety Report fax number or e-mail given in Section 10.3.1.10. Completed pregnancy forms must be signed by an investigator before faxing/mailing them to the sponsor. Blank reporting forms are provided to the investigator during the site initiation visit and are filed in the ISF.

The investigator will collect follow-up information on the trial subject/trial subject's partner and the neonate and the information will be forwarded to the sponsor. Pregnancy follow-up should describe the outcome of the pregnancy, including any voluntary or spontaneous termination, details of the birth, the presence or absence of any congenital abnormalities, birth defects, maternal or newborn complications and their presumed relation to the IMP.

<sup>&</sup>lt;sup>a</sup> Contraception methods that in the context of this guidance are considered to have low user dependency.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Generally, the follow-up will be of a duration determined in consultation with the pediatrician.

While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE.

A spontaneous abortion is always considered to be an SAE and will be reported as such. Any post-trial pregnancy related SAE considered reasonably related to the trial intervention by the investigator will be reported to the sponsor. While the investigator is not obligated to actively seek this information in former trial subjects, he or she may learn of an SAE through spontaneous reporting.

### 10.4.4 Sperm donation

Men must refrain from sperm donation, starting after Visit 0 and continuously until 60 d after receiving the last immunization.

#### 10.5 Genetics

Not applicable.

## 10.6 Liver safety: Suggested actions and follow-up assessments Not applicable.

## 10.7 Investigators and trial administrative structure

### 10.7.1 Investigators and trial site personnel

There must be an investigator at each trial site.

If the trial is conducted by a team of individuals at the trial site, the investigator leading and responsible for the team is called the principal investigator.

All persons assigned responsibility as principal investigator must sign a declaration of their responsibilities and their agreement to this protocol before any trial-related procedure is performed.

Curriculum vitae and/or other relevant documents confirming the current qualification of the investigators must be provided to the sponsor. This should include any previous training in the principles of GCP, experience obtained from work with clinical trials, and experience with trial subject care.

Documentation of all involved investigators must be maintained according to GCP and applicable regulatory requirements.

## 10.7.2 Trial site personnel assigned trial-related duties

The principal investigator or deputy may define appropriately qualified personnel at a trial site to perform significant trial-related procedures and/or to make trial-related decisions under his/her supervision. In this case, the principal investigator must maintain a signed

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


list of the persons to whom they delegate significant trial-related duties/responsibilities; the delegated trial-related duties/responsibilities must be specified in the list.

When personnel or responsibility changes are made, the principal investigator or deputy must ensure that the relevant documentation is updated before any trial-related activities are performed.

Documentation of all involved trial site personnel performing significant trial-related procedures and/or making trial-related decisions must be maintained according to GCP and applicable regulatory requirements.

### 10.7.3 Contract research organizations

Documentation of all involved CROs must be maintained according to GCP and applicable regulatory requirements. This includes documentation of any delegation of responsibilities to CROs.

### 10.7.4 The sponsor and sponsor's personnel

The trial sponsor listed on the title page accepts the responsibilities of the sponsor according to GCP and applicable regulatory requirements.

The sponsor must designate appropriately qualified personnel to advise on trial-related topics. The trial site will be provided with contact details for these personnel before any trial-related procedure is performed.

A list of key sponsor personnel involved in the preparation of this protocol and the conduct of the trial, including their full names, titles, roles, and responsibilities, must be maintained.

## 10.8 Country-specific requirements

Not applicable.


## 10.9 Other standard abbreviations and definitions

For trial-specific abbreviations, see the list of trial-specific abbreviations.

For definitions related to safety, see Section 10.3.

| Abbreviation | Explanation |
|---|---|
| AE | Adverse Event |
| BMI | Body Mass Index |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| D | Day(s) |
| DLT | Dose limit toxicity(ies) |
| DMC | Data Monitoring Committee |
| EDC | Electronic Data Capture (system) |
| EMA | European Medicines Agency |
| EoT | End of Treatment |
| FDA | (US) Food and Drug Administration |
| FSH | Follicle Stimulating Hormone |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practice |
| Н | Hour(s) |
| HIV | Human Immunodeficiency Virus |
| HRT | Hormonal Replacement Therapy |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation (of technical requirements for registration of pharmaceuticals for human use) |
| IEC | Independent Ethics Committee |
| IMP | Investigational Medicinal Product; in this trial, BNT162 vaccines |
| ISF | Investigator's Site File |
| min | Minute(s) |
| NSAID | Nonsteroidal Anti-Inflammatory Drug |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SoA | Schedule of Activities |
| SOC | System Organ Class |
| SRC | Safety Review Committee |
| SUSAR | Suspected Unexpected Serious Adverse Reactions |
| TEAE | Treatment-Emergent Adverse Event |
| TMF | Trial Master File |

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


| Abbreviation | Explanation |
|--------------|---------------------------------|
| US | United States (of America) |
| WHO | World Health Organization |
| wks | Week(s) |
| WOCBP | Women Of Childbearing Potential |

## 10.10 Protocol amendments and version updates

Changes made to the protocol using the protocol amendments are described in detail in the document Protocol Amendment History which is available upon request. This Protocol Amendment History is filed together with the protocol in the TMF.

#### 10.10.1 Protocol amendment no. 01

#### Amendment rationale

This amendment describes the replacement of the product codes BNT162c1 with BNT162c2. The RNA component of BNT162c1 encoded only the RBD of the S protein, the RNA component of BNT162c2 encodes a modified version of the full length S protein. BNT162c1 was replaced with BNT162c2 because of its superior immunogenicity profile in non-clinical studies.

This amendment describes changes made in response to feedback from the PEI (April 16<sup>th</sup>, 2020).

This amendment was issued before any trial subjects were enrolled into the trial.

#### 10.10.2 Protocol amendment no. 02

#### Amendment rationale

This amendment describes a dose adjustment for the vaccine BNT162c2 and the corrections of some inconsistencies and ambiguities.

This amendment was issued after some of the planned trial subjects have already been enrolled into the trial.

#### 10.10.3 Protocol amendment no. 03

#### Amendment rationale

This amendment describes updates in response to PEI and IEC feedback on protocol version 4.0.

This amendment was issued after some of the planned trial subjects have already been enrolled into the trial.


### 10.10.4 Protocol amendment no. 04

#### Amendment rationale

The changes planned by amendment 04 were discussed with the PEI on the basis of the submitted protocol version 6.0. Amendment 04 was revised in response to received feedback, to yield protocol version 7.0.

This amendment describes adaption of the protocol to:

- Allow the assessment of additional intermediate and low dose cohorts for BNT162b modRNA vaccine candidates to support identification of a suitable dose for Phase II/III evaluation.
- Allow the assessment of BNT162b1 modRNA vaccine candidate in elderly subjects, given its favorable safety, tolerability, and immunogenicity profile in younger adults to date and recently available non-human primate immunogenicity data for the BNT162b1 and other modRNA vaccine candidates.
- Plan the assessment of BNT162b2 modRNA vaccine candidate in elderly subjects.
- Allow the assessment of P/B cohorts for the BNT162c2 saRNA vaccine candidate.
- · Allow revision of safety assessment & dose limiting toxicity criteria.
- Add additional for blood draws for explorative biomarker/immunogenicity research purposes.

This amendment was issued after some of the planned trial subjects have already been enrolled into the trial.

#### 10.10.5 Protocol amendment no. 05

#### **Amendment rationale**

Amendment 05 address feedback obtained from the PEI and the IEC on protocol version 7.0. Some changes were also implemented to align data collection and reporting in this trial with the data collection and reporting in other trials with BNT162 vaccines candidates (to facilitate data merging).

This amendment will be issued after some of the planned trial subjects have already been enrolled into the trial.

### 10.10.6 Protocol amendment no. 06

#### Amendment rationale

Protocol amendment 6.0 implemented three additional cohorts (Cohorts 11, 12, and 13) comprising up to additional 150 trial subjects aged from 18 to 85 years receiving BNT162b2 only.

BNT162b2 has entered a Phase II/III evaluation of efficacy, with the intent to support an application for marketing authorization. The dosing regimen under investigation is two 30 µg BNT162b2 doses given ~21 d apart.

# Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


The expansion cohorts implemented by this amendment are intended to provide a more indepth characterization of the adaptive immune responses induced by BNT162b2, associated vaccine safety, and the impact of factors such as subject disposition and dosing posology on humoral and cell-mediated immunity. These cohorts will extend the safety data of BNT162b2 to a broader trial population and thus closer to the vaccine target population.



For further background on the scientific rationale for the expansion cohorts, see Section 4.2.

The planned dose of BNT162b2, two 30  $\mu$ g BNT162b2 doses given ~21 d apart, the same regime that has already been tested in the dose escalation phase of this trial and in almost 17,000 adult subjects, including those with acute and chronic illnesses, in the ongoing global Phase I/II/III trial BNT162-02/C4591001 (NCT04368728).

The three expansion cohorts are as follows:

- Cohort 11: Alternative posology cohort with 30 healthy adults who will receive BNT162b2 using one 3 μg prime dose and one 30 μg boost dose of BNT162b2 given approximately 21 d apart (P/B regimen).
- Cohort 12: Adaptive immune response cohort (including safety and long term immune response) with 90 healthy adults who will receive of two 30 μg BNT162b2 doses given approximately 21 d apart (P/B regimen).
- Cohort 13: Population expansion cohort (including safety and long term immune response) with 30 immunocompromised adults who will receive of two 30 μg BNT162b2 doses given approximately 21 d apart (P/B regimen).

This amendment also addresses feedback obtained from the PEI and the IEC on protocol version 8.0.

This amendment also introduces logistical simplifications, i.e., except for Cohorts 1 and 8, the minimum interval between dosed trial subjects has been reduced from 30 min to 15 min for the prime and boost doses in the still to be completed Cohorts 2 to 10 (inclusive). Also, the minimum interval has been set to at least 5 min for the prime and boost doses in Cohorts 11 and 12, and to 15 min (prime) and 5 min (boost for Cohort 13. This simplification/design is considered justified:

 Because all FIH cohorts for the different BNT162 vaccine variants have been completed.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


• Due to the extensive experience and exposure already achieved with BNT162 vaccine candidates, including that almost 17,000 trial subjects have been dosed at least once with BNT162b2 (see Table 10).

Further changes were implemented to align data collection and reporting in this trial with the data collection and reporting in other trials with BNT162 vaccines candidates (to facilitate data merging).

This amendment will be issued after some of the planned trial subjects have already been enrolled into the trial.

### 10.10.7 Protocol amendment no. 06 (protocol version 10.0)

#### **Update rationale**

As requested by the IEC, this update reverses the reductions of the intervals between the dosing of trial subjects implemented in protocol amendment no. 06 (protocol version 9.0) for Cohorts 1 to 10 and Cohort 13.

This update will be issued after some of the planned trial subjects have already been enrolled into the trial.

## 10.10.8 Protocol amendment no. 07 (protocol version 11.0)

#### **Update rationale**

This update implements: a change in the sponsor name; deletion of the subject wellbeing calls given the available clinical data for BNT162b2; added text to avoid under reporting of mild COVID-19 related events arising in the trial; addition of a blood draw for CD4<sup>+</sup> T-cell counting; removal of outdated content; correction of some errors; updates for clarification; updates of outdated data.

This update will be issued after some of the planned trial subjects have already been enrolled into the trial.

## 10.10.9 Protocol amendment no. 08 (protocol version 12.0)

### **Update rationale**

This update implements one additional independent cohort (Cohort 14) comprising an additional 20 trial subjects receiving BNT162b2. Biomarker data from Cohort 14 are intended to provide characterization of B cell and plasma cell immune responses induced by BNT162b2, and to allow assessment of the durability of responses induced by vaccination in addition to continued follow-up of vaccine safety.

There is also a change to concomitant medication reporting to allow capture of vaccinations, e.g., SARS-CoV-2 vaccinations.

Date: 12 JAN 2022


Version: 13.0

### 10.10.10 Protocol amendment no. 09 (protocol version 13.0)

#### **Update rationale**

This update implements changes to the follow-up visits of subjects in Cohorts 11 to 13 who receive non-trial SARS-CoV-2 vaccinations. For these subjects, blood samples for immunogenicity and cell-mediated immune testing will not be collected, and they will be discontinued from the BNT162-01 trial.

## 10.11 Data collection and management

The trial documentation must be adequate for the reconstruction of the trial.

## 10.11.1 Case report forms

The CRFs will be completed through use of an electronic data capture (EDC) system. Trial site personnel will receive training and have access to a manual for appropriate CRF completion. The CRFs will be submitted electronically to the sponsor via the system and should be handled in accordance with instructions from the sponsor.

All CRFs should be completed by designated, trained trial site personnel. CRFs should be reviewed, verified, and then electronically signed and dated by the investigator or a designee.

At the end of the trial, the investigator will receive trial subject data for his/her trial site in a readable format that must be kept with the trial records. Acknowledgment of receipt of the trial subject data will be required.

## 10.11.2 Trial subject reported outcomes

Not applicable.

### 10.11.3 Data management

The CRO (see the title page) will be responsible for data management of this trial, including quality checking of the data.

Data entered manually will be submitted to the sponsor through use of an EDC system, data extracts and reports. Trial sites will be responsible for data entry into the EDC system. In the event of discrepant data, the data management service provider will request data clarification from the trial sites, which the trial sites will resolve electronically in the EDC system.

The data management service provider will produce a Trial Data Validation Specification document that describes the quality checking to be performed on the data. CRFs and correction documentation will be maintained in the EDC system's audit trail.

Central laboratory data will be sent directly to the data management service provider.

System backups for data stored by the sponsor and records retention for the trial data will be in accordance with regulatory requirements.


## 10.11.4 Investigator's Site File and the Trial Master File

The principal investigator or deputy is responsible for the filing of all essential documents in an ISF. The sponsor is responsible for the timely filing of all essential documents in the TMF. As applicable, these files must be available at monitoring visits and during audits or regulatory inspections.

After trial completion, the principal investigator or deputy must ensure that all source data and documentation related to the trial is recorded, handled, and stored in a way that allows its accurate reporting, interpretation, and verification. The principal investigator or deputy must take measures to prevent accidental or premature destruction of these documents.

The principal investigator or deputy must keep the ISF, the source data/documentation arising from the trial according to the prescribed record retention period in the country and/or according to the hospital policy, but at least until informed by the sponsor that the trial-related records are no longer required.

#### 10.12 Other data

### 10.12.1 Demographic data

At screening, the following demographic data will be recorded for all trial subjects:

- Age (in years/months)
- Gender (male/female)
- Ethnic group

#### 10.12.2 Medical history

Medical history information will be recorded for at the times given in the SoA (Section 1.3).

#### 11 REFERENCES

BNT162 Investigator's brochure, current edition.

EMA 2017 guidance. Strategies to Identify and Mitigate Risks for First-in-Human and Early Clinical Trials with Investigational Medicinal Products. European Medicines Agency (EMA) Science Medicines Health (2017).

FDA Guidance 2007. US FDA Guidance for Industry. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.

Feldman RA, Fuhr R, Smolenov I, et al. mRNA vaccines against H10N8 and H7N9 influenza viruses of pandemic potential are immunogenic and well tolerated in healthy adults in phase 1 randomized clinical trials. Vaccine. 2019; 37(25): 3326-34.

ICH E7. Guideline for Industry - Studies in Support of Special Populations: Geriatrics. March 1994.

## Clinical Trial Protocol including Amendments Nos. 01 to 09 BNT162-01


Moyo N, Vogel AB, Buus S, et al. Efficient Induction of T Cells against Conserved HIV-1 Regions by Mosaic Vaccines Delivered as Self-Amplifying mRNA. Mol Ther Methods Clin Dev. 2018;12:32-46.

NCT02410733. Evaluation of the safety and tolerability of IV administration of a cancer vaccine in patients with advanced melanoma (Lipo-MERIT). Ongoing BioNTech clinical trial.

NCT03871348. A first-in-human dose escalation and expansion study to evaluate intratumoral administration of SAR441000 as monotherapy and in combination with cemiplimab in patients with advanced solid tumors. Ongoing BioNTech clinical trial.

NCT04368728. BNT162-02/C4591001. Study to describe the safety, tolerability, immunogenicity, and efficacy of RNA vaccine candidates against COVID-19 in healthy individuals.

Pardi N, Hogan MJ, Pelc RS, et al. Zika virus protection by a single low-dose nucleoside-modified mRNA vaccination. Nature. 2017;543(7644):248-251.

Rauch S, Jasny E, Schmidt KE, Petsch B. New Vaccine Technologies to Combat Outbreak Situations. Front Immunol. 2018;9:1963.

Sahin U, Karikó K, Türeci Ö. mRNA-based therapeutics - developing a new class of drugs. Nat Rev Drug Discov. 2014;13(10):759-780.

Vogel AB, Lambert L, Kinnear E, et al. Self-Amplifying RNA Vaccines Give Equivalent Protection against Influenza to mRNA Vaccines but at Much Lower Doses. Mol Ther. 2018;26(2):446-455.

WHO "Protection measures for persons who are in or have recently visited (past 14 days) areas where COVID-19 is spreading". Accessed at:

https://www.who.int/emergencies/diseases/novel-coronavirus-2019/advice-for-public

WHO Situation Report Nr. 85, April 15th, 2020. Accessed at:

https://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports/